CLINICAL TRIAL: NCT02443155
Title: A Randomised, Double-blind, Double-dummy, Placebo-controlled, Parallel-group Multi-centre Clinical Proof-of-principle Trial in Adult Subjects With Newly Diagnosed Type 1 Diabetes Mellitus Investigating the Effect of NNC0114-0006 and Liraglutide on Preservation of Beta-cell Function
Brief Title: A Clinical Proof-of-principle Trial in Adult Subjects With Newly Diagnosed Type 1 Diabetes Mellitus Investigating the Effect of NNC0114-0006 and Liraglutide on Preservation of Beta-cell Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9828-4150; 2014-001215-39 (EudraCT Number); U1111-1154-7172 (Other: WHO); REec-2015-1768 (Registry Identifier: Spanish registry)
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Results first posted 2021-01-11 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- NNC0114-0006 + Liraglutide (Experimental)
  Interventions: Drug: NNC0114-0006; Drug: liraglutide
- NNC0114-0006 + Placebo (Experimental)
  Interventions: Drug: NNC0114-0006; Drug: placebo
- Liraglutide + Placebo (Active Comparator)
  Interventions: Drug: liraglutide; Drug: placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: NNC0114-0006 — NNC0114-0006 12 mg/kg administered i.v (intravenously) every 6 weeks. Subjects will continue their pre-trial insulin treatment
  Arms: NNC0114-0006 + Liraglutide; NNC0114-0006 + Placebo
Drug: liraglutide — Liraglutide 1.8 mg administered s.c. (subcutaneously) daily. Subjects will continue their pre-trial insulin treatment
  Arms: Liraglutide + Placebo; NNC0114-0006 + Liraglutide
Drug: placebo — Placebo administered s.c (subcutaneously) or i.v ( intravenously). Subjects will continue their pre-trial insulin treatment
  Arms: Liraglutide + Placebo; NNC0114-0006 + Placebo; Placebo

SUMMARY:
This trial is conducted globally. The aim of this trial is to assess the clinical proof-of-principle of NNC0114-0006 and liraglutide on preservation of beta-cell function in adult subjects with newly diagnosed type 1 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* T1DM (type 1 diabetes mellitus) (as diagnosed clinically) for not more than 20 weeks prior to screening - Male or female, aged 18-45 (both inclusive) at the time of signing the informed consent form
* Non-fasting peak C-peptide higher or equal to 0.2 nmol/l at visit 2
* BMI (body mass index) higher or equal to 18.5 kg/m^2
* Presence of one or more islet specific auto antibodies (glutamic acid decarboxylase (GAD), islet antigen-2 (IA2) or zinc-transporter 8 (ZnT8)) at screening
* Insulin dependence unless in temporary spontaneous remission (honeymoon period)

Exclusion Criteria:

* Daily insulin usage above 1 U/kg per day at screening or use of continuous subcutaneous insulin infusion (CSII)
* History of recurrent (e.g. several times a year) of severe (e.g. pneumonia) or chronic infections or conditions predisposing to chronic infections (e.g., bronchiectasis and chronic osteomyelitis)
* History of severe systemic fungal infection within the past 12 months prior to screening unless treated and resolved with appropriate documented therapy
* Vaccination within 4 weeks before randomisation, Visit 3 (V3)
* Receipt of any other concomitant medications or herbal products that can influence the immune system within 90 days prior to screening (V1)
* History of pancreatitis (acute or chronic)
* Family or personal history of Multiple Endocrine Neoplasia Type 2 (MEN2) or Medullary Thyroid Carcinoma (MTC)
* Any past or current diagnosis of malignant neoplasms
* Known impairment of the immune system, except for T1DM, coeliac disease, alopecia, autoimmune antibodies not considered clinical important (e.g. thyroid antibodies without any clinically important thyroid disease), and vitiligo

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 308 (Actual)
Dates: Start 2015-11-10 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2019-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (97):
- United States (13):
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, Northridge, California
  - Novo Nordisk Investigational Site, Aurora, Colorado
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Teaneck, New Jersey
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Mesquite, Texas
- Austria (4):
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Innsbruck
  - Novo Nordisk Investigational Site, Salzburg
  - Novo Nordisk Investigational Site, Vienna
- Belgium (3):
  - Novo Nordisk Investigational Site, Brussels
  - Novo Nordisk Investigational Site, Edegem
  - Novo Nordisk Investigational Site, Leuven
- Canada (10):
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Vancouver, British Columbia
  - Novo Nordisk Investigational Site, Winnipeg, Manitoba
  - Novo Nordisk Investigational Site, Halifax, Nova Scotia
  - Novo Nordisk Investigational Site, Kingston, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Laval, Quebec
  - Novo Nordisk Investigational Site, Montreal, Quebec
  - Novo Nordisk Investigational Site, PQ, Quebec
  - Novo Nordisk Investigational Site, Sherbrooke, Quebec
- Denmark (3):
  - Novo Nordisk Investigational Site, Aarhus N
  - Novo Nordisk Investigational Site, Esbjerg
  - Novo Nordisk Investigational Site, Hellerup
- Finland (3):
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Oulu
  - Novo Nordisk Investigational Site, Tampere
- Ireland (2):
  - Novo Nordisk Investigational Site, Dublin
  - Novo Nordisk Investigational Site, Galway
- Israel (4):
  - Novo Nordisk Investigational Site, Holon
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Rehovot
- Italy (4):
  - Novo Nordisk Investigational Site, Bergamo
  - Novo Nordisk Investigational Site, Catanzaro
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Siena
- Norway (2):
  - Novo Nordisk Investigational Site, Oslo
  - Novo Nordisk Investigational Site, Stavanger
- Poland (3):
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Zabrze
- Portugal (6):
  - Novo Nordisk Investigational Site, Almada
  - Novo Nordisk Investigational Site, Amadora
  - Novo Nordisk Investigational Site, Braga
  - Novo Nordisk Investigational Site, Matosinhos Municipality
  - Novo Nordisk Investigational Site, Porto
  - Novo Nordisk Investigational Site, Viana do Castelo
- Russia (12):
  - Novo Nordisk Investigational Site, Arkhangelsk
  - Novo Nordisk Investigational Site, Chelyabinsk
  - Novo Nordisk Investigational Site, Dzerzhinskiy
  - Novo Nordisk Investigational Site, Kazan'
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Penza
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Saratov
  - Novo Nordisk Investigational Site, Syktyvkar
  - Novo Nordisk Investigational Site, Ulyanovsk
  - Novo Nordisk Investigational Site, Yoshkar-Ola
- Serbia (2):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Kragujevac
- Spain (7):
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Girona
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, Palma de Mallorca
  - Novo Nordisk Investigational Site, Sabadell
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Valencia
- Sweden (4):
  - Novo Nordisk Investigational Site, Gothenburg
  - Novo Nordisk Investigational Site, Karlstad
  - Novo Nordisk Investigational Site, Lund
  - Novo Nordisk Investigational Site, Stockholm
- Ukraine (3):
  - Novo Nordisk Investigational Site, Kyiv
  - Novo Nordisk Investigational Site, Vinnytsia
  - Novo Nordisk Investigational Site, Zhytomyr
- United Kingdom (12):
  - Novo Nordisk Investigational Site, Belfast
  - Novo Nordisk Investigational Site, Blackburn
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Cardiff
  - Novo Nordisk Investigational Site, Chester
  - Novo Nordisk Investigational Site, Edgbaston, Birmingham
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Newcastle upon Tyne
  - Novo Nordisk Investigational Site, Plymouth
  - Novo Nordisk Investigational Site, Sheffield
  - Novo Nordisk Investigational Site, Stevenage
  - Novo Nordisk Investigational Site, Swansea

REFERENCES:
- [Result] von Herrath M, Bain SC, Bode B, Clausen JO, Coppieters K, Gaysina L, Gumprecht J, Hansen TK, Mathieu C, Morales C, Mosenzon O, Segel S, Tsoukas G, Pieber TR; Anti-IL-21-liraglutide Study Group investigators and contributors. Anti-interleukin-21 antibody and liraglutide for the preservation of beta-cell function in adults with recent-onset type 1 diabetes: a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Diabetes Endocrinol. 2021 Apr;9(4):212-224. doi: 10.1016/S2213-8587(21)00019-X. Epub 2021 Mar 1. PMID 33662334
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 94 sites in Austria, Belgium, Canada, Denmark, Finland, Ireland, Israel, Italy, Norway, Poland, Portugal, Russian Federation, Spain, Sweden, Ukraine, the United Kingdom (UK), and the United States (US).
Pre-assignment Details: Participants were randomised in a 1:1:1:1 manner to one of the four treatment groups. One participant was randomised to liraglutide arm but was withdrawn from the trial before exposure to trial products as per investigator's decision.
Groups:
- NNC0114-0006 + Liraglutide (Experimental): Participants received 12 mg/kg dose of NNC0114-0006 every 6 weeks, intravenously for 54 weeks. Participants took 0.6 mg of liraglutide, once daily, subcutaneously, for first two weeks, 1.2 mg for next 2 weeks and 1.8 mg for rest of the treatment period. Participants received treatment for 54 weeks followed by an off-treatment observation period of 26 weeks. Participants continued their pre-trial insulin treatment throughout the trial.
- NNC0114-0006 (Experimental): Participants received 12 mg/kg dose of NNC0114-0006 every 6 weeks, intravenously for 54 weeks. Participants took liraglutide placebo once daily, subcutaneously, with the volume of placebo equivalent to the volume liraglutide 0.6 mg, 1.2 mg and 1.8 mg. Participants received treatment for 54 weeks followed by an off-treatment observation period of 26 weeks. Participants continued their pre-trial insulin treatment throughout the trial.
- Liraglutide (Experimental): Participants received NNC0114-0006 placebo (volume equivalent to NNC0114-0006 dose of 12 mg/kg) every 6 weeks, intravenously for 54 weeks. Participants took 0.6 mg of liraglutide, once daily, subcutaneously, for first two weeks, 1.2 mg for next 2 weeks and 1.8 mg for rest of the treatment period. Participants received treatment for 54 weeks followed by an off-treatment observation period of 26 weeks. Participants continued their pre-trial insulin treatment throughout the trial.
- Placebo (Placebo): Participants received NNC0114-0006 placebo (volume equivalent to NNC0114-0006 dose of 12 mg/kg) every 6 weeks, intravenously for 54 weeks. In addition to that, participants took liraglutide placebo once daily subcutaneously, with the volume of placebo equivalent to the volume liraglutide 0.6 mg, 1.2 mg and 1.8 mg. Participants received treatment for 54 weeks followed by an off-treatment observation period of 26 weeks. Participants continued their pre-trial insulin treatment throughout the trial.
Period: Overall Study
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Started | 77 | 77 | 76 | 77
Full Analysis Set | 77 | 77 | 76 | 77
PK Analysis Set | 21 | 21 | 22 | 20
Safety Analysis Set | 77 | 77 | 76 | 77
Completed | 65 | 63 | 67 | 61
Not Completed | 12 | 14 | 9 | 16
Not completed — Adverse Event | 3 | 4 | 1 | 2
Not completed — Unclassified | 0 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 4 | 7 | 3 | 9
Not completed — Pregnancy | 3 | 1 | 1 | 2
Not completed — Lost to Follow-up | 1 | 2 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 1 | 1
Not completed — Death | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Full analysis set (FAS) included all randomised participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo) | Total
Number analyzed (Participants) | 77 | 77 | 76 | 77 | 307
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (7.5) | 28.6 (7.9) | 28.0 (7.1) | 29.0 (7.0) | 28.4 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 32 | 25 | 28 | 106
  Male | 56 | 45 | 51 | 49 | 201
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 2 | 1 | 10
  Not Hispanic or Latino | 73 | 74 | 74 | 76 | 297
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 1 | 4
  White | 73 | 70 | 73 | 76 | 292
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 2 | 0 | 10

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve (AUC) 0-4h of Mixed Meal Tolerance Test (MMTT) Stimulated C-peptide at Week 54 Relative to Baseline
Description: Area under the concentration-time curve, from 0 to 4 hours (AUC0-4h) of a mixed meal tolerance test (MMTT) stimulated C-peptide at week 54 is presented as ratio to baseline. AUC of C-peptide was measured as Nano moles*hour per liter (nmol*h/L).
Time Frame: 0 - 4 hours post-dose on week 0 and week 54
Population: The FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AUC
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 66 | 65 | 68 | 63
Ratio of AUC | 0.934 (61.9) | 0.783 (45.5) | 0.709 (104.8) | 0.660 (86.3)
Statistical Analysis 1: Comparison: NNC0114-0006 + Liraglutide (Experimental) vs Placebo (Placebo); Ratio of week 54 to baseline are analysed using mixed model for repeated measurements (MMRM) with an unstructured covariance matrix. Treatment, stratum and sex as factors and log baseline value and age as covariates, including the interaction between visit and all variables; Test type: Superiority; p = 0.0017, Mixed model repeated measurements; Treatment ratio = 1.48, 95% CI 2-sided [1.16 to 1.89] — NNC0114-0006 + liraglutide / Placebo
Statistical Analysis 2: Comparison: NNC0114-0006 (Experimental) vs Placebo (Placebo); Ratio of week 54 to baseline are analysed using MMRM with an unstructured covariance matrix. Treatment, stratum and sex as factors and log baseline value and age as covariates, including the interaction between visit and all variables; Test type: Superiority; p = 0.0927, Mixed model repeated measurements; Treatment Ratio = 1.23, 95% CI 2-sided [0.97 to 1.57]
Statistical Analysis 3: Comparison: Liraglutide (Experimental) vs Placebo (Placebo); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.3780, Mixed model repeated measurements; Treatment Ratio = 1.12, 95% CI 2-sided [0.87 to 1.42]
Statistical Analysis 4: Comparison: NNC0114-0006 + Liraglutide (Experimental) vs NNC0114-0006 (Experimental); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.1377, Mixed model repeated measurements; Treatment ratio = 1.20, 95% CI 2-sided [0.94 to 1.53]
Statistical Analysis 5: Comparison: NNC0114-0006 + Liraglutide (Experimental) vs Liraglutide (Experimental); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0214, Mixed model repeated measurements; Treatment ratio = 1.33, 95% CI 2-sided [1.04 to 1.69]
Statistical Analysis 6: Comparison: NNC0114-0006 (Experimental) vs Liraglutide (Experimental); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.4187, Mixed model repeated measurements; Treatmrnt ratio = 1.10, 95% CI 2-sided [0.87 to 1.41]

2. Secondary Outcome: AUC0-2h of C-peptide at Week 54 Relative to Baseline
Description: Area under the concentration-time curve, from 0 to 2 hours (AUC0-2h) of a MMTT stimulated C-peptide at week 54 is presented as ratio to baseline. AUC of C-peptide was measured as 'nmol*h/L'.
Time Frame: 0-2 hours post-dose on week 0 and week 54
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AUC
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 66 | 65 | 68 | 63
Ratio of AUC | 0.961 (65.4) | 0.824 (53.0) | 0.646 (97.4) | 0.655 (87.3)

3. Secondary Outcome: Cmax of C-peptide at Week 54 Relative to Baseline
Description: Maximum observed concentration (Cmax) of a MMTT stimulated C-peptide at week 54 is presented as ratio to baseline. Cmax of C-peptide was measured as nanomoles per liter (nmol/L).
Time Frame: 0-4 hours post-dose on week 0 and week 54
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of Cmax
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 66 | 65 | 68 | 63
Ratio of Cmax | 0.978 (70.3) | 0.779 (47.6) | 0.733 (110.4) | 0.644 (89.4)

4. Secondary Outcome: AUC0-4h of Glucose at Week 54 Relative to Baseline
Description: Area under the concentration-time curve, from 0 to 4 hours (AUC0-4h) of a MMTT stimulated glucose at week 54 is presented as ratio to baseline. AUC of glucose was measured as Milli moles*hour per liter (mmol*h/L).
Time Frame: 0 - 4 hours post-dose on week 0 and week 54
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AUC
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 65 | 65 | 67 | 62
Ratio of AUC | 0.904 (33.1) | 1.078 (31.8) | 0.993 (34.2) | 1.089 (36.7)

5. Secondary Outcome: AUC0-2h of Glucose at Week 54 Relative to Baseline
Description: Area under the concentration-time curve, from 0 to 2 hours (AUC0-2h) of a MMTT stimulated glucose at week 54 is presented as ratio to baseline. AUC of glucose is measured as 'mmol*h/L'.
Time Frame: 0-2 hours post-dose on week 0 and week 54
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AUC
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 65 | 65 | 67 | 62
Ratio of AUC | 0.939 (28.5) | 1.066 (24.8) | 0.978 (31.9) | 1.057 (31.3)

6. Secondary Outcome: Cmax of Glucose at Week 54 Relative to Baseline
Description: Maximum observed concentration (Cmax) of a MMTT stimulated glucose at week 54 is presented as ratio to baseline. Cmax of C-peptide was measured as 'mmol/L'.
Time Frame: 0-4 hours post-dose on week 0 and week 54
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of Cmax
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 65 | 65 | 67 | 62
Ratio of Cmax | 0.937 (27.8) | 1.068 (25.4) | 1.004 (29.1) | 1.057 (30.9)

7. Secondary Outcome: Number of Treatment Emergent Adverse Events
Description: An adverse event was any untoward medical occurrence in a participants administered a product, and which did not necessarily have a causal relationship with this treatment. An adverse event was defined as treatment emergent if the onset of the adverse event occurs on or after the first day of trial product administration. Number of treatment emergent adverse events from first dose of trial product to week 54 and week 80 are presented. Results are based on the on-treatment and on-observation period.
  On-treatment period: From the day of first trial product administration to the day of the visit at week 54. On-observation: From the day after the visit at week 54 to the day of the last visit.
Time Frame: Week 0-54; Week 54-80
Population: The SAS included all participants who received at least one dose of the investigational product or comparator. Overall number of participants analyzed = participants with available data.
Measure: Number; unit: Adverse events
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Adverse events
  Week 0-54 | 434 | 327 | 410 | 364
  Week 54-80 | 70 | 73 | 78 | 87

8. Secondary Outcome: Number of Treatment Emergent Hyperglycaemic Episodes
Description: Hyperglycaemic episodes were defined as treatment-emergent if the onset occurred on or after the first day of trial product administration. Number of treatment emergent episodes of hyperglycaemic episodes from first dose of trial product to week 54 and from week 54 to week 80 are presented. Results are based on the on-treatment and on-observation period.
  On-treatment period: From the day of first trial product administration to the day of the visit at week 54. On-observation: From the day after the visit at week 54 to the day of the last visit.
Time Frame: Week 0-54; Week 54-80
Population: as for outcome 7
Measure: Number; unit: Episodes
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Episodes
  Week 0-54 | 302 | 256 | 217 | 291
  Week 54-80 | 306 | 74 | 352 | 112

9. Secondary Outcome: Number of Treatment Emergent Episodes of Diabetic Ketoacidosis
Description: Diabetic ketoacidosis episodes were defined as treatment-emergent if the onset occurred on or after the first day of trial product administration. Number of treatment emergent episodes of hyperglycaemic episodes from first dose of trial product to week 54 and from week 54 to week 80 are presented. Results are based on the on-treatment and on-observation period.
  On-treatment period: From the day of first trial product administration to the day of the visit at week 54. On-observation: From the day after the visit at week 54 to the day of the last visit.
Time Frame: Weeks 0-54; Weeks 54-80
Population: as for outcome 7
Measure: Number; unit: Episodes
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Episodes
  Week 0-54 | 0 | 0 | 0 | 0
  Week 54-80 | 0 | 0 | 1 | 1

10. Secondary Outcome: Number of Participants Experiencing Treatment Emergent Injection/Infusion Site Reactions Caused by NNC0114-0006/Liraglutide/Placebo Injection/Infusion
Description: Injection/infusion site reactions episodes were defined as treatment-emergent if the onset occurred on or after the first day of trial product administration. Number of participants experiencing treatment emergent episodes of injection/infusion site reactions episodes from first dose of trial product to week 54 (treatment period) is presented.
Time Frame: Week 0-54
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Participants | 2 | 0 | 0 | 1

11. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to the American Diabetes Association (ADA)
Description: Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 1 day after the date of last contact. Number of treatment-emergent hypoglycaemic episodes according to American Diabetes Association (ADA) classification from first dose of trial product to week 54 and from week 54 to week 80 are presented.
  Results presented hypoglycaemia episodes were recorded as per ADA definition: Severe hypoglycaemia, Documented symptomatic hypoglycaemia, Asymptomatic hypoglycaemia, Probable symptomatic hypoglycaemia and Pseudo-hypoglycaemia.
Time Frame: Weeks 0-54; Weeks 54-80
Population: as for outcome 7
Measure: Number; unit: Episodes
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Episodes
  Severe hypoglycaemia (Week 0-54) | 1 | 2 | 0 | 0
  Asymptomatic hypoglycaemia (Week 0-54) | 2038 | 1956 | 2092 | 1774
  Documented symptomatic hypoglycaemia (Week 0-54) | 1305 | 1461 | 1114 | 1625
  Pseudo-hypoglycaemia (Week 0-54) | 1 | 1 | 14 | 2
  Probable symptomatic hypoglycaemia (Week 0-54) | 9 | 0 | 4 | 10
  Severe hypoglycaemia (Week 54-80) | 3 | 1 | 0 | 1
  Asymptomatic hypoglycaemia (Week 54-80) | 609 | 522 | 670 | 449
  Documented symptomatic hypoglycaemia (Week 54-80) | 514 | 362 | 651 | 527
  Pseudo-hypoglycaemia (Week 54-80) | 0 | 0 | 1 | 2
  Probable symptomatic hypoglycaemia (Week 54-80) | 1 | 0 | 0 | 2

12. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to Novo Nordisk Definitions
Description: Hypoglycaemia episodes were recorded as per Novo Nordisk definition: Symptomatic BG-confirmed: An episode that is blood glucose (BG) confirmed by plasma glucose (PG) value <3.1 mmol/L with symptoms consistent with hypoglycaemia. Asymptomatic BG-confirmed: An episode that is BG-confirmed by PG value <3.1 mmol/L without symptoms consistent with hypoglycaemia. Severe or BG-confirmed symptomatic: An episode that is severe according to the ISPAD classification or BG-confirmed by a PG value <3.1 mmol/L with symptoms consistent with hypoglycaemia. BG-confirmed: An episode that is BG-confirmed by a PG value <3.1 mmol/L with or without symptoms consistent with hypoglycaemia. Severe or BG-confirmed: An episode that is severe according to the International Society for Pediatric and Adolescent Diabetes (ISPAD) classification or BG-confirmed by a PG value <3.1 mmol/L with or without symptoms consistent with hypoglycaemia.
Time Frame: Weeks 0-54; Weeks 54-80
Population: as for outcome 7
Measure: Number; unit: Episodes
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Episodes
  Severe or BG confirmed (Week 0-54) | 396 | 394 | 315 | 503
  Symptomatic BG confirmed (Week 0-54) | 576 | 616 | 479 | 646
  Severe or BG confirmed (Week 54-80) | 216 | 130 | 244 | 240
  Symptomatic BG confirmed (Week 54-80) | 368 | 207 | 332 | 292

13. Secondary Outcome: Change in Body Weight (kg)
Description: Change in body weight is measured at week 54 and week 80 respective to baseline. Body weight was measured in unit 'Kg'.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Kilogram (Kg)
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Kilogram (Kg)
  Change from week 0 to week 54: number analyzed (Participants) | 68 | 65 | 68 | 67
  Change from week 0 to week 54 | -1.8 (4.2) | 1.2 (5.0) | -2.5 (4.0) | 1.1 (6.1)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 64 | 68 | 62
  Change from week 0 to week 80 | 1.9 (4.6) | 1.6 (5.2) | 0.4 (4.7) | 2.8 (5.5)

14. Secondary Outcome: Diabetes Retinopathy
Description: Number of participants evaluated for diabetic retinopathy at baseline (Day -28 to -14), week 54 and week 80 are presented as 'yes', 'no' or 'unknown'.
Time Frame: Baseline, week 54 and week 80
Population: The SAS included all participants who received at least one dose of the investigational product or comparator. Number analyzed = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Participants
  Baseline (Day:-28 to -14): Yes | 4 | 2 | 1 | 1
  Baseline (Day:-28 to -14): No | 73 | 75 | 75 | 76
  Baseline (Day:-28 to -14): Unknown | 0 | 0 | 0 | 0
  Week 54: number analyzed (Participants) | 68 | 65 | 69 | 68
  Week 54: Yes | 3 | 2 | 1 | 0
  Week 54: No | 65 | 63 | 68 | 68
  Week 54: Unknown | 0 | 0 | 0 | 0
  Week 80: number analyzed (Participants) | 69 | 65 | 69 | 64
  Week 80: Yes | 3 | 2 | 1 | 0
  Week 80: No | 65 | 62 | 67 | 63
  Week 80: Unknown | 1 | 1 | 1 | 1

15. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR)- Ratio to Baseline
Description: The eGFR was measured using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula. Change in eGFR (measured in milliliters per minute per 1.73 square meters) from baseline (week 0) at week 54 and week 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of eGFR
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of eGFR
  Change from week 0 to week 54: number analyzed (Participants) | 67 | 65 | 67 | 66
  Change from week 0 to week 54 | 0.98 (10.3) | 0.95 (8.2) | 0.97 (10.2) | 1.00 (8.8)
  Change from week 0 to week 80: number analyzed (Participants) | 66 | 63 | 68 | 62
  Change from week 0 to week 80 | 0.97 (9.3) | 0.94 (11.4) | 0.96 (11.5) | 0.99 (10.9)

16. Secondary Outcome: Change in Haematology: Erythrocytes
Description: Change in erythrocytes (measured in 10^12 cells per liter) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio of erythrocytes
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
ratio of erythrocytes
  Change from week 0 to week 54: number analyzed (Participants) | 65 | 64 | 67 | 66
  Change from week 0 to week 54 | 0.99 (6.00) | 1.01 (6.3) | 0.99 (7.2) | 1.00 (6.0)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 64 | 68 | 62
  Change from week 0 to week 80 | 0.99 (6.7) | 1.00 (6.7) | 0.99 (7.00) | 1.00 (5.5)

17. Secondary Outcome: Change in Haematology: Haematocrit
Description: Change in haematocrit (measured in percentage '%') from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio of haematocrit
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
ratio of haematocrit
  Change from week 0 to week 54: number analyzed (Participants) | 65 | 64 | 67 | 66
  Change from week 0 to week 54 | 0.99 (6.6) | 1.00 (7.00) | 0.99 (7.8) | 1.00 (5.9)
  Change from week 0 to week 80: number analyzed (Participants) | 66 | 63 | 68 | 62
  Change from week 0 to week 80 | 0.98 (7.5) | 1.00 (7.3) | 0.98 (7.2) | 0.99 (5.8)

18. Secondary Outcome: Change in Haematology: Haemoglobin
Description: Change in haemoglobin (measured in millimoles per liter 'mmol/L') from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio of haemoglobin
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
ratio of haemoglobin
  Change from week 0 to week 54 | 1.01 (6.1) | 1.02 (7.2) | 1.00 (7.9) | 1.01 (5.6)
  Change from week 0 to week 80 | 1.00 (7.5) | 1.02 (8.2) | 1.00 (7.4) | 1.01 (5.6)

19. Secondary Outcome: Change in Haematology: Leukocytes
Description: Change in leukocytes (measured in 10^9 cells/L) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio of leukocytes
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
ratio of leukocytes
  Change from week 0 to week 54: number analyzed (Participants) | 65 | 64 | 67 | 66
  Change from week 0 to week 54 | 0.96 (27.1) | 0.98 (21.9) | 0.97 (23.2) | 1.02 (24.8)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 64 | 68 | 62
  Change from week 0 to week 80 | 0.99 (33.0) | 0.95 (19.9) | 0.99 (29.5) | 1.00 (24.9)

20. Secondary Outcome: Change in Haematology: Mean Corpuscular Hemoglobin
Description: Change in mean Corpuscular hemoglobin (measured in femtomole 'fmol') from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ratio of mean Corpuscular hemoglobin
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
ratio of mean Corpuscular hemoglobin
  Change from week 0 to week 54: number analyzed (Participants) | 65 | 64 | 67 | 66
  Change from week 0 to week 54 | 1.02 (3.6) | 1.01 (4.8) | 1.01 (4.0) | 1.01 (4.1)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 64 | 68 | 62
  Change from week 0 to week 80 | 1.02 (5.1) | 1.01 (6.6) | 1.01 (5.4) | 1.02 (4.3)

21. Secondary Outcome: Change in Haematology: Mean Corpuscular Hemoglobin Concentration
Description: Change in mean corpuscular hemoglobin concentration (MCHC) (measured in gram per liter 'g/L') from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of MCHC
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of MCHC
  Change from week 0 to week 54: number analyzed (Participants) | 65 | 64 | 67 | 66
  Change from week 0 to week 54 | 1.02 (2.9) | 1.01 (2.1) | 1.02 (2.6) | 1.02 (3.0)
  Change from week 0 to week 80: number analyzed (Participants) | 66 | 63 | 68 | 62
  Change from week 0 to week 80 | 1.02 (3.5) | 1.02 (3.1) | 1.02 (3.0) | 1.02 (0.29)

22. Secondary Outcome: Change in Haematology: Mean Corpuscular Volume
Description: Change in Mean Corpuscular volume (measured in femtoliter 'fL') from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio of mean corpuscular volume
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
ratio of mean corpuscular volume
  Change from week 0 to week 54: number analyzed (Participants) | 65 | 64 | 67 | 66
  Change from week 0 to week 54 | 1.00 (2.8) | 0.99 (3.8) | 1.00 (3.3) | 0.99 (3.3)
  Change from week 0 to week 80: number analyzed (Participants) | 66 | 63 | 68 | 62
  Change from week 0 to week 80 | 1.00 (4.3) | 1.00 (5.2) | 1.00 (4.3) | 0.99 (3.7)

23. Secondary Outcome: Change in Haematology: Thrombocytes
Description: Change in thrombocytes (measured in 10^9 cells per liter) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio of thrombocytes
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
ratio of thrombocytes
  Change from week 0 to week 54: number analyzed (Participants) | 65 | 64 | 66 | 65
  Change from week 0 to week 54 | 0.98 (14.5) | 0.98 (15.0) | 1.03 (13.2) | 0.98 (14.1)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 63 | 66 | 62
  Change from week 0 to week 80 | 1.00 (15.0) | 1.03 (15.7) | 1.04 (15.6) | 1.00 (17.3)

24. Secondary Outcome: Change in Haematology: Eosinophil
Description: Change in eosinophil (measured in percentage '%') from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Ratio of eosinophils
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of eosinophils
  Change from week 0 to week 54: number analyzed (Participants) | 64 | 64 | 66 | 66
  Change from week 0 to week 54 | 1.15 (0.65) | 1.30 (1.71) | 3.10 (13.79) | 1.37 (1.15)
  Change from week 0 to week 80: number analyzed (Participants) | 65 | 63 | 66 | 61
  Change from week 0 to week 80 | 1.31 (1.24) | 1.23 (1.03) | 1.54 (1.78) | 1.36 (1.27)

25. Secondary Outcome: Change in Haematology: Neutrophils
Description: Change in neutrophils (measured in percentage '%') from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio of neutrophils
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
ratio of neutrophils
  Change from week 0 to week 54: number analyzed (Participants) | 62 | 63 | 65 | 64
  Change from week 0 to week 54 | 0.98 (18.8) | 0.99 (17.6) | 0.97 (18.5) | 1.04 (17.8)
  Change from week 0 to week 80: number analyzed (Participants) | 63 | 62 | 65 | 59
  Change from week 0 to week 80 | 0.97 (17.5) | 0.99 (14.2) | 0.98 (20.7) | 1.04 (17.2)

26. Secondary Outcome: Change in Haematology: Basophils
Description: Change in basophils (measured in percentage '%') from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Ratio of basophils
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of basophils
  Change from week 0 to week 54: number analyzed (Participants) | 64 | 64 | 66 | 66
  Change from week 0 to week 54 | 1.73 (2.11) | 1.58 (1.52) | 1.52 (1.47) | 1.43 (1.06)
  Change from week 0 to week 80: number analyzed (Participants) | 65 | 63 | 66 | 61
  Change from week 0 to week 80 | 2.17 (2.17) | 1.73 (1.41) | 2.09 (1.86) | 1.96 (1.27)

27. Secondary Outcome: Change in Haematology: Lymphocytes
Description: Change in lymphocytes (measured in percentage '%') from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio of lymphocytes
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
ratio of lymphocytes
  Change from week 0 to week 54: number analyzed (Participants) | 64 | 64 | 66 | 66
  Change from week 0 to week 54 | 1.00 (28.5) | 1.00 (28.3) | 1.02 (28.4) | 0.91 (30.7)
  Change from week 0 to week 80: number analyzed (Participants) | 65 | 63 | 66 | 61
  Change from week 0 to week 80 | 1.01 (28.0) | 0.98 (21.8) | 0.99 (35.1) | 0.91 (30.6)

28. Secondary Outcome: Change in Haematology: Monocytes
Description: Change in monocytes (measured in percentage '%') from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio of monocytes
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
ratio of monocytes
  Change from week 0 to week 54: number analyzed (Participants) | 64 | 64 | 66 | 66
  Change from week 0 to week 54 | 1.05 (40.8) | 1.02 (34.8) | 1.01 (41.1) | 1.01 (34.9)
  Change from week 0 to week 80: number analyzed (Participants) | 65 | 63 | 66 | 61
  Change from week 0 to week 80 | 1.12 (44.0) | 1.07 (37.5) | 1.04 (42.9) | 1.12 (35.4)

29. Secondary Outcome: Change in Biochemistry: Alanine Aminotransferase (ALAT)
Description: Change in ALAT (measured in units per liter [U/L]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio of ALT
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
ratio of ALT
  Change from week 0 to week 54: number analyzed (Participants) | 66 | 65 | 66 | 65
  Change from week 0 to week 54 | 0.96 (47.7) | 0.98 (35.9) | 0.97 (46.0) | 0.90 (44.1)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 63 | 67 | 62
  Change from week 0 to week 80 | 0.95 (54.7) | 0.98 (39.5) | 1.06 (40.7) | 0.92 (40.6)

30. Secondary Outcome: Change in Biochemistry: Albumin
Description: Change in albumin (measured in gram per deciliter [g/dL]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ratio of albumin
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
ratio of albumin
  Change from week 0 to week 54: number analyzed (Participants) | 67 | 65 | 67 | 66
  Change from week 0 to week 54 | 0.99 (7.3) | 1.00 (6.00) | 1.02 (7.4) | 0.99 (7.5)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 63 | 68 | 62
  Change from week 0 to week 80 | 1.00 (6.7) | 1.01 (6.9) | 1.00 (6.7) | 0.99 (6.9)

31. Secondary Outcome: Change in Biochemistry: Amylase
Description: Change in amylase (measured in units per liter [U/L]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio of Amylase
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
ratio of Amylase
  Change from week 0 to week 54: number analyzed (Participants) | 66 | 65 | 67 | 66
  Change from week 0 to week 54 | 1.07 (20.7) | 0.98 (16.6) | 1.04 (18.9) | 1.01 (19.2)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 63 | 68 | 62
  Change from week 0 to week 80 | 1.04 (24.3) | 0.99 (14.9) | 1.03 (19.8) | 1.04 (26.1)

32. Secondary Outcome: Change in Biochemistry: Alkaline Phosphatase (ALP)
Description: Change in ALP (measured in units per liter [U/L]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of ALP
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of ALP
  Change from week 0 to week 54: number analyzed (Participants) | 66 | 65 | 67 | 66
  Change from week 0 to week 54 | 1.03 (28.6) | 0.99 (17.8) | 0.99 (18.1) | 1.03 (17.9)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 63 | 68 | 62
  Change from week 0 to week 80 | 1.07 (30.3) | 1.05 (16.5) | 1.04 (22.1) | 1.04 (21.7)

33. Secondary Outcome: Change in Biochemistry: Aspartate Aminotransferase (ASAT)
Description: Change in ASAT (measured in units per liter [U/L]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AST
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of AST
  Change from week 0 to week 54: number analyzed (Participants) | 66 | 64 | 64 | 65
  Change from week 0 to week 54 | 0.99 (39.3) | 0.99 (34.5) | 1.00 (57.0) | 0.98 (43.1)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 61 | 68 | 61
  Change from week 0 to week 80 | 0.98 (39.1) | 0.98 (32.4) | 1.09 (34.6) | 0.99 (39.3)

34. Secondary Outcome: Change in Biochemistry: Total Bilirubin
Description: Change in Total bilirubin (measured in micromole per liter [umol/L]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio of total bilirubin
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
ratio of total bilirubin
  Change from week 0 to week 54: number analyzed (Participants) | 66 | 65 | 67 | 66
  Change from week 0 to week 54 | 0.81 (61.7) | 1.10 (56.5) | 0.99 (49.8) | 1.01 (59.4)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 62 | 68 | 62
  Change from week 0 to week 80 | 0.91 (44.7) | 1.04 (74.8) | 0.98 (55.1) | 0.99 (58.7)

35. Secondary Outcome: Change in Biochemistry: Calcium Corrected
Description: Change in calcium corrected (measured in millimole per liter [mmol/L]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio of calcium
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
ratio of calcium
  Change from week 0 to week 54: number analyzed (Participants) | 67 | 65 | 67 | 66
  Change from week 0 to week 54 | 0.99 (3.7) | 0.98 (3.6) | 0.98 (4.0) | 0.99 (4.2)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 63 | 68 | 62
  Change from week 0 to week 80 | 0.96 (3.5) | 0.97 (4.0) | 0.98 (3.9) | 0.98 (4.0)

36. Secondary Outcome: Change in Biochemistry: Chloride
Description: Change in chloride (measured in millimole per liter [mmol/L]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio of chloride
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
ratio of chloride
  Change from week 0 to week 54: number analyzed (Participants) | 67 | 65 | 67 | 66
  Change from week 0 to week 54 | 1.01 (2.4) | 1.00 (2.2) | 1.00 (2.8) | 1.00 (3.1)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 63 | 68 | 62
  Change from week 0 to week 80 | 1.00 (2.3) | 1.01 (2.7) | 1.00 (3.0) | 1.00 (3.0)

37. Secondary Outcome: Change in Biochemistry: Creatine Kinase
Description: Change in creatine kinase (measured in units per liter [U/L]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of Creatine Kinase
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of Creatine Kinase
  Change from week 0 to week 54: number analyzed (Participants) | 66 | 64 | 64 | 65
  Change from week 0 to week 54 | 1.16 (86.3) | 1.17 (64.5) | 1.08 (140.2) | 1.02 (72.8)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 62 | 68 | 61
  Change from week 0 to week 80 | 1.11 (48.1) | 1.09 (68.3) | 1.24 (87.2) | 1.13 (76.5)

38. Secondary Outcome: Change in Biochemistry: Creatinine
Description: Change in creatinine (measured in micromole per liter [umol/L]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of Creatinine
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of Creatinine
  Change from week 0 to week 54: number analyzed (Participants) | 67 | 65 | 67 | 66
  Change from week 0 to week 54 | 1.01 (12.0) | 1.05 (10.6) | 1.04 (12.8) | 1.01 (9.9)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 63 | 68 | 62
  Change from week 0 to week 80 | 1.02 (11.2) | 1.05 (14.3) | 1.05 (13.1) | 1.02 (12.3)

39. Secondary Outcome: Change in Biochemistry: Gamma-glutamyl Transferase (GGT)
Description: Change in GGT (measured in units per liter [U/L]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of GGT
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of GGT
  Change from week 0 to week 54: number analyzed (Participants) | 66 | 65 | 66 | 66
  Change from week 0 to week 54 | 1.02 (38.6) | 1.08 (27.7) | 1.03 (37.2) | 1.02 (41.8)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 62 | 68 | 62
  Change from week 0 to week 80 | 1.05 (41.9) | 1.13 (29.4) | 1.10 (41.1) | 1.00 (36.8)

40. Secondary Outcome: Change in Biochemistry: C-reactive Protein Serum
Description: Change in C-reactive protein serum (measured in milligrams per liter [mg/L]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of C-reactive protein
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of C-reactive protein
  Change from week 0 to week 54: number analyzed (Participants) | 67 | 65 | 67 | 66
  Change from week 0 to week 54 | 0.92 (141.6) | 1.04 (93.0) | 0.89 (87.8) | 1.06 (78.0)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 63 | 68 | 62
  Change from week 0 to week 80 | 1.08 (103.8) | 0.94 (81.0) | 1.25 (134.7) | 1.06 (70.1)

41. Secondary Outcome: Change in Biochemistry: Lactate Dehydrogenase
Description: Change in Lactate Dehydrogenase (measured in units per liter [U/L]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of Lactate Dehydrogenase
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of Lactate Dehydrogenase
  Change from week 0 to week 54: number analyzed (Participants) | 64 | 61 | 62 | 59
  Change from week 0 to week 54 | 0.99 (12.6) | 1.03 (18.4) | 1.04 (23.3) | 1.03 (16.5)
  Change from week 0 to week 80: number analyzed (Participants) | 64 | 60 | 64 | 58
  Change from week 0 to week 80 | 1.02 (12.1) | 1.04 (19.6) | 1.09 (19.3) | 1.03 (17.8)

42. Secondary Outcome: Change in Biochemistry: Lipase
Description: Change in lipase (measured in units per liter [U/L]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of lipase
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of lipase
  Change from week 0 to week 54: number analyzed (Participants) | 67 | 65 | 67 | 66
  Change from week 0 to week 54 | 1.49 (36.6) | 1.00 (27.4) | 1.34 (36.2) | 1.01 (29.4)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 63 | 68 | 62
  Change from week 0 to week 80 | 1.05 (40.4) | 0.94 (27.2) | 1.02 (26.5) | 0.96 (37.2)

43. Secondary Outcome: Change in Biochemistry: Magnesium
Description: Change in magnesium (measured in millimole per liter [mmol/L]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of magnesium
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of magnesium
  Change from week 0 to week 54: number analyzed (Participants) | 66 | 65 | 67 | 66
  Change from week 0 to week 54 | 1.02 (8.9) | 1.01 (7.6) | 1.02 (7.8) | 0.99 (8.1)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 62 | 68 | 62
  Change from week 0 to week 80 | 1.01 (10.7) | 1.03 (11.2) | 1.02 (9.0) | 0.98 (9.2)

44. Secondary Outcome: Change in Biochemistry: Phosphate
Description: Change in phosphate (measured in millimole per liter [mmol/L]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of phosphate
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of phosphate
  Change from week 0 to week 54: number analyzed (Participants) | 66 | 65 | 66 | 66
  Change from week 0 to week 54 | 0.99 (16.0) | 0.99 (16.6) | 1.02 (13.9) | 0.96 (18.6)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 63 | 68 | 62
  Change from week 0 to week 80 | 1.02 (20.5) | 1.01 (16.9) | 1.03 (19.9) | 0.99 (17.4)

45. Secondary Outcome: Change in Biochemistry: Potassium
Description: Change in potassium (measured in millimole per liter [mmol/L]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of potassium
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of potassium
  Change from week 0 to week 54: number analyzed (Participants) | 66 | 64 | 64 | 65
  Change from week 0 to week 54 | 1.01 (8.1) | 0.98 (6.9) | 0.99 (8.3) | 0.98 (10.4)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 62 | 68 | 61
  Change from week 0 to week 80 | 0.99 (8.3) | 0.99 (6.9) | 0.98 (8.5) | 0.98 (10.0)

46. Secondary Outcome: Change in Biochemistry: Sodium
Description: Change in sodium (measured in millimole per liter [mmol/L]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of sodium
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of sodium
  Change from week 0 to week 54: number analyzed (Participants) | 67 | 65 | 67 | 66
  Change from week 0 to week 54 | 1.00 (1.9) | 1.00 (1.4) | 1.00 (1.9) | 1.00 (2.0)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 63 | 68 | 62
  Change from week 0 to week 80 | 0.99 (1.8) | 1.00 (2.1) | 1.00 (2.3) | 1.00 (1.8)

47. Secondary Outcome: Change in Biochemistry: Total Protein
Description: Change in total protein (measured in gram per liter [g/dL]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total protein
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of total protein
  Change from week 0 to week 54: number analyzed (Participants) | 66 | 65 | 67 | 66
  Change from week 0 to week 54 | 0.99 (6.8) | 1.00 (6.0) | 1.01 (7.2) | 1.00 (7.6)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 62 | 68 | 62
  Change from week 0 to week 80 | 0.99 (6.5) | 1.00 (6.4) | 1.00 (6.6) | 1.00 (7.4)

48. Secondary Outcome: Change in Biochemistry: Blood Urea Nitrogen Serum
Description: Change in blood urea nitrogen serum (measured in milligram per deciliter [mg/dL]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of Blood Urea Nitrogen serum
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of Blood Urea Nitrogen serum
  Change from week 0 to week 54: number analyzed (Participants) | 67 | 65 | 67 | 66
  Change from week 0 to week 54 | 1.00 (27.0) | 1.05 (22.4) | 0.98 (22.0) | 0.94 (23.3)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 63 | 68 | 62
  Change from week 0 to week 80 | 0.97 (33.2) | 0.97 (26.2) | 0.98 (28.9) | 0.97 (28.2)

49. Secondary Outcome: Change in Biochemistry: Uric Acid
Description: Change in Uric Acid (measured in milligram per deciliter [mg/dL]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of uric acid
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of uric acid
  Change from week 0 to week 54: number analyzed (Participants) | 67 | 65 | 67 | 66
  Change from week 0 to week 54 | 0.93 (21.3) | 0.98 (17.6) | 0.98 (18.8) | 0.96 (18.0)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 62 | 68 | 62
  Change from week 0 to week 80 | 0.95 (17.1) | 0.94 (19.1) | 0.96 (22.2) | 0.95 (19.6)

50. Secondary Outcome: Change in International Normalised Ratio (INR)
Description: Change in INR (measured in ratio]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of INR
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of INR
  Change from week 0 to week 54: number analyzed (Participants) | 64 | 64 | 64 | 64
  Change from week 0 to week 54 | 0.97 (9.5) | 0.96 (10.4) | 0.95 (9.8) | 0.96 (13.7)
  Change from week 0 to week 80: number analyzed (Participants) | 66 | 61 | 66 | 59
  Change from week 0 to week 80 | 0.98 (12.4) | 0.99 (12.9) | 0.96 (9.2) | 0.97 (11.5)

51. Secondary Outcome: Change in D-Dimer
Description: Change in D-Dimer (measured in mg/L) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of D-dimer
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of D-dimer
  Change from week 0 to week 54: number analyzed (Participants) | 65 | 65 | 66 | 66
  Change from week 0 to week 54 | 0.96 (37.6) | 0.98 (53.9) | 0.98 (56.8) | 1.15 (107.1)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 62 | 66 | 61
  Change from week 0 to week 80 | 0.96 (43.7) | 0.92 (61.3) | 1.05 (60.0) | 1.10 (74.3)

52. Secondary Outcome: Change in Lipids: Total Cholesterol (Ratio to Baseline)
Description: Change in total cholesterol (measured in mmol/L) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of total cholesterol
  Change from week 0 to week 54: number analyzed (Participants) | 66 | 65 | 67 | 66
  Change from week 0 to week 54 | 1.00 (13.8) | 1.02 (14.1) | 1.03 (16.2) | 1.04 (16.8)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 63 | 68 | 62
  Change from week 0 to week 80 | 1.02 (15.5) | 1.03 (14.1) | 1.07 (15.0) | 1.03 (18.4)

53. Secondary Outcome: Change in Lipids: Free Fatty Acids (Ratio to Baseline)
Description: Change in total free fatty acids (measured in mmol/L) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of free fatty acids
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of free fatty acids
  Change from week 0 to week 54: number analyzed (Participants) | 66 | 60 | 65 | 66
  Change from week 0 to week 54 | 0.86 (94.5) | 1.01 (114.4) | 1.18 (82.5) | 0.97 (68.7)
  Change from week 0 to week 80: number analyzed (Participants) | 66 | 59 | 64 | 61
  Change from week 0 to week 80 | 0.89 (85.3) | 1.06 (112.8) | 1.19 (92.8) | 0.94 (84.0)

54. Secondary Outcome: Change in Lipids: HDL Cholesterol (Ratio to Baseline)
Description: Change in HDL cholesterol (measured in mmol/L) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL cholesterol
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of HDL cholesterol
  Change from week 0 to week 54: number analyzed (Participants) | 67 | 65 | 67 | 66
  Change from week 0 to week 54 | 1.04 (17.3) | 1.08 (18.2) | 1.12 (19.6) | 1.10 (20.2)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 62 | 68 | 62
  Change from week 0 to week 80 | 1.04 (18.7) | 1.06 (16.7) | 1.14 (21.5) | 1.07 (22.2)

55. Secondary Outcome: Change in Lipids: LDL Cholesterol (Ratio to Baseline)
Description: Change in LDL cholesterol (measured in mmol/L) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL cholesterol
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of LDL cholesterol
  Change from week 0 to week 54: number analyzed (Participants) | 66 | 65 | 67 | 66
  Change from week 0 to week 54 | 0.96 (17.8) | 0.97 (20.9) | 0.98 (24.0) | 1.01 (23.6)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 62 | 68 | 62
  Change from week 0 to week 80 | 0.99 (22.2) | 1.02 (21.2) | 1.02 (21.2) | 1.03 (29.2)

56. Secondary Outcome: Change in Lipids: Triglycerides (TG) (Ratio to Baseline)
Description: Change in Triglycerides (measured in mmol/L) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of TG
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of TG
  Change from week 0 to week 54: number analyzed (Participants) | 66 | 65 | 67 | 66
  Change from week 0 to week 54 | 1.03 (46.2) | 0.96 (39.5) | 1.03 (49.2) | 1.02 (54.7)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 63 | 68 | 62
  Change from week 0 to week 80 | 1.08 (45.6) | 0.94 (45.1) | 1.09 (51.5) | 0.95 (50.4)

57. Secondary Outcome: Change in Total Immunoglobulin E (IgE)
Description: Change in IgE (measured in kilo international units per liter [kIU/L]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of IgE
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of IgE
  Change from week 0 to week 54: number analyzed (Participants) | 68 | 65 | 68 | 66
  Change from week 0 to week 54 | 1.31 (71.6) | 1.05 (63.1) | 1.08 (45.7) | 1.02 (41.8)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 64 | 68 | 62
  Change from week 0 to week 80 | 1.32 (65.4) | 1.18 (38.5) | 1.16 (55.1) | 0.94 (61.2)

58. Secondary Outcome: Change in Urinalysis: Urine Dipsticks
Description: Urinalysis was performed by urine dipsticks for protein, glucose, erythrocytes, ketones leukocytes, nitrite, pH and specific gravity and categorised as normal, abnormal not clinically significant (NCS) and abnormal clinially significant (CS). Number of participants in each category at baseline (week 0), week 54 and 80 are presented.
Time Frame: Week 0, week 54 and week 80
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Participants
  Week 0: Glucose dipstick: Normal | 72 | 71 | 67 | 71
  Week 0: Glucose dipstick: Abnormal, NCS | 5 | 6 | 9 | 6
  Week 0: Glucose dipstick: Abnormal, CS | 0 | 0 | 0 | 0
  Week 54: Glucose dipstick: number analyzed (Participants) | 68 | 65 | 68 | 65
  Week 54: Glucose dipstick: Normal | 57 | 56 | 63 | 59
  Week 54: Glucose dipstick: Abnormal, NCS | 9 | 9 | 5 | 6
  Week 54: Glucose dipstick: Abnormal, CS | 2 | 0 | 0 | 0
  Week 80: Glucose dipstick: number analyzed (Participants) | 66 | 64 | 68 | 62
  Week 80: Glucose dipstick: Normal | 54 | 54 | 54 | 51
  Week 80: Glucose dipstick: Abnormal, NCS | 12 | 10 | 13 | 11
  Week 80: Glucose dipstick: Abnormal, CS | 0 | 0 | 1 | 0
  Week 0: Ketone dipstick: Normal | 74 | 73 | 73 | 76
  Week 0: Ketone dipstick: Abnormal, NCS | 2 | 4 | 3 | 1
  Week 0: Ketone dipstick: Abnormal, CS | 1 | 0 | 0 | 0
  Week 54: Ketone dipstick: number analyzed (Participants) | 68 | 65 | 68 | 65
  Week 54: Ketone dipstick: Normal | 68 | 64 | 65 | 64
  Week 54: Ketone dipstick: Abnormal, NCS | 0 | 1 | 3 | 1
  Week 54: Ketone dipstick: Abnormal, CS | 0 | 0 | 0 | 0
  Week 80: Ketone dipstick: number analyzed (Participants) | 66 | 64 | 68 | 62
  Week 80: Ketone dipstick: Normal | 65 | 61 | 66 | 61
  Week 80: Ketone dipstick: Abnormal, NCS | 1 | 3 | 1 | 1
  Week 80: Ketone dipstick: Abnormal, CS | 0 | 0 | 1 | 0
  Week 0: pH dipstick: Normal | 75 | 77 | 76 | 75
  Week 0: pH dipstick: Abnormal, NCS | 2 | 0 | 0 | 2
  Week 0: pH dipstick: Abnormal, CS | 0 | 0 | 0 | 0
  Week 54: pH dipstick: number analyzed (Participants) | 68 | 65 | 68 | 65
  Week 54: pH dipstick: Normal | 67 | 65 | 68 | 64
  Week 54: pH dipstick: Abnormal, NCS | 1 | 0 | 0 | 1
  Week 54: pH dipstick: Abnormal, CS | 0 | 0 | 0 | 0
  Week 80: pH dipstick: number analyzed (Participants) | 66 | 64 | 68 | 62
  Week 80: pH dipstick: Normal | 66 | 64 | 68 | 62
  Week 80: pH dipstick: Abnormal, NCS | 0 | 0 | 0 | 0
  Week 80: pH dipstick: Abnormal, CS | 0 | 0 | 0 | 0
  Week 0: Erythrocytes in urine: Normal | 74 | 74 | 74 | 72
  Week 0: Erythrocytes in urine: Abnormal, NCS | 2 | 3 | 2 | 4
  Week 0: Erythrocytes in urine: Abnormal, CS | 1 | 0 | 0 | 1
  Week 54: Erythrocytes in urine: number analyzed (Participants) | 68 | 65 | 68 | 65
  Week 54: Erythrocytes in urine: Normal | 66 | 63 | 66 | 63
  Week 54: Erythrocytes in urine: Abnormal, NCS | 2 | 2 | 2 | 2
  Week 54: Erythrocytes in urine: Abnormal, CS | 0 | 0 | 0 | 0
  Week 80: Erythrocytes in urine: number analyzed (Participants) | 66 | 64 | 68 | 62
  Week 80: Erythrocytes in urine: Normal | 63 | 61 | 65 | 60
  Week 80: Erythrocytes in urine: Abnormal, NCS | 3 | 3 | 3 | 2
  Week 80: Erythrocytes in urine: Abnormal, CS | 0 | 0 | 0 | 0
  Week 0: Leukocytes in urine: Normal | 77 | 73 | 76 | 77
  Week 0: Leukocytes in urine: Abnormal, NCS | 0 | 4 | 0 | 0
  Week 0: Leukocytes in urine: Abnormal, CS | 0 | 0 | 0 | 0
  Week 54: Leukocytes in urine: number analyzed (Participants) | 68 | 65 | 68 | 65
  Week 54: Leukocytes in urine: Normal | 64 | 62 | 67 | 64
  Week 54: Leukocytes in urine: Abnormal, NCS | 4 | 3 | 1 | 1
  Week 54: Leukocytes in urine: Abnormal, CS | 0 | 0 | 0 | 0
  Week 80: Leukocytes in urine: number analyzed (Participants) | 66 | 64 | 68 | 62
  Week 80: Leukocytes in urine: Normal | 62 | 61 | 67 | 60
  Week 80: Leukocytes in urine: Abnormal, NCS | 4 | 3 | 1 | 2
  Week 80: Leukocytes in urine: Abnormal, CS | 0 | 0 | 0 | 0
  Week 0: Nitrite: Normal | 77 | 77 | 76 | 77
  Week 0: Nitrite: Abnormal, NCS | 0 | 0 | 0 | 0
  Week 0: Nitrite: Abnormal, CS | 0 | 0 | 0 | 0
  Week 54: Nitrite: number analyzed (Participants) | 68 | 65 | 68 | 65
  Week 54: Nitrite: Normal | 68 | 65 | 68 | 65
  Week 54: Nitrite: Abnormal, NCS | 0 | 0 | 0 | 0
  Week 54: Nitrite: Abnormal, CS | 0 | 0 | 0 | 0
  Week 80: Nitrite: number analyzed (Participants) | 66 | 64 | 68 | 62
  Week 80: Nitrite: Normal | 65 | 64 | 68 | 61
  Week 80: Nitrite: Abnormal, NCS | 1 | 0 | 0 | 1
  Week 80: Nitrite: Abnormal, CS | 0 | 0 | 0 | 0
  Week 0: Protein urine: Normal | 77 | 71 | 75 | 76
  Week 0: Protein urine: Abnormal, NCS | 0 | 6 | 1 | 1
  Week 0: Protein urine: Abnormal, CS | 0 | 0 | 0 | 0
  Week 54: Protein urine: number analyzed (Participants) | 68 | 65 | 68 | 65
  Week 54: Protein urine: Normal | 67 | 64 | 62 | 61
  Week 54: Protein urine: Abnormal, NCS | 1 | 1 | 6 | 4
  Week 54: Protein urine: Abnormal, CS | 0 | 0 | 0 | 0
  Week 80: Protein urine: number analyzed (Participants) | 66 | 64 | 68 | 62
  Week 80: Protein urine: Normal | 63 | 62 | 65 | 59
  Week 80: Protein urine: Abnormal, NCS | 3 | 1 | 3 | 2
  Week 80: Protein urine: Abnormal, CS | 0 | 1 | 0 | 1
  Week 0: Specific Gravity: Normal | 75 | 77 | 76 | 75
  Week 0: Specific Gravity: Abnormal, NCS | 2 | 0 | 0 | 2
  Week 0: Specific Gravity: Abnormal, CS | 0 | 0 | 0 | 0
  Week 54: Specific Gravity: number analyzed (Participants) | 68 | 65 | 68 | 65
  Week 54: Specific Gravity: Normal | 67 | 65 | 68 | 64
  Week 54: Specific Gravity: Abnormal, NCS | 1 | 0 | 0 | 1
  Week 54: Specific Gravity: Abnormal, CS | 0 | 0 | 0 | 0
  Week 80: Specific Gravity: number analyzed (Participants) | 66 | 64 | 68 | 62
  Week 80: Specific Gravity: Normal | 65 | 64 | 68 | 62
  Week 80: Specific Gravity: Abnormal, NCS | 1 | 0 | 0 | 0
  Week 80: Specific Gravity: Abnormal, CS | 0 | 0 | 0 | 0

59. Secondary Outcome: Change in Cytokines: Interleukin (IL)-6
Description: IL-6 levels at baseline (week 0), weeks 54 and 80 are evaluated and presented.
Time Frame: Week 0, week 54 and week 80
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
picogram per milliliter (pg/mL)
  Week 0: number analyzed (Participants) | 77 | 76 | 74 | 75
  Week 0 | 0.9 (0.6) | 0.8 (0.1) | 1.2 (1.8) | 0.8 (0.3)
  Week 54: number analyzed (Participants) | 68 | 64 | 68 | 67
  Week 54 | 0.8 (0.3) | 0.8 (0.4) | 1.0 (0.8) | 0.8 (0.2)
  Week 80: number analyzed (Participants) | 67 | 63 | 68 | 62
  Week 80 | 0.9 (0.4) | 0.8 (0.2) | 0.9 (0.8) | 0.9 (0.4)

60. Secondary Outcome: Change in Cytokines- Interleukin (IL)-10
Description: IL-10 levels at baseline (week 0), weeks 54 and 80 are evaluated and presented.
Time Frame: Week 0, week 54 and week 80
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
pg/mL
  Week 0: number analyzed (Participants) | 77 | 75 | 74 | 75
  Week 0 | 0.7 (1.4) | 0.5 (1.1) | 0.4 (0.3) | 0.4 (0.2)
  Week 54: number analyzed (Participants) | 68 | 64 | 68 | 67
  Week 54 | 0.4 (0.2) | 0.4 (0.1) | 0.4 (0.3) | 0.4 (0.3)
  Week 80: number analyzed (Participants) | 67 | 63 | 68 | 62
  Week 80 | 0.4 (0.5) | 0.4 (0.2) | 0.5 (0.7) | 0.4 (0.1)

61. Secondary Outcome: Change in Cytokines: Interleukin (IL)-17
Description: IL-17 levels at baseline (week 0), weeks 54 and 80 are evaluated and presented.
Time Frame: Week 0, week 54 and week 80
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
pg/mL
  Week 0: number analyzed (Participants) | 77 | 76 | 74 | 76
  Week 0 | 4.9 (2.0) | 4.7 (0.7) | 4.7 (0.0) | 4.8 (0.9)
  Week 54: number analyzed (Participants) | 68 | 65 | 68 | 67
  Week 54 | 4.9 (1.9) | 4.8 (1.3) | 5.1 (3.5) | 5.4 (5.0)
  Week 80: number analyzed (Participants) | 67 | 63 | 68 | 62
  Week 80 | 4.9 (1.7) | 4.7 (0.0) | 4.8 (1.2) | 4.8 (1.0)

62. Secondary Outcome: Change in Cytokines: Interferon (IFN) Gamma
Description: IFN gamma levels at baseline (week 0), weeks 54 and 80 are evaluated and presented.
Time Frame: Week 0, week 54 and week 80
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
pg/mL
  Week 0: number analyzed (Participants) | 77 | 76 | 74 | 75
  Week 0 | 7.3 (16.1) | 7.8 (24.0) | 5.8 (11.6) | 4.3 (2.8)
  Week 54: number analyzed (Participants) | 68 | 64 | 68 | 67
  Week 54 | 4.6 (4.2) | 7.5 (19.6) | 5.0 (6.8) | 5.8 (7.0)
  Week 80: number analyzed (Participants) | 67 | 63 | 68 | 62
  Week 80 | 4.4 (2.8) | 4.9 (6.4) | 13.0 (57.5) | 4.5 (3.4)

63. Secondary Outcome: Change in Cytokines: TNF-alpha
Description: TNF-alpha levels at baseline (week 0), weeks 54 and 80 are evaluated and presented.
Time Frame: Week 0, week 54 and week 80
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
pg/mL
  Week 0: number analyzed (Participants) | 77 | 76 | 74 | 75
  Week 0 | 2.60 (1.69) | 2.32 (0.82) | 2.70 (1.73) | 3.06 (3.75)
  Week 54: number analyzed (Participants) | 68 | 64 | 68 | 67
  Week 54 | 2.36 (0.75) | 2.33 (0.59) | 2.56 (1.11) | 2.43 (0.65)
  Week 80: number analyzed (Participants) | 67 | 63 | 68 | 62
  Week 80 | 2.43 (0.66) | 2.36 (0.68) | 2.96 (2.39) | 2.75 (2.47)

64. Secondary Outcome: Change in Hormone Level: Thyroid Stimulating Hormone (TSH)
Description: Change in TSH (measured in milli international units per liter [mIU/L]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of Thyroid Stimulating Hormone
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of Thyroid Stimulating Hormone
  Change from week 0 to week 54: number analyzed (Participants) | 66 | 65 | 67 | 66
  Change from week 0 to week 54 | 1.00 (49.9) | 1.12 (54.1) | 0.89 (46.6) | 0.91 (66.1)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 63 | 68 | 62
  Change from week 0 to week 80 | 1.04 (46.7) | 0.99 (116.1) | 0.99 (48.5) | 0.93 (84.5)

65. Secondary Outcome: Change in Hormone Level: Calcitonin
Description: Change in Calcitonin (measured in nanogram per liter [ng/L]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of Calcitonin
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of Calcitonin
  Change from week 0 to week 54: number analyzed (Participants) | 66 | 63 | 65 | 67
  Change from week 0 to week 54 | 1.00 (43.5) | 0.90 (48.5) | 0.89 (57.2) | 0.88 (47.4)
  Change from week 0 to week 80: number analyzed (Participants) | 66 | 63 | 67 | 62
  Change from week 0 to week 80 | 0.85 (50.9) | 0.93 (41.8) | 0.82 (71.5) | 0.90 (64.5)

66. Secondary Outcome: Change in Systolic and Diastolic Blood Pressure
Description: Change in systolic blood pressure (SBP) and diastolic blood pressure (DBP) are evaluated from baseline (week 0) to weeks 54 and 80.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Millimeters of mercury (mmHg)
  Week 54: Systolic blood pressure: number analyzed (Participants) | 68 | 65 | 68 | 67
  Week 54: Systolic blood pressure | -3 (9) | 3 (9) | -2 (14) | 1 (11)
  Week 80: Systolic blood pressure: number analyzed (Participants) | 67 | 64 | 68 | 62
  Week 80: Systolic blood pressure | -1 (10) | 2 (11) | 1 (12) | 4 (10)
  Week 54: Diastolic blood pressure: number analyzed (Participants) | 68 | 65 | 68 | 67
  Week 54: Diastolic blood pressure | -0 (9) | 2 (9) | -1 (10) | -1 (8)
  Week 80: Diastolic blood pressure: number analyzed (Participants) | 67 | 64 | 68 | 62
  Week 80: Diastolic blood pressure | -0 (9) | 2 (9) | 1 (10) | 1 (10)

67. Secondary Outcome: Change in Pulse
Description: Change in pulse is evaluated from baseline (week 0) to weeks 54 and 80
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Beats/min
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Beats/min
  Change from week 0 to week 54: number analyzed (Participants) | 68 | 65 | 68 | 67
  Change from week 0 to week 54 | 3 (12) | 0 (12) | 6 (9) | 2 (8)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 64 | 68 | 62
  Change from week 0 to week 80 | -1 (10) | -1 (10) | 2 (10) | 1 (9)

68. Secondary Outcome: Change in Body Temperature
Description: Change in body temperature is evaluated from baseline (week 0) to weeks 54 and 80.
Time Frame: Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Degree celsius (C)
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Degree celsius (C)
  Change from week 0 to week 54: number analyzed (Participants) | 68 | 65 | 68 | 67
  Change from week 0 to week 54 | -0.1 (0.4) | 0.0 (0.6) | -0.1 (0.5) | -0.0 (0.3)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 64 | 67 | 62
  Change from week 0 to week 80 | -0.0 (0.4) | 0.1 (0.5) | 0.0 (0.5) | 0.0 (0.4)

69. Secondary Outcome: Change in Respiratory Rate
Description: Change in respiratory rate is evaluated from baseline (week 0) to weeks 54 and 80.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Breaths per minute
  Change from week 0 to week 54: number analyzed (Participants) | 68 | 65 | 68 | 67
  Change from week 0 to week 54 | -0.3 (2.2) | 0.1 (3.0) | 0.1 (2.5) | 0.6 (2.4)
  Change from week 0 to week 80: number analyzed (Participants) | 67 | 64 | 68 | 62
  Change from week 0 to week 80 | -0.3 (2.0) | -0.2 (2.7) | 0.1 (2.5) | 0.1 (2.2)

70. Secondary Outcome: Change in Electrocardiogram (ECG)
Description: The ECG was assessed by the investigator at baseline (week 0), week 54 and week 80 and categorised as normal, abnormal NCS or abnormal CS. Number of participants in each ECG category at baseline, week 54 and week 80 are presented.
Time Frame: Week 0, week 54 and week 80
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Participants
  Week 0: Normal | 62 | 65 | 60 | 63
  Week 0: Abnormal, NCS | 15 | 12 | 16 | 13
  Week 0: Abnormal, CS | 0 | 0 | 0 | 1
  Week 54: number analyzed (Participants) | 68 | 65 | 67 | 65
  Week 54: Normal | 54 | 48 | 55 | 46
  Week 54: Abnormal, NCS | 14 | 17 | 12 | 19
  Week 54: Abnormal, CS | 0 | 0 | 0 | 0
  Week 80: number analyzed (Participants) | 66 | 64 | 68 | 62
  Week 80: Normal | 51 | 48 | 53 | 50
  Week 80: Abnormal, NCS | 15 | 16 | 15 | 12
  Week 80: Abnormal, CS | 0 | 0 | 0 | 0

71. Secondary Outcome: Change in Eye-examination
Description: Dilated fundoscopy or fundus photography was performed by the investigator at week 0, week 54 and week 80. The results of the examination were interpreted for each eye (left/right) are categorised as normal, abnormal NCS or abnormal CS. Number of participants in each category at week 0, week 54 and week 80 are presented.
Time Frame: Week 0, week 54 and week 80
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Participants
  Week 0: Left eye ophthalmoscopy: Normal | 64 | 68 | 70 | 66
  Week 0: Left eye ophthalmoscopy: Abnormal, NCS | 13 | 9 | 6 | 11
  Week 0: Left eye ophthalmoscopy: Abnormal, CS | 0 | 0 | 0 | 0
  Week 54: Left eye ophthalmoscopy: number analyzed (Participants) | 68 | 63 | 69 | 64
  Week 54: Left eye ophthalmoscopy: Normal | 55 | 56 | 60 | 54
  Week 54: Left eye ophthalmoscopy: Abnormal, NCS | 12 | 7 | 9 | 9
  Week 54: Left eye ophthalmoscopy: Abnormal, CS | 1 | 0 | 0 | 1
  Week 80: Left eye ophthalmoscopy: number analyzed (Participants) | 66 | 62 | 65 | 59
  Week 80: Left eye ophthalmoscopy: Normal | 52 | 54 | 59 | 51
  Week 80: Left eye ophthalmoscopy: Abnormal, NCS | 11 | 8 | 6 | 8
  Week 80: Left eye ophthalmoscopy: Abnormal, CS | 3 | 0 | 0 | 0
  Week 0: Right eye ophthalmoscopy: Normal | 58 | 66 | 69 | 67
  Week 0: Right eye ophthalmoscopy: Abnormal, NCS | 18 | 11 | 7 | 10
  Week 0: Right eye ophthalmoscopy: Abnormal, CS | 1 | 0 | 0 | 0
  Week 54: Right eye ophthalmoscopy: number analyzed (Participants) | 68 | 63 | 69 | 64
  Week 54: Right eye ophthalmoscopy: Normal | 55 | 55 | 60 | 55
  Week 54: Right eye ophthalmoscopy: Abnormal, NCS | 13 | 8 | 9 | 8
  Week 54: Right eye ophthalmoscopy: Abnormal, CS | 0 | 0 | 0 | 1
  Week 80: Right eye ophthalmoscopy: number analyzed (Participants) | 66 | 62 | 65 | 59
  Week 80: Right eye ophthalmoscopy: Normal | 52 | 53 | 58 | 51
  Week 80: Right eye ophthalmoscopy: Abnormal, NCS | 12 | 9 | 7 | 8
  Week 80: Right eye ophthalmoscopy: Abnormal, CS | 2 | 0 | 0 | 0

72. Secondary Outcome: Change in Physical Examination
Description: Physical examination parameters are categorised as general appearance; head, ears, eyes, nose, throat, neck; respiratory system;cardiovascular system; gastrointestinal system including mouth; musculoskeletal system; central and peripheral nervous system; skin; lymph node palpation and thyroid gland. Investigator assessed the participants with normal, abnormal not clinically significant (NCS) and abnormal clinically significant (CS) findings at week 0, week 54 and week 80 are presented.
Time Frame: Week 0, week 54 and week 80
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Participants
  Week 0: General Appearance: Normal | 76 | 77 | 76 | 76
  Week 0: General Appearance: Abnormal, NCS | 1 | 0 | 0 | 1
  Week 0: General Appearance: Abnormal, CS | 0 | 0 | 0 | 0
  Week 54: General Appearance: number analyzed (Participants) | 68 | 65 | 66 | 66
  Week 54: General Appearance: Normal | 68 | 64 | 66 | 65
  Week 54: General Appearance: Abnormal, NCS | 0 | 0 | 0 | 1
  Week 54: General Appearance: Abnormal, CS | 0 | 1 | 0 | 0
  Week 80: General Appearance: number analyzed (Participants) | 67 | 64 | 68 | 62
  Week 80: General Appearance: Normal | 67 | 64 | 68 | 61
  Week 80: General Appearance: Abnormal, NCS | 0 | 0 | 0 | 1
  Week 80: General Appearance: Abnormal, CS | 0 | 0 | 0 | 0
  Week 0: Head, Ears, Eyes, Nose, Throat, Neck: Normal | 75 | 77 | 76 | 76
  Week 0: Head, Ears, Eyes, Nose, Throat, Neck: Abnormal, NCS | 2 | 0 | 0 | 1
  Week 0: Head, Ears, Eyes, Nose, Throat, Neck: Abnormal, CS | 0 | 0 | 0 | 0
  Week 54: Head, Ears, Eyes, Nose, Throat, Neck: number analyzed (Participants) | 68 | 65 | 66 | 66
  Week 54: Head, Ears, Eyes, Nose, Throat, Neck: Normal | 66 | 65 | 66 | 66
  Week 54: Head, Ears, Eyes, Nose, Throat, Neck: Abnormal, NCS | 1 | 0 | 0 | 0
  Week 54: Head, Ears, Eyes, Nose, Throat, Neck: Abnormal, CS | 1 | 0 | 0 | 0
  Week 80: Head, Ears, Eyes, Nose, Throat, Neck: number analyzed (Participants) | 67 | 64 | 68 | 62
  Week 80: Head, Ears, Eyes, Nose, Throat, Neck: Normal | 65 | 64 | 66 | 60
  Week 80: Head, Ears, Eyes, Nose, Throat, Neck: Abnormal, NCS | 2 | 0 | 2 | 2
  Week 80: Head, Ears, Eyes, Nose, Throat, Neck: Abnormal, CS | 0 | 0 | 0 | 0
  Week 0: Respiratory System: Normal | 77 | 77 | 76 | 77
  Week 0: Respiratory System: Abnormal, NCS | 0 | 0 | 0 | 0
  Week 0: Respiratory System: Abnormal, CS | 0 | 0 | 0 | 0
  Week 54: Respiratory System: number analyzed (Participants) | 68 | 65 | 66 | 66
  Week 54: Respiratory System: Normal | 68 | 65 | 66 | 66
  Week 54: Respiratory System: Abnormal, NCS | 0 | 0 | 0 | 0
  Week 54: Respiratory System: Abnormal, CS | 0 | 0 | 0 | 0
  Week 80: Respiratory System: number analyzed (Participants) | 67 | 64 | 68 | 62
  Week 80: Respiratory System: Normal | 67 | 64 | 68 | 61
  Week 80: Respiratory System: Abnormal, NCS | 0 | 0 | 0 | 1
  Week 80: Respiratory System: Abnormal, CS | 0 | 0 | 0 | 0
  Week 0: Cardiovascular System: Normal | 74 | 76 | 76 | 73
  Week 0: Cardiovascular System: Abnormal, NCS | 3 | 1 | 0 | 4
  Week 0: Cardiovascular System: Abnormal, CS | 0 | 0 | 0 | 0
  Week 54: Cardiovascular System: number analyzed (Participants) | 68 | 65 | 66 | 66
  Week 54: Cardiovascular System: Normal | 67 | 65 | 65 | 66
  Week 54: Cardiovascular System: Abnormal, NCS | 1 | 0 | 1 | 0
  Week 54: Cardiovascular System: Abnormal, CS | 0 | 0 | 0 | 0
  Week 80: Cardiovascular System: number analyzed (Participants) | 67 | 64 | 68 | 62
  Week 80: Cardiovascular System: Normal | 67 | 64 | 67 | 62
  Week 80: Cardiovascular System: Abnormal, NCS | 0 | 0 | 1 | 0
  Week 80: Cardiovascular System: Abnormal, CS | 0 | 0 | 0 | 0
  Week 0: Gastrointestinal System incl. Mouth: Normal | 75 | 76 | 76 | 76
  Week 0: Gastrointestinal System incl. Mouth: Abnormal, NCS | 2 | 1 | 0 | 1
  Week 0: Gastrointestinal System incl. Mouth: Abnormal, CS | 0 | 0 | 0 | 0
  Week 54: Gastrointestinal System incl. Mouth: number analyzed (Participants) | 68 | 65 | 66 | 66
  Week 54: Gastrointestinal System incl. Mouth: Normal | 68 | 64 | 66 | 65
  Week 54: Gastrointestinal System incl. Mouth: Abnormal, NCS | 0 | 1 | 0 | 1
  Week 54: Gastrointestinal System incl. Mouth: Abnormal, CS | 0 | 0 | 0 | 0
  Week 80: Gastrointestinal System incl. Mouth: number analyzed (Participants) | 67 | 64 | 68 | 62
  Week 80: Gastrointestinal System incl. Mouth: Normal | 67 | 63 | 68 | 61
  Week 80: Gastrointestinal System incl. Mouth: Abnormal, NCS | 0 | 1 | 0 | 1
  Week 80: Gastrointestinal System incl. Mouth: Abnormal, CS | 0 | 0 | 0 | 0
  Week 0: Musculoskeletal System: Normal | 76 | 75 | 74 | 77
  Week 0: Musculoskeletal System: Abnormal, NCS | 1 | 2 | 2 | 0
  Week 0: Musculoskeletal System: Abnormal, CS | 0 | 0 | 0 | 0
  Week 54: Musculoskeletal System: number analyzed (Participants) | 68 | 65 | 66 | 66
  Week 54: Musculoskeletal System: Normal | 65 | 63 | 66 | 65
  Week 54: Musculoskeletal System: Abnormal, NCS | 1 | 2 | 0 | 1
  Week 54: Musculoskeletal System: Abnormal, CS | 2 | 0 | 0 | 0
  Week 80: Musculoskeletal System: number analyzed (Participants) | 67 | 64 | 68 | 62
  Week 80: Musculoskeletal System: Normal | 66 | 64 | 68 | 62
  Week 80: Musculoskeletal System: Abnormal, NCS | 1 | 0 | 0 | 0
  Week 80: Musculoskeletal System: Abnormal, CS | 0 | 0 | 0 | 0
  Week 0: Central and Peripheral Nervous System: Normal | 77 | 76 | 76 | 76
  Week 0: Central and Peripheral Nervous System: Abnormal, NCS | 0 | 1 | 0 | 1
  Week 0: Central and Peripheral Nervous System: Abnormal, CS | 0 | 0 | 0 | 0
  Week 54: Central and Peripheral Nervous System: number analyzed (Participants) | 68 | 65 | 66 | 66
  Week 54: Central and Peripheral Nervous System: Normal | 68 | 64 | 66 | 65
  Week 54: Central and Peripheral Nervous System: Abnormal, NCS | 0 | 1 | 0 | 1
  Week 54: Central and Peripheral Nervous System: Abnormal, CS | 0 | 0 | 0 | 0
  Week 80: Central and Peripheral Nervous System: number analyzed (Participants) | 67 | 64 | 68 | 62
  Week 80: Central and Peripheral Nervous System: Normal | 66 | 63 | 68 | 62
  Week 80: Central and Peripheral Nervous System: Abnormal, NCS | 1 | 1 | 0 | 0
  Week 80: Central and Peripheral Nervous System: Abnormal, CS | 0 | 0 | 0 | 0
  Week 0: Skin: Normal | 70 | 75 | 69 | 74
  Week 0: Skin: Abnormal, NCS | 6 | 2 | 7 | 3
  Week 0: Skin: Abnormal, CS | 1 | 0 | 0 | 0
  Week 54: Skin: number analyzed (Participants) | 68 | 65 | 66 | 66
  Week 54: Skin: Normal | 61 | 63 | 63 | 66
  Week 54: Skin: Abnormal, NCS | 5 | 1 | 3 | 0
  Week 54: Skin: Abnormal, CS | 2 | 1 | 0 | 0
  Week 80: Skin: number analyzed (Participants) | 67 | 64 | 68 | 62
  Week 80: Skin: Normal | 61 | 62 | 65 | 62
  Week 80: Skin: Abnormal, NCS | 6 | 2 | 3 | 0
  Week 80: Skin: Abnormal, CS | 0 | 0 | 0 | 0
  Week 0: Lymph Node Palpation: Normal | 77 | 76 | 76 | 77
  Week 0: Lymph Node Palpation: Abnormal, NCS | 0 | 1 | 0 | 0
  Week 0: Lymph Node Palpation: Abnormal, CS | 0 | 0 | 0 | 0
  Week 54: Lymph Node Palpation: number analyzed (Participants) | 68 | 65 | 66 | 65
  Week 54: Lymph Node Palpation: Normal | 68 | 65 | 66 | 64
  Week 54: Lymph Node Palpation: Abnormal, NCS | 0 | 0 | 0 | 1
  Week 54: Lymph Node Palpation: Abnormal, CS | 0 | 0 | 0 | 0
  Week 80: Lymph Node Palpation: number analyzed (Participants) | 67 | 63 | 68 | 62
  Week 80: Lymph Node Palpation: Normal | 67 | 63 | 67 | 62
  Week 80: Lymph Node Palpation: Abnormal, NCS | 0 | 0 | 1 | 0
  Week 80: Lymph Node Palpation: Abnormal, CS | 0 | 0 | 0 | 0
  Week 0: Thyroid Gland: Normal | 77 | 76 | 76 | 75
  Week 0: Thyroid Gland: Abnormal, NCS | 0 | 1 | 0 | 2
  Week 0: Thyroid Gland: Abnormal, CS | 0 | 0 | 0 | 0
  Week 54: Thyroid Gland: number analyzed (Participants) | 68 | 65 | 66 | 65
  Week 54: Thyroid Gland: Normal | 67 | 65 | 66 | 65
  Week 54: Thyroid Gland: Abnormal, NCS | 1 | 0 | 0 | 0
  Week 54: Thyroid Gland: Abnormal, CS | 0 | 0 | 0 | 0
  Week 80: Thyroid Gland: number analyzed (Participants) | 67 | 64 | 68 | 62
  Week 80: Thyroid Gland: Normal | 67 | 64 | 68 | 62
  Week 80: Thyroid Gland: Abnormal, NCS | 0 | 0 | 0 | 0
  Week 80: Thyroid Gland: Abnormal, CS | 0 | 0 | 0 | 0

73. Secondary Outcome: Occurrence of Anti-NNC0114-0006 Antibodies
Description: This outcome measure was applicable for NNC0114-0006 + Liraglutide treatment arm and NNC0114-0006 treatment arm. Participants was assessed for anti-NNC0114-0006 antibodies. Participant who reported anti-NNC0114-0006 antibodies were further analyzed for cross-reactivity. Number of participants who measured with anti-NNC0114-0006 antibodies at week 54 and week 80 are presented.
Time Frame: Week 0, week 54 and week 80
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental)
Number analyzed (Participants) | 77 | 77
Participants
  Week 0: Anti-NNC0114-0006 antibodies: number analyzed (Participants) | 77 | 76
  Week 0: Anti-NNC0114-0006 antibodies: Negative | 68 | 62
  Week 0: Anti-NNC0114-0006 antibodies: Positive | 9 | 14
  Week 0: Cross-reactivity: number analyzed (Participants) | 9 | 14
  Week 0: Cross-reactivity: Negative | 4 | 7
  Week 0: Cross-reactivity: Positive | 5 | 7
  Week 54: Anti-NNC0114-0006: number analyzed (Participants) | 68 | 65
  Week 54: Anti-NNC0114-0006: Negative | 68 | 62
  Week 54: Anti-NNC0114-0006: Positive | 0 | 3
  Week 54: Cross-reactivity: number analyzed (Participants) | 0 | 3
  Week 54: Cross-reactivity: Negative | 0 | 3
  Week 54: Cross-reactivity: Positive | 0 | 0
  Week 80: Anti-NNC0114-0006 antibodies: number analyzed (Participants) | 67 | 64
  Week 80: Anti-NNC0114-0006 antibodies: Negative | 65 | 60
  Week 80: Anti-NNC0114-0006 antibodies: Positive | 2 | 4
  Week 80: Cross-reactivity: number analyzed (Participants) | 2 | 4
  Week 80: Cross-reactivity: Negative | 1 | 2
  Week 80: Cross-reactivity: Positive | 1 | 2

74. Secondary Outcome: Occurrence of Anti-liraglutide Antibodies
Description: This outcome measure is applicable for NNC0114-0006 + Liraglutide treatment arm and Liraglutide treatment arm. Participants was assessed for anti-liraglutide antibodies. Participant who reported anti-liraglutide antibodies were further analyzed for cross-reactivity. Number of participants who measured with anti-liraglutide antibodies at week 54 and week 80 are presented.
Time Frame: Week 0, week 54 and week 80
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | Liraglutide (Experimental)
Number analyzed (Participants) | 77 | 76
Participants
  Week 0: Anti-Liraglutide antibodies: number analyzed (Participants) | 77 | 75
  Week 0: Anti-Liraglutide antibodies: Negative | 77 | 75
  Week 0: Anti-Liraglutide antibodies: Positive | 0 | 0
  Week 0: Cross-reactivity to native GLP-1: number analyzed (Participants) | 0 | 0
  Week 0: Cross-reactivity to native GLP-1: Negative | 0 | 0
  Week 0: Cross-reactivity to native GLP-1: Positive | 0 | 0
  Week 54: Anti-Liraglutide antibodies: number analyzed (Participants) | 68 | 67
  Week 54: Anti-Liraglutide antibodies: Negative | 67 | 65
  Week 54: Anti-Liraglutide antibodies: Positive | 1 | 2
  Week 54: Cross-reactivity to native GLP-1: number analyzed (Participants) | 1 | 2
  Week 54: Cross-reactivity to native GLP-1: Negative | 1 | 1
  Week 54: Cross-reactivity to native GLP-1: Positive | 0 | 1
  Week 80: Anti-Liraglutide antibodies: number analyzed (Participants) | 67 | 68
  Week 80: Anti-Liraglutide antibodies: Negative | 67 | 66
  Week 80: Anti-Liraglutide antibodies: Positive | 0 | 2
  Week 80: Cross-reactivity to native GLP-1: number analyzed (Participants) | 0 | 0
  Week 80: Cross-reactivity to native GLP-1: Negative | 0 | 0
  Week 80: Cross-reactivity to native GLP-1: Positive | 0 | 0

75. Secondary Outcome: Change in Insulin Dose
Description: The total daily insulin dose was derived as the average of the doses reported on the three days prior to the visit. Change in daily total insulin dose from baseline (week 0) after 54 weeks of treatment and week 80 are presented.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: The FAS included all randomised participants. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Units per kilograms
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Units per kilograms
  Change from week 0 to week 54: number analyzed (Participants) | 49 | 52 | 55 | 49
  Change from week 0 to week 54 | -0.05 (0.18) | 0.02 (0.18) | 0.01 (0.23) | 0.09 (0.19)
  Change from week 0 to week 80: number analyzed (Participants) | 46 | 53 | 50 | 43
  Change from week 0 to week 80 | 0.10 (0.20) | 0.05 (0.19) | 0.11 (0.22) | 0.12 (0.18)

76. Secondary Outcome: Change in Number of Insulin Injections
Description: The number of insulin injections was derived as the average of the reported number on the three days prior to the visit. The change in number of insulin injections per day (count) from baseline (week 0) after 54 weeks of treatment and week 80 are presented.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: The FAS included all randomised participants. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Injections per day
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Injections per day
  Change from week 0 to week 54: number analyzed (Participants) | 49 | 52 | 55 | 49
  Change from week 0 to week 54 | -0.3 (1.5) | -0.1 (1.2) | -0.5 (1.7) | 0.2 (1.4)
  Change from week 0 to week 80: number analyzed (Participants) | 46 | 53 | 50 | 43
  Change from week 0 to week 80 | 0.2 (1.5) | -0.3 (1.3) | -0.2 (1.5) | 0.2 (1.3)

77. Secondary Outcome: Number of Weeks Off Bolus Insulin
Description: The number of weeks off bolus insulin after 54 weeks of treatment and week 80 are presented.
Time Frame: (Week 0 to week 54) and (week 0 to week 80)
Population: The FAS included all randomised participants. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Weeks
  Week 0 to week 54: number analyzed (Participants) | 62 | 55 | 56 | 58
  Week 0 to week 54 | 10 (18) | 5 (14) | 9 (18) | 4 (11)
  Week 0 to week 80: number analyzed (Participants) | 54 | 52 | 52 | 51
  Week 0 to week 80 | 14 (25) | 9 (20) | 12 (24) | 6 (14)

78. Secondary Outcome: Change in HbA1c
Description: Change in glycosylated haemoglobin (HbA1c) is evaluated from baseline (week 0) to weeks 54 and 80.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: The FAS included all randomised participants. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage point of HbA1c
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Percentage point of HbA1c
  Change from week 0 to week 54: number analyzed (Participants) | 68 | 65 | 67 | 65
  Change from week 0 to week 54 | -0.7 (1.9) | -0.5 (1.4) | -0.3 (1.5) | -0.3 (1.9)
  Change from week 0 to week 80: number analyzed (Participants) | 66 | 64 | 68 | 62
  Change from week 0 to week 80 | -0.1 (1.6) | -0.2 (1.5) | 0.5 (2.1) | -0.4 (1.8)

79. Secondary Outcome: Change in Fasting Plasma Glucose
Description: Change in fasting plasma glucose is evaluated from baseline (week 0) to weeks 54 and 80.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: The FAS included all randomised participants. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
mmol/L
  Change from week 0 to week 54: number analyzed (Participants) | 66 | 64 | 66 | 64
  Change from week 0 to week 54 | 0.5 (3.2) | 0.2 (2.4) | -0.3 (3.1) | 0.5 (2.4)
  Change from week 0 to week 80: number analyzed (Participants) | 62 | 61 | 65 | 60
  Change from week 0 to week 80 | 1.1 (3.3) | 0.3 (2.4) | 0.2 (4.0) | 1.0 (2.4)

80. Secondary Outcome: Change in Fasting C-peptide- Ratio to Baseline
Description: Change in fasting C-peptide (measured in nanomole per liter [nmol/L]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: The FAS included all randomised participants. Number analyzed = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of C-peptide
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of C-peptide
  Ratio from week 0 to week 54: number analyzed (Participants) | 68 | 64 | 66 | 64
  Ratio from week 0 to week 54 | 1.01 (76.8) | 0.70 (71.1) | 0.65 (102.4) | 0.66 (116.3)
  Ratio from week 0 to week 80: number analyzed (Participants) | 65 | 63 | 64 | 60
  Ratio from week 0 to week 80 | 0.58 (112.9) | 0.53 (106.2) | 0.42 (132.5) | 0.54 (154.4)

81. Secondary Outcome: Change in Fasting Glucagon- Ratio to Baseline
Description: Change in fasting glucagon (measured in picogram per milliliter [pg/mL]) from baseline (week 0) to weeks 54 and 80 is presented as ratio to baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: The FAS included all randomised participants. Number analyzed = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of glucagon
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Ratio of glucagon
  Ratio from week 0 to week 54: number analyzed (Participants) | 67 | 64 | 68 | 66
  Ratio from week 0 to week 54 | 1.01 (32.1) | 0.95 (32.5) | 0.96 (31.3) | 1.00 (31.4)
  Ratio from week 0 to week 80: number analyzed (Participants) | 66 | 63 | 67 | 61
  Ratio from week 0 to week 80 | 0.89 (36.2) | 0.85 (30.7) | 0.96 (32.8) | 0.93 (37.8)

82. Secondary Outcome: 7-point SMPG Profiles
Description: Participants measured plasma glucose values using the blood glucose meter at 7 time points: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner, bedtime. 7-point SMPG profile values are presented for week 54 and week 80.
Time Frame: Week 54 and Week 80
Population: The FAS included all randomised participants. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
mmol/L
  Week 54: Before breakfast: number analyzed (Participants) | 51 | 51 | 57 | 45
  Week 54: Before breakfast | 6.8 (3.4) | 6.8 (2.7) | 6.4 (2.2) | 6.3 (1.4)
  Week 54: 90 minutes after start of breakfast: number analyzed (Participants) | 47 | 46 | 53 | 39
  Week 54: 90 minutes after start of breakfast | 8.9 (3.7) | 7.5 (2.4) | 7.4 (2.1) | 7.6 (2.4)
  Week 54: Before lunch: number analyzed (Participants) | 52 | 51 | 58 | 46
  Week 54: Before lunch | 5.5 (1.8) | 6.4 (2.3) | 6.1 (1.8) | 6.0 (1.6)
  Week 54: 90 minutes after start of lunch: number analyzed (Participants) | 47 | 47 | 54 | 39
  Week 54: 90 minutes after start of lunch | 8.2 (2.6) | 7.5 (2.7) | 7.8 (2.4) | 7.7 (2.0)
  Week 54: Before dinner: number analyzed (Participants) | 52 | 48 | 56 | 47
  Week 54: Before dinner | 6.5 (1.9) | 6.5 (2.5) | 6.6 (2.2) | 6.1 (1.7)
  Week 54: 90 minutes after start of dinner: number analyzed (Participants) | 44 | 43 | 50 | 35
  Week 54: 90 minutes after start of dinner | 8.2 (3.4) | 7.0 (2.5) | 7.2 (2.3) | 6.8 (1.9)
  Week 54: Bedtime: number analyzed (Participants) | 52 | 49 | 56 | 43
  Week 54: Bedtime | 7.8 (3.9) | 7.4 (2.6) | 7.5 (2.5) | 7.2 (2.1)
  Week 80: Before breakfast: number analyzed (Participants) | 46 | 46 | 41 | 44
  Week 80: Before breakfast | 6.5 (1.7) | 6.4 (2.0) | 7.2 (2.7) | 6.8 (2.0)
  Week 80: 90 minutes after start of breakfast: number analyzed (Participants) | 43 | 43 | 36 | 40
  Week 80: 90 minutes after start of breakfast | 8.5 (2.8) | 7.2 (3.0) | 8.3 (3.7) | 7.5 (2.7)
  Week 80: Before lunch: number analyzed (Participants) | 44 | 46 | 39 | 45
  Week 80: Before lunch | 6.2 (2.2) | 6.2 (2.0) | 6.9 (3.3) | 6.1 (1.8)
  Week 80: 90 minutes after start of lunch: number analyzed (Participants) | 43 | 43 | 35 | 40
  Week 80: 90 minutes after start of lunch | 7.8 (2.6) | 7.6 (2.7) | 8.5 (4.5) | 8.0 (3.0)
  Week 80: Before dinner: number analyzed (Participants) | 44 | 45 | 41 | 45
  Week 80: Before dinner | 6.5 (2.2) | 6.7 (2.9) | 7.6 (4.1) | 6.5 (1.6)
  Week 80: 90 minutes after start of dinner: number analyzed (Participants) | 41 | 42 | 34 | 40
  Week 80: 90 minutes after start of dinner | 7.6 (2.5) | 7.0 (2.1) | 9.0 (5.0) | 7.6 (2.5)
  Week 80: Bedtime: number analyzed (Participants) | 38 | 44 | 38 | 41
  Week 80: Bedtime | 7.8 (3.0) | 6.6 (1.8) | 7.8 (4.4) | 7.4 (2.2)

83. Secondary Outcome: Change in 7- Points Self-measured Plasma Glucose (SMPG) Postprandial Glucose /Prandial Increment: Breakfast, Lunch, Dinner
Description: Participants measured plasma glucose values using the blood glucose meter at 7 time points: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner and at bedtime. Change from baseline (week 0) to week 54 and week 80 in 7-point SMPG postprandial glucose /prandial increment (breakfast, lunch and dinner) value are presented.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: The FAS included all randomised participants. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
mmol/L
  Change from week 0 to week 54: Breakfast: number analyzed (Participants) | 29 | 29 | 28 | 21
  Change from week 0 to week 54: Breakfast | 1.3 (4.0) | 0.4 (3.0) | -0.1 (3.8) | -0.6 (2.4)
  Change from week 0 to week 80: Breakfast: number analyzed (Participants) | 26 | 28 | 20 | 19
  Change from week 0 to week 80: Breakfast | 1.9 (4.2) | 0.5 (4.0) | -0.1 (4.5) | -0.5 (4.5)
  Change from week 0 to week 54: Lunch: number analyzed (Participants) | 31 | 32 | 28 | 22
  Change from week 0 to week 54: Lunch | 0.9 (4.5) | 0.5 (3.4) | 1.5 (2.9) | 0.7 (2.7)
  Change from week 0 to week 80: Lunch: number analyzed (Participants) | 29 | 30 | 19 | 20
  Change from week 0 to week 80: Lunch | 0.0 (4.5) | 0.1 (3.0) | 1.0 (3.5) | 0.8 (4.5)
  Change from week 0 to week 54: Dinner: number analyzed (Participants) | 28 | 27 | 22 | 18
  Change from week 0 to week 54: Dinner | 0.1 (4.5) | 1.1 (4.0) | -0.8 (4.7) | -0.3 (3.1)
  Change from week 0 to week 80: Dinner: number analyzed (Participants) | 25 | 26 | 15 | 19
  Change from week 0 to week 80: Dinner | 0.5 (5.0) | 0.5 (3.4) | -0.4 (4.3) | -0.4 (3.2)

84. Secondary Outcome: Change in 7- Points Self-measured Plasma Glucose (SMPG) Postprandial Glucose /Prandial Increment (Average Over the Three Meals)
Description: Participants measured plasma glucose values using the blood glucose meter at 7 time points: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner, bedtime. Change from baseline (week 0) to week 54 and week 80 in 7-point self-measured plasma glucose (SMPG) postprandial glucose /prandial increment (average over the three meals) value is presented.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: The FAS included all randomised participants. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
mmol/L
  Change from week 0 to week 54: number analyzed (Participants) | 32 | 33 | 29 | 22
  Change from week 0 to week 54 | 0.9 (2.3) | 0.6 (2.2) | 0.2 (2.0) | -0.1 (2.0)
  Change from week 0 to week 80: number analyzed (Participants) | 30 | 31 | 20 | 21
  Change from week 0 to week 80 | 0.8 (2.6) | 0.4 (2.2) | 0.0 (2.5) | -0.0 (2.9)

85. Secondary Outcome: Change in Mean of 7-point Profiles
Description: Participants measured plasma glucose values using the blood glucose meter at 7 time points: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner, bedtime. Change from baseline (week 0) to week 54 and week 80 in mean of 7-point profiles value is presented.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: The FAS included all randomised participants. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
mmol/L
  Change from week 0 to week 54: number analyzed (Participants) | 36 | 40 | 34 | 28
  Change from week 0 to week 54 | 0.5 (2.0) | 0.3 (2.4) | -0.1 (1.9) | 0.0 (1.2)
  Change from week 0 to week 80: number analyzed (Participants) | 34 | 36 | 26 | 27
  Change from week 0 to week 80 | 0.1 (2.1) | 0.0 (2.3) | 0.7 (1.6) | 0.3 (1.7)

86. Secondary Outcome: Before Breakfast 7- Points Self Measured Plasma Glucose (SMPG)
Description: Participants measured plasma glucose values using the blood glucose meter at 7 time points: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner and at bedtime. Before breakfast 7-point self-measured plasma glucose (SMPG) profile values are presented at week 54 and week 80.
Time Frame: Week 54 and week 80
Population: The FAS included all randomised participants. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
mmol/L
  Week 54: number analyzed (Participants) | 51 | 51 | 57 | 45
  Week 54 | 6.8 (3.4) | 6.8 (2.7) | 6.4 (2.2) | 6.3 (1.4)
  Week 80: number analyzed (Participants) | 46 | 46 | 41 | 44
  Week 80 | 6.5 (1.7) | 6.4 (2.0) | 7.2 (2.7) | 6.8 (2.0)

87. Secondary Outcome: Area Under the NNC0114-0006 Concentration-time Curve Over a Dosing Interval at Steady State (AUCtau, NNC0114-0006)
Description: AUCtau, NNC0114-0006 was derived as the area under the concentration-time curve using the linear trapezoidal technique based on observed values and actual measurement times between 0 and 6 weeks (after the last dose). This outcome measure was applicable for NNC0114-0006 + Liraglutide and NNC0114-0006 treatment arms.
Time Frame: Pre-dose and 1 hour post-dose during week 48 to week 54
Population: The PK analysis set comprised all randomized participants with at least one valid PK measurement. Overall number of participants analyzed = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*microgram per milliliter (day*ug/mL)
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental)
Number analyzed (Participants) | 17 | 16
day*microgram per milliliter (day*ug/mL) | 3969 (17.9) | 4115 (23.1)

88. Secondary Outcome: Terminal Half-life (t½) After Last Dose of NNC0114-0006
Description: Terminal half life was calculated as log(2)/λz. The terminal rate constant λz was determined through linear regression with the logarithm to concentration as the response variable and actual measurement time as the explanatory variable. Valid observations from the terminal part of the curve, which is approximately linear, were used for the determination. This outcome measure was applicable for NNC0114-0006 + Liraglutide and NNC0114-0006 treatment arms.
Time Frame: Pre-dose and 1 hour post-dose during week 48 to week 80
Population: as for outcome 87
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental)
Number analyzed (Participants) | 17 | 16
Days | 22.3 (17.9) | 22.2 (16.5)

89. Secondary Outcome: Apparent Volume of Distribution of NNC0114-0006 at Steadystate (Vss, NNC0114-0006)
Description: The apparent volume of distribution of NNC0114-0006 at steady-state was calculated as mean residence time of (MRT) of NNC0114-0006 multiplied by clearance of NNC0114-0006 at steady state. This outcome measure was applicable for NNC0114-0006 + Liraglutide and NNC0114-0006 treatment arms.
Time Frame: Pre-dose and 1 hour post-dose during week 48 to week 80
Population: as for outcome 87
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliters per kilogram (mL/kg)
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental)
Number analyzed (Participants) | 17 | 16
Milliliters per kilogram (mL/kg) | 83.7 (23.1) | 79.3 (17.6)

90. Secondary Outcome: Clearance of NNC0114-0006 at Steady State (CLss, NNC0114-0006)
Description: Clearance of NNC0114-0006 at steady state was calculated as dose/AUCtau, NNC0114-0006. This outcome measure was applicable for NNC0114-0006 + Liraglutide and NNC0114-0006 treatment arms.
Time Frame: Pre-dose and 1 hour post-dose during week 48 to week 54
Population: as for outcome 87
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (Milliliters/day)/kilogram ([mL/day]/kg)
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental)
Number analyzed (Participants) | 17 | 16
(Milliliters/day)/kilogram ([mL/day]/kg) | 3.02 (17.9) | 2.92 (23.1)

91. Secondary Outcome: Mean Residence Time of NNC0114-0006 (MRT, NNC0114-0006)
Description: This outcome measure was applicable for NNC0114-0006 + Liraglutide and NNC0114-0006 treatment arms. Mean residence time of NNC0114-0006 is presented.
Time Frame: Pre-dose and 1 hour post-dose during week 48 to week 80
Population: as for outcome 87
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental)
Number analyzed (Participants) | 17 | 16
Days | 27.7 (24.5) | 27.2 (22.6)

92. Secondary Outcome: Accumulation Ratio of NNC114-0006 (RA,AUC, NNC0114-0006)
Description: Accumulation ratio of NNC114-0006 was defined as AUC48-54 weeks/AUC0-6 weeks. This outcome measure was applicable for NNC0114-0006 + Liraglutide and NNC0114-0006 treatment arms.
Time Frame: Pre-dose and 1 hour post-dose during (week 0 to week 6) and (week 48 to week 54)
Population: as for outcome 87
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AUC
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental)
Number analyzed (Participants) | 16 | 16
Ratio of AUC | 1.24 (17.8) | 1.26 (17.4)

93. Secondary Outcome: Observed NNC0114-0006 Concentration Prior to Dosing of NNC0114-0006 at Steady State (Ctrough, NNC0114-0006)
Description: Ctrough of NNC0114-0006 was defined as concentration prior to dosing of NNC0114-0006 at steady state. This outcome measure was applicable for NNC0114-0006 + Liraglutide and NNC0114-0006 treatment arms.
Time Frame: Week 48 (predose)
Population: as for outcome 87
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (ug/mL)
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental)
Number analyzed (Participants) | 17 | 16
microgram/milliliter (ug/mL) | 34.7 (42.3) | 36.7 (36.8)

94. Secondary Outcome: Observed NNC0114-0006 Concentration 1 Hour After Dosing of NNC0114-0006 at Steady State (C1h, NNC0114-0006)
Description: C1h, NNC0114-0006 was defined as concentration of NNC0114-0006 at 1 hour after dosing of NNC0114-0006 at steady state. This outcome measure was applicable for NNC0114-0006 + Liraglutide and NNC0114-0006 treatment arms.
Time Frame: Week 48 (1 hour post-dose)
Population: as for outcome 87
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental)
Number analyzed (Participants) | 14 | 15
ug/mL | 298.6 (16.8) | 282.6 (56.4)

95. Secondary Outcome: Liraglutide Concentration at Steady State (C Liraglutide)
Description: C liraglutide was defined as the liraglutide concentration at steady state. This outcome measure was applicable for NNC0114-0006 + Liraglutide and Liraglutide treatment arms.
Time Frame: Week 54 (post-dose)
Population: as for outcome 87
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole per liter (pmol/L)
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | Liraglutide (Experimental)
Number analyzed (Participants) | 17 | 19
picomole per liter (pmol/L) | 16287 (41.7) | 15920 (66.0)

96. Secondary Outcome: Change in Biomarker: Immune Phenotyping- B Cell Panel
Description: B cell panel is evaluated by Immune phenotyping of peripheral blood mononuclear cells (PBMC) at baseline (week 0), week 54 and week 80.
  In below table CD refer to Cluster of Differentiation; IgMNeg refers to Immunoglobulin M negative; IgDNeg refers to Immunoglobulin D negative.
Time Frame: Week 0, week 54 and week 80
Population: The FAS included all randomised participants. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of B cells (%)
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Percentage of B cells (%)
  Week 0: Activated Memory B-Cells: number analyzed (Participants) | 71 | 70 | 62 | 71
  Week 0: Activated Memory B-Cells | 1.3 (0.9) | 1.4 (1.0) | 1.6 (1.1) | 1.5 (1.0)
  Week 54: Activated Memory B-Cells: number analyzed (Participants) | 64 | 56 | 57 | 58
  Week 54: Activated Memory B-Cells | 1.2 (0.8) | 1.1 (1.0) | 1.5 (1.3) | 1.3 (0.8)
  Week 80: Activated Memory B-Cells: number analyzed (Participants) | 61 | 53 | 55 | 56
  Week 80: Activated Memory B-Cells | 1.2 (0.9) | 1.1 (0.7) | 1.5 (1.1) | 1.5 (1.2)
  Week 0: Mature Naive B-Cells: number analyzed (Participants) | 71 | 70 | 62 | 71
  Week 0: Mature Naive B-Cells | 15.1 (6.7) | 14.0 (7.1) | 13.6 (6.9) | 13.3 (7.4)
  Week 54: Mature Naive B-Cells: number analyzed (Participants) | 64 | 56 | 57 | 58
  Week 54: Mature Naive B-Cells | 14.0 (6.2) | 14.3 (7.9) | 13.6 (7.6) | 13.5 (6.9)
  Week 80: Mature Naive B-Cells: number analyzed (Participants) | 61 | 53 | 55 | 56
  Week 80: Mature Naive B-Cells | 14.3 (7.3) | 14.2 (8.7) | 12.0 (5.2) | 12.8 (7.6)
  Week 0: Antibody-Secreting Cells: number analyzed (Participants) | 71 | 70 | 62 | 71
  Week 0: Antibody-Secreting Cells | 0.6 (0.4) | 0.5 (0.5) | 0.6 (0.3) | 0.6 (0.6)
  Week 54: Antibody-Secreting Cells: number analyzed (Participants) | 64 | 56 | 57 | 58
  Week 54: Antibody-Secreting Cells | 0.6 (0.5) | 0.4 (0.4) | 0.5 (0.3) | 0.6 (0.7)
  Week 80: Antibody-Secreting Cells: number analyzed (Participants) | 61 | 53 | 55 | 56
  Week 80: Antibody-Secreting Cells | 0.5 (0.4) | 0.4 (0.3) | 0.4 (0.4) | 0.6 (0.5)
  Week 0: B-Cells Positive For Both CD19 & CD20: number analyzed (Participants) | 71 | 70 | 62 | 71
  Week 0: B-Cells Positive For Both CD19 & CD20 | 71.9 (9.7) | 71.1 (11.1) | 72.1 (8.9) | 72.2 (8.8)
  Week 54: B-Cells Positive For Both CD19 & CD20: number analyzed (Participants) | 64 | 56 | 57 | 58
  Week 54: B-Cells Positive For Both CD19 & CD20 | 71.1 (12.4) | 70.8 (12.4) | 72.1 (8.4) | 65.9 (13.6)
  Week 80: B-Cells Positive For Both CD19 & CD20: number analyzed (Participants) | 61 | 53 | 55 | 56
  Week 80: B-Cells Positive For Both CD19 & CD20 | 71.0 (10.7) | 69.8 (11.2) | 72.8 (10.6) | 69.6 (13.5)
  Week 0: CD20Neg B-Cell: number analyzed (Participants) | 71 | 70 | 62 | 71
  Week 0: CD20Neg B-Cell | 0.6 (0.5) | 0.6 (0.7) | 0.6 (0.7) | 0.6 (0.5)
  Week 54: CD20Neg B-Cell: number analyzed (Participants) | 64 | 56 | 57 | 58
  Week 54: CD20Neg B-Cell | 0.6 (0.7) | 0.5 (0.9) | 0.5 (0.4) | 0.6 (0.7)
  Week 80: CD20Neg B-Cell: number analyzed (Participants) | 61 | 53 | 55 | 56
  Week 80: CD20Neg B-Cell | 0.5 (0.3) | 0.5 (0.4) | 0.6 (1.8) | 0.7 (1.0)
  Week 0: CD24- B-Cells: number analyzed (Participants) | 71 | 70 | 62 | 71
  Week 0: CD24- B-Cells | 29.8 (10.2) | 31.0 (11.5) | 31.5 (11.8) | 32.0 (11.1)
  Week 54: CD24- B-Cells: number analyzed (Participants) | 64 | 56 | 57 | 58
  Week 54: CD24- B-Cells | 30.2 (9.4) | 30.6 (10.8) | 31.3 (11.9) | 28.3 (8.9)
  Week 80: CD24- B-Cells: number analyzed (Participants) | 61 | 53 | 55 | 56
  Week 80: CD24- B-Cells | 30.0 (8.9) | 31.6 (10.9) | 33.4 (12.4) | 30.7 (11.8)
  Week 0: Class-Switched Memory B Cells: number analyzed (Participants) | 71 | 70 | 62 | 71
  Week 0: Class-Switched Memory B Cells | 5.0 (3.3) | 4.6 (2.5) | 4.8 (3.3) | 4.9 (3.0)
  Week 54: Class-Switched Memory B Cells: number analyzed (Participants) | 64 | 56 | 57 | 58
  Week 54: Class-Switched Memory B Cells | 5.0 (3.7) | 4.2 (2.3) | 4.6 (2.9) | 4.8 (2.9)
  Week 80: Class-Switched Memory B Cells: number analyzed (Participants) | 61 | 53 | 55 | 56
  Week 80: Class-Switched Memory B Cells | 4.6 (3.3) | 3.6 (2.0) | 4.6 (3.0) | 4.5 (2.5)
  Week 0: IgMNeg IgDNeg Switched Memory B-cells: number analyzed (Participants) | 71 | 70 | 62 | 71
  Week 0: IgMNeg IgDNeg Switched Memory B-cells | 0.1 (0.1) | 0.1 (0.1) | 0.1 (0.1) | 0.1 (0.1)
  Week 54: IgMNeg IgDNeg Switched Memory B-cells: number analyzed (Participants) | 64 | 56 | 57 | 58
  Week 54: IgMNeg IgDNeg Switched Memory B-cells | 0.1 (0.1) | 0.1 (0.1) | 0.1 (0.2) | 0.1 (0.1)
  Week 80: IgMNeg IgDNeg Switched Memory B-cells: number analyzed (Participants) | 61 | 53 | 55 | 56
  Week 80: IgMNeg IgDNeg Switched Memory B-cells | 0.1 (0.1) | 0.2 (0.2) | 0.1 (0.1) | 0.1 (0.1)
  Week 0: Non-Class Switched Memory B-Cells: number analyzed (Participants) | 71 | 70 | 62 | 71
  Week 0: Non-Class Switched Memory B-Cells | 10.2 (6.4) | 9.6 (5.8) | 9.6 (5.8) | 10.1 (6.4)
  Week 54: Non-Class Switched Memory B-Cells: number analyzed (Participants) | 64 | 56 | 57 | 58
  Week 54: Non-Class Switched Memory B-Cells | 8.5 (4.8) | 9.0 (5.7) | 8.7 (5.8) | 8.9 (5.8)
  Week 80: Non-Class Switched Memory B-Cells: number analyzed (Participants) | 61 | 53 | 55 | 56
  Week 80: Non-Class Switched Memory B-Cells | 8.2 (4.9) | 7.2 (4.1) | 8.0 (5.1) | 8.9 (6.2)
  Week 0: Total B-Cell Population: number analyzed (Participants) | 71 | 70 | 62 | 71
  Week 0: Total B-Cell Population | 72.5 (9.8) | 71.7 (11.2) | 72.7 (9.0) | 72.8 (8.6)
  Week 54: Total B-Cell Population: number analyzed (Participants) | 64 | 56 | 57 | 58
  Week 54: Total B-Cell Population | 71.7 (12.1) | 71.3 (11.9) | 72.6 (8.4) | 66.5 (13.3)
  Week 80: Total B-Cell Population: number analyzed (Participants) | 61 | 53 | 55 | 56
  Week 80: Total B-Cell Population | 71.4 (10.7) | 70.3 (11.2) | 73.5 (9.6) | 70.4 (13.0)
  Week 0: Transitional B-Cells: number analyzed (Participants) | 71 | 70 | 62 | 71
  Week 0: Transitional B-Cells | 11.4 (6.1) | 9.9 (6.5) | 9.5 (5.5) | 9.6 (6.6)
  Week 54: Transitional B-Cells: number analyzed (Participants) | 64 | 56 | 57 | 58
  Week 54: Transitional B-Cells | 10.2 (5.6) | 10.7 (7.7) | 9.5 (6.3) | 9.8 (6.4)
  Week 80: Transitional B-Cells: number analyzed (Participants) | 61 | 53 | 55 | 56
  Week 80: Transitional B-Cells | 10.8 (6.8) | 10.5 (8.1) | 8.1 (4.0) | 8.9 (6.1)

97. Secondary Outcome: Change in Biomarker: Immune Phenotyping- Natural Killer (NK) Cell Panel
Description: NK cell panel is evaluated by Immune phenotyping of peripheral blood mononuclear cells (PBMC) at baseline (week 0), week 54 and week 80.
  In below table ADCC refer to Antibody-dependent cellular cytotoxicity; CD refer to Cluster of Differentiation.
Time Frame: Week 0, week 54 and week 80
Population: The FAS included all randomised participants. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of NK cells (%)
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Percentage of NK cells (%)
  Week 0: ADCC-Competent NK: number analyzed (Participants) | 71 | 65 | 65 | 68
  Week 0: ADCC-Competent NK | 39.5 (17.1) | 36.3 (14.9) | 36.0 (16.6) | 34.7 (14.6)
  Week 54: ADCC-Competent NK: number analyzed (Participants) | 60 | 53 | 53 | 53
  Week 54: ADCC-Competent NK | 37.1 (16.1) | 32.5 (14.1) | 33.9 (14.0) | 31.5 (14.0)
  Week 80: ADCC-Competent NK: number analyzed (Participants) | 59 | 44 | 52 | 50
  Week 80: ADCC-Competent NK | 37.1 (16.0) | 33.2 (13.7) | 31.9 (15.1) | 34.1 (16.3)
  Week 0: CD16+ Highly Functional NK Cells: number analyzed (Participants) | 71 | 65 | 65 | 68
  Week 0: CD16+ Highly Functional NK Cells | 0.8 (0.8) | 0.8 (0.7) | 0.7 (0.6) | 0.7 (0.6)
  Week 54: CD16+ Highly Functional NK Cells: number analyzed (Participants) | 60 | 53 | 53 | 53
  Week 54: CD16+ Highly Functional NK Cells | 0.7 (0.7) | 0.7 (0.8) | 0.7 (0.7) | 0.6 (0.5)
  Week 80: CD16+ Highly Functional NK Cells: number analyzed (Participants) | 59 | 44 | 52 | 50
  Week 80: CD16+ Highly Functional NK Cells | 0.7 (0.8) | 0.6 (0.5) | 0.6 (0.6) | 0.8 (0.7)
  Week 0: CD56- Cells: number analyzed (Participants) | 71 | 65 | 65 | 68
  Week 0: CD56- Cells | 34.5 (15.9) | 36.8 (15.5) | 38.0 (17.1) | 38.0 (13.6)
  Week 54: CD56- Cells: number analyzed (Participants) | 60 | 53 | 53 | 53
  Week 54: CD56- Cells | 34.8 (12.8) | 36.6 (12.9) | 38.1 (14.3) | 41.1 (15.7)
  Week 80: CD56- Cells: number analyzed (Participants) | 59 | 44 | 52 | 50
  Week 80: CD56- Cells | 36.2 (14.3) | 37.6 (13.7) | 37.1 (11.7) | 37.6 (12.7)
  Week 0: CD56High NK Pool: number analyzed (Participants) | 71 | 65 | 65 | 68
  Week 0: CD56High NK Pool | 4.9 (3.3) | 5.1 (3.5) | 4.5 (2.9) | 4.9 (3.7)
  Week 54: CD56High NK Pool: number analyzed (Participants) | 60 | 53 | 53 | 53
  Week 54: CD56High NK Pool | 4.9 (3.1) | 5.3 (3.4) | 4.2 (2.9) | 4.4 (3.0)
  Week 80: CD56High NK Pool: number analyzed (Participants) | 59 | 44 | 52 | 50
  Week 80: CD56High NK Pool | 4.5 (2.9) | 5.1 (3.1) | 4.3 (2.8) | 5.4 (4.0)
  Week 0: CD57+ MatNK Effectors: number analyzed (Participants) | 71 | 65 | 65 | 68
  Week 0: CD57+ MatNK Effectors | 22.6 (12.5) | 20.4 (10.3) | 21.0 (11.8) | 19.0 (10.1)
  Week 54: CD57+ MatNK Effectors: number analyzed (Participants) | 60 | 53 | 53 | 53
  Week 54: CD57+ MatNK Effectors | 21.0 (12.5) | 18.0 (10.1) | 18.9 (10.6) | 16.6 (9.4)
  Week 80: CD57+ MatNK Effectors: number analyzed (Participants) | 59 | 44 | 52 | 50
  Week 80: CD57+ MatNK Effectors | 20.0 (11.2) | 18.3 (9.0) | 17.5 (11.1) | 17.3 (9.6)
  Week 0: Functional NK Cells; Efficient At ADCC: number analyzed (Participants) | 71 | 65 | 65 | 68
  Week 0: Functional NK Cells; Efficient At ADCC | 14.5 (7.8) | 13.3 (8.5) | 13.1 (9.7) | 12.1 (6.4)
  Week 54: Functional NK Cells; Efficient At ADCC: number analyzed (Participants) | 60 | 53 | 53 | 53
  Week 54: Functional NK Cells; Efficient At ADCC | 13.2 (8.5) | 11.1 (7.2) | 12.1 (7.1) | 11.0 (7.2)
  Week 80: Functional NK Cells; Efficient At ADCC: number analyzed (Participants) | 59 | 44 | 52 | 50
  Week 80: Functional NK Cells; Efficient At ADCC | 13.3 (7.4) | 11.3 (7.1) | 10.9 (7.2) | 12.6 (9.4)
  Week 0: Highly Cytolytic Subset Of NK Cells: number analyzed (Participants) | 71 | 65 | 65 | 68
  Week 0: Highly Cytolytic Subset Of NK Cells | 18.8 (10.4) | 20.9 (10.3) | 20.6 (11.0) | 21.4 (9.4)
  Week 54: Highly Cytolytic Subset Of NK Cells: number analyzed (Participants) | 60 | 53 | 53 | 53
  Week 54: Highly Cytolytic Subset Of NK Cells | 22.2 (10.7) | 24.5 (11.0) | 22.8 (11.5) | 22.1 (11.0)
  Week 80: Highly Cytolytic Subset Of NK Cells: number analyzed (Participants) | 59 | 44 | 52 | 50
  Week 80: Highly Cytolytic Subset Of NK Cells | 21.1 (9.7) | 23.0 (9.1) | 25.5 (11.4) | 21.9 (9.9)
  Week 0: Mature CD16+ Highly Functional NK Cells: number analyzed (Participants) | 71 | 65 | 65 | 68
  Week 0: Mature CD16+ Highly Functional NK Cells | 0.7 (0.7) | 0.7 (0.6) | 0.6 (0.6) | 0.7 (0.6)
  Week 54: Mature CD16+ Highly Functional NK Cells: number analyzed (Participants) | 60 | 53 | 53 | 53
  Week 54: Mature CD16+ Highly Functional NK Cells | 0.6 (0.6) | 0.6 (0.8) | 0.6 (0.7) | 0.6 (0.5)
  Week 80: Mature CD16+ Highly Functional NK Cells: number analyzed (Participants) | 59 | 44 | 52 | 50
  Week 80: Mature CD16+ Highly Functional NK Cells | 0.6 (0.7) | 0.6 (0.5) | 0.5 (0.6) | 0.7 (0.7)
  Week 0: Mature CD16+ Terminally Differentiated: number analyzed (Participants) | 71 | 65 | 65 | 68
  Week 0: Mature CD16+ Terminally Differentiated | 1.3 (1.3) | 1.1 (1.2) | 1.1 (1.1) | 1.3 (1.1)
  Week 54: Mature CD16+ Terminally Differentiated: number analyzed (Participants) | 60 | 53 | 53 | 53
  Week 54: Mature CD16+ Terminally Differentiated | 0.9 (0.7) | 0.8 (0.7) | 1.0 (0.9) | 1.1 (0.9)
  Week 80: Mature CD16+ Terminally Differentiated: number analyzed (Participants) | 59 | 44 | 52 | 50
  Week 80: Mature CD16+ Terminally Differentiated | 1.1 (1.1) | 1.0 (1.0) | 0.8 (0.9) | 1.3 (1.0)
  Week 0: Mature CD16- Terminally Differentiate NK: number analyzed (Participants) | 71 | 65 | 65 | 68
  Week 0: Mature CD16- Terminally Differentiate NK | 0.3 (0.2) | 0.3 (0.2) | 0.4 (0.4) | 0.4 (0.3)
  Week 54: Mature CD16- Terminally Differentiate NK: number analyzed (Participants) | 60 | 53 | 53 | 53
  Week 54: Mature CD16- Terminally Differentiate NK | 0.3 (0.2) | 0.3 (0.2) | 0.3 (0.3) | 0.4 (0.2)
  Week 80: Mature CD16- Terminally Differentiate NK: number analyzed (Participants) | 59 | 44 | 52 | 50
  Week 80: Mature CD16- Terminally Differentiate NK | 0.3 (0.2) | 0.3 (0.3) | 0.4 (0.3) | 1.0 (4.2)
  Week 0: Mature Cytolytic NK Cells: number analyzed (Participants) | 71 | 65 | 65 | 68
  Week 0: Mature Cytolytic NK Cells | 2.3 (1.4) | 2.2 (1.1) | 2.4 (1.7) | 2.3 (1.3)
  Week 54: Mature Cytolytic NK Cells: number analyzed (Participants) | 60 | 53 | 53 | 53
  Week 54: Mature Cytolytic NK Cells | 2.4 (1.4) | 2.7 (1.5) | 2.5 (1.6) | 2.4 (1.7)
  Week 80: Mature Cytolytic NK Cells: number analyzed (Participants) | 59 | 44 | 52 | 50
  Week 80: Mature Cytolytic NK Cells | 2.3 (1.2) | 2.9 (3.7) | 2.6 (2.3) | 2.5 (1.5)
  Week 0: Mature Rapid Cytokine-Producing NK Cell: number analyzed (Participants) | 71 | 65 | 65 | 68
  Week 0: Mature Rapid Cytokine-Producing NK Cell | 3.6 (2.5) | 3.8 (2.8) | 3.3 (2.2) | 3.6 (2.8)
  Week 54: Mature Rapid Cytokine-Producing NK Cell: number analyzed (Participants) | 60 | 53 | 53 | 53
  Week 54: Mature Rapid Cytokine-Producing NK Cell | 3.6 (2.4) | 3.9 (2.4) | 3.0 (2.0) | 3.3 (2.4)
  Week 80: Mature Rapid Cytokine-Producing NK Cell: number analyzed (Participants) | 59 | 44 | 52 | 50
  Week 80: Mature Rapid Cytokine-Producing NK Cell | 3.2 (2.0) | 3.7 (2.4) | 3.0 (1.9) | 3.9 (3.0)
  Week 0: Rapid Cytokine-Producing NK Cell Subset: number analyzed (Participants) | 71 | 65 | 65 | 68
  Week 0: Rapid Cytokine-Producing NK Cell Subset | 4.1 (2.7) | 4.4 (3.1) | 3.8 (2.6) | 4.1 (3.2)
  Week 54: Rapid Cytokine-Producing NK Cell Subset: number analyzed (Participants) | 60 | 53 | 53 | 53
  Week 54: Rapid Cytokine-Producing NK Cell Subset | 4.2 (2.7) | 4.5 (2.8) | 3.5 (2.3) | 3.8 (2.6)
  Week 80: Rapid Cytokine-Producing NK Cell Subset: number analyzed (Participants) | 59 | 44 | 52 | 50
  Week 80: Rapid Cytokine-Producing NK Cell Subset | 3.8 (2.3) | 4.4 (2.7) | 3.7 (2.3) | 4.6 (3.4)
  Week 0: Senescent CD16+ CD56- NK cells: number analyzed (Participants) | 71 | 65 | 65 | 68
  Week 0: Senescent CD16+ CD56- NK cells | 1.3 (1.8) | 1.2 (1.9) | 1.0 (1.1) | 1.2 (1.2)
  Week 54: Senescent CD16+ CD56- NK cells: number analyzed (Participants) | 60 | 53 | 53 | 53
  Week 54: Senescent CD16+ CD56- NK cells | 1.0 (1.1) | 1.2 (1.5) | 0.9 (0.9) | 1.1 (1.1)
  Week 80: Senescent CD16+ CD56- NK cells: number analyzed (Participants) | 59 | 44 | 52 | 50
  Week 80: Senescent CD16+ CD56- NK cells | 1.1 (1.4) | 1.4 (1.5) | 0.9 (0.9) | 1.2 (1.0)
  Week 0: Senescent CD16+CD56hi NK: number analyzed (Participants) | 71 | 65 | 65 | 68
  Week 0: Senescent CD16+CD56hi NK | 0.1 (0.2) | 0.1 (0.1) | 0.1 (0.1) | 0.1 (0.1)
  Week 54: Week 0: Senescent CD16+CD56hi NK: number analyzed (Participants) | 60 | 53 | 53 | 53
  Week 54: Week 0: Senescent CD16+CD56hi NK | 0.1 (0.1) | 0.0 (0.1) | 0.1 (0.1) | 0.0 (0.1)
  Week 80: Week 0: Senescent CD16+CD56hi NK: number analyzed (Participants) | 59 | 44 | 52 | 50
  Week 80: Week 0: Senescent CD16+CD56hi NK | 0.1 (0.1) | 0.0 (0.0) | 0.1 (0.1) | 0.1 (0.1)
  Week 0: Senescent CD16- CD56- NK cells: number analyzed (Participants) | 71 | 65 | 65 | 68
  Week 0: Senescent CD16- CD56- NK cells | 1.3 (1.0) | 1.5 (1.6) | 1.3 (1.0) | 1.5 (1.1)
  Week 54: Senescent CD16- CD56- NK cells: number analyzed (Participants) | 60 | 53 | 53 | 53
  Week 54: Senescent CD16- CD56- NK cells | 1.5 (1.2) | 1.8 (1.3) | 1.6 (1.3) | 2.0 (2.9)
  Week 80: Senescent CD16- CD56- NK cells: number analyzed (Participants) | 59 | 44 | 52 | 50
  Week 80: Senescent CD16- CD56- NK cells | 1.9 (2.0) | 2.4 (3.7) | 1.9 (1.3) | 2.2 (3.3)
  Week 0: Senescent Cytolytic NK Cells: number analyzed (Participants) | 71 | 65 | 65 | 68
  Week 0: Senescent Cytolytic NK Cells | 8.7 (6.6) | 9.9 (7.2) | 9.8 (7.2) | 9.9 (6.0)
  Week 54: Senescent Cytolytic NK Cells: number analyzed (Participants) | 60 | 53 | 53 | 53
  Week 54: Senescent Cytolytic NK Cells | 9.9 (6.3) | 11.3 (7.6) | 10.9 (7.9) | 9.6 (6.7)
  Week 80: Senescent Cytolytic NK Cells: number analyzed (Participants) | 59 | 44 | 52 | 50
  Week 80: Senescent Cytolytic NK Cells | 9.4 (6.1) | 11.1 (7.1) | 11.5 (7.9) | 9.8 (7.3)
  Week 0: Senescent Rapid Cytokine-Producing NK: number analyzed (Participants) | 71 | 65 | 65 | 68
  Week 0: Senescent Rapid Cytokine-Producing NK | 0.1 (0.3) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Week 54: Senescent Rapid Cytokine-Producing NK: number analyzed (Participants) | 60 | 53 | 53 | 53
  Week 54: Senescent Rapid Cytokine-Producing NK | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.1) | 0.0 (0.0)
  Week 80: Senescent Rapid Cytokine-Producing NK: number analyzed (Participants) | 59 | 44 | 52 | 50
  Week 80: Senescent Rapid Cytokine-Producing NK | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.1)
  Week 0: Total CD16+ CD56- NK: number analyzed (Participants) | 71 | 65 | 65 | 68
  Week 0: Total CD16+ CD56- NK | 6.7 (3.8) | 7.4 (5.1) | 6.4 (3.5) | 7.3 (3.8)
  Week 54: Total CD16+ CD56- NK: number analyzed (Participants) | 60 | 53 | 53 | 53
  Week 54: Total CD16+ CD56- NK | 5.9 (2.6) | 6.2 (3.8) | 6.0 (3.1) | 6.8 (3.5)
  Week 80: Total CD16+ CD56- NK: number analyzed (Participants) | 59 | 44 | 52 | 50
  Week 80: Total CD16+ CD56- NK | 6.8 (5.8) | 6.6 (4.1) | 6.2 (3.0) | 7.3 (3.5)
  Week 0: Total CD16- CD56- NK: number analyzed (Participants) | 71 | 65 | 65 | 68
  Week 0: Total CD16- CD56- NK | 27.6 (15.4) | 29.2 (13.2) | 31.4 (16.7) | 30.5 (13.0)
  Week 54: Week 0: Total CD16- CD56- NK: number analyzed (Participants) | 60 | 53 | 53 | 53
  Week 54: Week 0: Total CD16- CD56- NK | 28.6 (12.2) | 30.1 (11.9) | 31.9 (13.3) | 34.0 (14.1)
  Week 80: Week 0: Total CD16- CD56- NK: number analyzed (Participants) | 59 | 44 | 52 | 50
  Week 80: Week 0: Total CD16- CD56- NK | 29.2 (12.7) | 30.7 (13.2) | 30.7 (10.2) | 30.0 (12.2)
  Week 0: Total Mature NK Cells; Highly Cytolytic: number analyzed (Participants) | 71 | 65 | 65 | 68
  Week 0: Total Mature NK Cells; Highly Cytolytic | 58.6 (13.4) | 57.4 (15.1) | 56.8 (16.6) | 56.3 (13.7)
  Week 54: Total Mature NK Cells; Highly Cytolytic: number analyzed (Participants) | 60 | 53 | 53 | 53
  Week 54: Total Mature NK Cells; Highly Cytolytic | 59.6 (13.4) | 57.3 (12.9) | 56.9 (13.8) | 53.7 (15.0)
  Week 80: Total Mature NK Cells; Highly Cytolytic: number analyzed (Participants) | 59 | 44 | 52 | 50
  Week 80: Total Mature NK Cells; Highly Cytolytic | 58.5 (13.9) | 56.5 (13.4) | 57.7 (12.1) | 56.2 (11.6)

98. Secondary Outcome: Change in Biomarker: Immune Phenotyping- T Cell Panel
Description: T cell panel is evaluated by Immune phenotyping of peripheral blood mononuclear cells (PBMC) at baseline (week 0), week 54 and week 80.
  In below table CD refer to Cluster of Differentiation; TEMRA refers to terminally differentiated effector memory cells re-expressing CD45RA; CCR refers to C-C chemokine receptor; TREG refers to Regulatory T cells.
Time Frame: Week 0, week 54 and week 80
Population: The FAS included all randomised participants. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of T cells (%)
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Percentage of T cells (%)
  Week 0: Activated CD4 TEMRA: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: Activated CD4 TEMRA | 10.1 (7.1) | 9.7 (5.4) | 10.8 (6.8) | 9.7 (6.5)
  Week 54: Activated CD4 TEMRA: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: Activated CD4 TEMRA | 10.3 (5.9) | 8.7 (5.3) | 9.7 (5.4) | 9.3 (6.0)
  Week 80: Activated CD4 TEMRA: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: Activated CD4 TEMRA | 9.1 (5.5) | 8.1 (5.5) | 8.1 (4.9) | 8.7 (5.0)
  Week 0: Activated CD8 TEMRA: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: Activated CD8 TEMRA | 0.9 (1.2) | 0.8 (1.4) | 0.6 (0.6) | 1.0 (1.9)
  Week 54: Activated CD8 TEMRA: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: Activated CD8 TEMRA | 0.9 (1.5) | 0.6 (0.7) | 0.6 (0.6) | 0.7 (1.0)
  Week 80: Activated CD8 TEMRA: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: Activated CD8 TEMRA | 0.7 (0.9) | 0.6 (0.7) | 0.6 (0.6) | 1.1 (2.3)
  Week 0: Activated Central Memory CD4: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: Activated Central Memory CD4 | 6.3 (3.3) | 6.7 (3.1) | 7.1 (3.8) | 6.1 (3.2)
  Week 54: Activated Central Memory CD4: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: Activated Central Memory CD4 | 6.3 (3.1) | 6.1 (3.1) | 6.3 (2.9) | 6.2 (3.1)
  Week 80: Activated Central Memory CD4: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: Activated Central Memory CD4 | 6.5 (3.0) | 6.0 (2.6) | 6.0 (2.6) | 6.5 (2.8)
  Week 0: Activated Central Memory CD8: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: Activated Central Memory CD8 | 1.1 (1.2) | 1.7 (1.8) | 1.6 (1.7) | 1.1 (1.0)
  Week 54: Activated Central Memory CD8: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: Activated Central Memory CD8 | 1.4 (1.6) | 1.6 (1.8) | 1.5 (1.4) | 3.1 (13.3)
  Week 80: Activated Central Memory CD8: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: Activated Central Memory CD8 | 2.2 (6.5) | 1.4 (1.5) | 1.6 (2.3) | 1.9 (4.5)
  Week 0: Activated Effector Memory CD4: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: Activated Effector Memory CD4 | 10.3 (5.8) | 10.9 (5.6) | 11.3 (6.4) | 9.4 (4.8)
  Week 54: Activated Effector Memory CD4: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: Activated Effector Memory CD4 | 10.1 (5.4) | 9.6 (5.2) | 10.0 (4.9) | 9.2 (4.8)
  Week 80: Activated Effector Memory CD4: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: Activated Effector Memory CD4 | 10.2 (6.6) | 8.9 (4.3) | 9.5 (4.8) | 9.1 (4.3)
  Week 0: Activated Effector Memory CD8: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: Activated Effector Memory CD8 | 1.9 (3.6) | 1.7 (2.9) | 1.2 (1.4) | 0.9 (1.2)
  Week 54: Activated Effector Memory CD8: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: Activated Effector Memory CD8 | 2.0 (3.7) | 1.6 (2.4) | 1.2 (1.2) | 1.1 (1.4)
  Week 80: Activated Effector Memory CD8: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: Activated Effector Memory CD8 | 1.9 (3.4) | 1.5 (2.8) | 1.4 (2.0) | 1.1 (1.4)
  Week 0: Activated Mature Naive CD4 T-Cells: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: Activated Mature Naive CD4 T-Cells | 4.0 (2.0) | 4.0 (1.9) | 4.7 (2.4) | 3.9 (1.8)
  Week 54: Activated Mature Naive CD4 T-Cells: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: Activated Mature Naive CD4 T-Cells | 3.9 (2.1) | 3.8 (1.8) | 4.5 (2.3) | 3.7 (1.4)
  Week 80: Activated Mature Naive CD4 T-Cells: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: Activated Mature Naive CD4 T-Cells | 4.0 (2.4) | 3.8 (1.4) | 4.0 (1.9) | 3.9 (1.7)
  Week 0: Activated Mature Naive CD8 T-Cells: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: Activated Mature Naive CD8 T-Cells | 3.4 (3.7) | 2.8 (2.3) | 3.3 (3.5) | 3.5 (3.7)
  Week 54: Activated Mature Naive CD8 T-Cells: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: Activated Mature Naive CD8 T-Cells | 3.0 (3.3) | 2.6 (3.0) | 2.6 (2.7) | 3.1 (3.6)
  Week 80: Activated Mature Naive CD8 T-Cells: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: Activated Mature Naive CD8 T-Cells | 2.7 (2.1) | 2.6 (2.5) | 2.5 (2.7) | 3.1 (3.2)
  Week 0: CCR5+ CD4 TEMRA: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: CCR5+ CD4 TEMRA | 17.7 (12.2) | 16.4 (8.1) | 16.9 (11.1) | 18.9 (12.8)
  Week 54: CCR5+ CD4 TEMRA: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: CCR5+ CD4 TEMRA | 18.4 (12.2) | 17.7 (10.3) | 18.8 (13.5) | 21.0 (17.3)
  Week 80: CCR5+ CD4 TEMRA: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: CCR5+ CD4 TEMRA | 18.3 (11.0) | 19.5 (13.6) | 18.6 (11.9) | 21.4 (15.1)
  Week 0: CCR5+ CD4 Treg TEMRA: number analyzed (Participants) | 65 | 65 | 60 | 67
  Week 0: CCR5+ CD4 Treg TEMRA | 3.7 (10.6) | 1.7 (1.8) | 2.7 (4.7) | 3.9 (8.6)
  Week 54: CCR5+ CD4 Treg TEMRA: number analyzed (Participants) | 59 | 52 | 52 | 52
  Week 54: CCR5+ CD4 Treg TEMRA | 4.2 (9.1) | 4.2 (10.4) | 4.6 (10.5) | 4.6 (9.3)
  Week 80: CCR5+ CD4 Treg TEMRA: number analyzed (Participants) | 58 | 46 | 53 | 50
  Week 80: CCR5+ CD4 Treg TEMRA | 2.8 (4.6) | 4.4 (10.4) | 3.2 (5.7) | 4.4 (9.3)
  Week 0: CCR5+ CD8 EM: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: CCR5+ CD8 EM | 35.3 (14.5) | 35.5 (13.8) | 38.2 (14.1) | 37.7 (15.8)
  Week 54: CCR5+ CD8 EM: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: CCR5+ CD8 EM | 37.9 (14.1) | 36.4 (13.5) | 38.0 (14.4) | 38.8 (15.5)
  Week 80: CCR5+ CD8 EM: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: CCR5+ CD8 EM | 38.8 (15.3) | 34.7 (12.4) | 37.5 (14.1) | 40.0 (16.3)
  Week 0: CCR5+ CD8 TEMRA: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: CCR5+ CD8 TEMRA | 22.8 (10.2) | 22.9 (10.9) | 25.9 (12.9) | 24.3 (12.6)
  Week 54: CCR5+ CD8 TEMRA: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: CCR5+ CD8 TEMRA | 25.9 (10.7) | 25.0 (9.7) | 26.3 (12.1) | 25.4 (11.6)
  Week 80: CCR5+ CD8 TEMRA: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: CCR5+ CD8 TEMRA | 25.9 (11.3) | 24.4 (11.3) | 26.8 (13.4) | 26.9 (13.1)
  Week 0: CCR5+ Central Memory CD4 Cells: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: CCR5+ Central Memory CD4 Cells | 4.1 (2.4) | 4.3 (2.3) | 4.5 (2.9) | 4.5 (3.2)
  Week 54: CCR5+ Central Memory CD4 Cells: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: CCR5+ Central Memory CD4 Cells | 4.5 (2.5) | 4.1 (2.0) | 4.1 (2.8) | 4.9 (3.4)
  Week 80: CCR5+ Central Memory CD4 Cells: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: CCR5+ Central Memory CD4 Cells | 4.9 (2.5) | 4.9 (3.7) | 5.1 (3.4) | 5.7 (4.7)
  Week 0: CCR5+ Central Memory CD8 Cells: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: CCR5+ Central Memory CD8 Cells | 15.0 (10.6) | 14.4 (9.0) | 16.9 (10.3) | 16.7 (11.1)
  Week 54: CCR5+ Central Memory CD8 Cells: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: CCR5+ Central Memory CD8 Cells | 16.8 (9.0) | 14.2 (9.7) | 15.8 (9.7) | 18.5 (15.6)
  Week 80: CCR5+ Central Memory CD8 Cells: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: CCR5+ Central Memory CD8 Cells | 16.8 (8.9) | 15.5 (8.9) | 15.8 (9.2) | 19.3 (13.5)
  Week 0: CCR5+ Central Memory Regulatory T-Cells: number analyzed (Participants) | 65 | 65 | 60 | 67
  Week 0: CCR5+ Central Memory Regulatory T-Cells | 1.9 (1.7) | 1.8 (1.4) | 1.8 (1.9) | 1.5 (1.1)
  Week 54: CCR5+ Central Memory Regulatory T-Cells: number analyzed (Participants) | 59 | 52 | 52 | 52
  Week 54: CCR5+ Central Memory Regulatory T-Cells | 2.0 (1.7) | 1.5 (1.3) | 1.7 (1.8) | 1.7 (1.3)
  Week 80: CCR5+ Central Memory Regulatory T-Cells: number analyzed (Participants) | 58 | 46 | 53 | 50
  Week 80: CCR5+ Central Memory Regulatory T-Cells | 2.1 (1.9) | 1.8 (1.7) | 1.9 (1.9) | 2.2 (2.4)
  Week 0: CCR5+ Effector Memory CD4: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: CCR5+ Effector Memory CD4 | 15.5 (7.9) | 14.5 (7.6) | 15.5 (8.3) | 15.3 (7.4)
  Week 54: CCR5+ Effector Memory CD4: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: CCR5+ Effector Memory CD4 | 16.2 (7.7) | 15.7 (7.6) | 14.9 (7.5) | 16.9 (9.6)
  Week 80: CCR5+ Effector Memory CD4: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: CCR5+ Effector Memory CD4 | 17.5 (7.5) | 16.8 (9.2) | 16.4 (8.0) | 18.4 (10.9)
  Week 0: CCR5+ Effector Memory Regulatory T-Cells: number analyzed (Participants) | 65 | 65 | 60 | 67
  Week 0: CCR5+ Effector Memory Regulatory T-Cells | 4.7 (3.5) | 5.1 (3.3) | 4.5 (3.9) | 4.1 (2.3)
  Week 54: CCR5+ Effector Memory Regulatory T-Cells: number analyzed (Participants) | 59 | 52 | 52 | 52
  Week 54: CCR5+ Effector Memory Regulatory T-Cells | 4.8 (3.0) | 4.6 (3.1) | 4.4 (3.3) | 4.5 (2.5)
  Week 80: CCR5+ Effector Memory Regulatory T-Cells: number analyzed (Participants) | 58 | 46 | 53 | 50
  Week 80: CCR5+ Effector Memory Regulatory T-Cells | 5.2 (3.6) | 5.2 (4.0) | 5.4 (5.3) | 5.2 (3.2)
  Week 0: CCR5+ Naive CD4 T-Cells: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: CCR5+ Naive CD4 T-Cells | 1.9 (1.5) | 2.0 (1.3) | 2.1 (1.9) | 2.0 (1.8)
  Week 54: CCR5+ Naive CD4 T-Cells: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: CCR5+ Naive CD4 T-Cells | 2.0 (1.5) | 2.1 (2.1) | 2.1 (1.9) | 2.3 (2.2)
  Week 80: CCR5+ Naive CD4 T-Cells: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: CCR5+ Naive CD4 T-Cells | 2.3 (1.6) | 2.9 (3.9) | 2.8 (3.0) | 3.5 (5.1)
  Week 0: CCR5+ Naive CD8 T-Cells: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: CCR5+ Naive CD8 T-Cells | 3.7 (2.3) | 3.5 (1.9) | 4.1 (2.8) | 4.2 (3.2)
  Week 54: CCR5+ Naive CD8 T-Cells: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: CCR5+ Naive CD8 T-Cells | 3.4 (1.7) | 3.5 (2.4) | 3.5 (2.1) | 4.1 (2.9)
  Week 80: CCR5+ Naive CD8 T-Cells: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: CCR5+ Naive CD8 T-Cells | 3.8 (1.8) | 4.0 (4.3) | 4.3 (3.1) | 4.9 (4.7)
  Week 0: CCR5+ Naive Regulatory T-Cells: number analyzed (Participants) | 65 | 65 | 60 | 67
  Week 0: CCR5+ Naive Regulatory T-Cells | 6.1 (6.5) | 5.0 (3.6) | 6.5 (8.3) | 6.5 (8.8)
  Week 54: CCR5+ Naive Regulatory T-Cells: number analyzed (Participants) | 59 | 52 | 52 | 52
  Week 54: CCR5+ Naive Regulatory T-Cells | 6.7 (10.1) | 6.3 (7.3) | 4.8 (5.5) | 5.3 (5.2)
  Week 80: CCR5+ Naive Regulatory T-Cells: number analyzed (Participants) | 58 | 46 | 53 | 50
  Week 80: CCR5+ Naive Regulatory T-Cells | 5.8 (4.9) | 6.5 (8.4) | 5.7 (6.5) | 7.1 (8.0)
  Week 0: CD4 TEMRA: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: CD4 TEMRA | 3.7 (4.9) | 2.6 (1.7) | 3.1 (2.5) | 2.7 (2.3)
  Week 54: CD4 TEMRA: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: CD4 TEMRA | 3.8 (5.7) | 2.9 (2.3) | 3.3 (2.8) | 3.1 (3.2)
  Week 80: CD4 TEMRA: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: CD4 TEMRA | 4.4 (5.8) | 3.2 (2.3) | 3.6 (3.2) | 3.5 (2.6)
  Week 0: CD8 Central Memory: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: CD8 Central Memory | 2.0 (1.8) | 2.0 (2.1) | 1.8 (1.5) | 1.9 (1.3)
  Week 54: CD8 Central Memory: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: CD8 Central Memory | 1.8 (1.2) | 2.1 (2.3) | 1.7 (1.4) | 2.1 (1.6)
  Week 80: CD8 Central Memory: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: CD8 Central Memory | 1.8 (1.6) | 1.9 (2.0) | 1.8 (1.5) | 2.2 (2.0)
  Week 0: CD8 Effector Memory: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: CD8 Effector Memory | 14.3 (7.9) | 14.7 (7.6) | 13.4 (7.7) | 15.7 (6.9)
  Week 54: CD8 Effector Memory: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: CD8 Effector Memory | 15.1 (7.6) | 14.8 (7.8) | 11.3 (6.6) | 16.4 (7.4)
  Week 80: CD8 Effector Memory: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: CD8 Effector Memory | 15.1 (8.0) | 16.5 (9.0) | 13.9 (7.6) | 17.4 (7.5)
  Week 0: CD8 TEMRA: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: CD8 TEMRA | 31.6 (12.8) | 30.9 (13.9) | 29.0 (12.8) | 32.3 (13.8)
  Week 54: CD8 TEMRA: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: CD8 TEMRA | 29.8 (12.3) | 31.0 (13.9) | 30.3 (12.9) | 30.4 (13.3)
  Week 80: CD8 TEMRA: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: CD8 TEMRA | 31.9 (14.3) | 33.5 (13.1) | 30.4 (13.0) | 33.4 (14.6)
  Week 0: Conventional Central Memory CD4 T-Cells: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: Conventional Central Memory CD4 T-Cells | 20.0 (9.9) | 22.1 (8.0) | 20.3 (8.1) | 21.6 (8.0)
  Week 54: Conventional Central Memory CD4 T-Cells: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: Conventional Central Memory CD4 T-Cells | 20.4 (8.1) | 22.2 (9.3) | 19.9 (7.8) | 21.1 (8.0)
  Week 80: Conventional Central Memory CD4 T-Cells: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: Conventional Central Memory CD4 T-Cells | 19.4 (8.4) | 21.7 (7.8) | 19.9 (8.2) | 21.1 (8.7)
  Week 0: Conventional Effector Memory CD4 T-Cells: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: Conventional Effector Memory CD4 T-Cells | 19.2 (10.7) | 22.8 (10.3) | 19.5 (9.5) | 20.7 (9.2)
  Week 54: Conventional Effector Memory CD4 T-Cells: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: Conventional Effector Memory CD4 T-Cells | 20.3 (9.6) | 22.9 (11.0) | 20.5 (10.7) | 21.3 (9.7)
  Week 80: Conventional Effector Memory CD4 T-Cells: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: Conventional Effector Memory CD4 T-Cells | 20.0 (9.8) | 24.4 (11.3) | 20.9 (11.7) | 23.2 (10.0)
  Week 0: Naive CD4 T-Cells: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: Naive CD4 T-Cells | 57.0 (14.7) | 52.4 (14.4) | 57.0 (12.6) | 54.9 (13.2)
  Week 54: Naive CD4 T-Cells: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: Naive CD4 T-Cells | 55.4 (11.9) | 51.8 (15.0) | 56.3 (13.9) | 54.5 (12.5)
  Week 80: Naive CD4 T-Cells: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: Naive CD4 T-Cells | 56.1 (11.9) | 50.6 (16.2) | 55.6 (15.1) | 52.1 (14.5)
  Week 0: Naive CD8 T-Cells: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: Naive CD8 T-Cells | 52.0 (15.9) | 52.5 (19.1) | 55.8 (17.0) | 50.1 (17.4)
  Week 54: Naive CD8 T-Cells: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: Naive CD8 T-Cells | 53.2 (14.9) | 52.1 (18.1) | 54.7 (15.4) | 51.1 (17.4)
  Week 80: Naive CD8 T-Cells: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: Naive CD8 T-Cells | 51.1 (16.0) | 48.1 (19.2) | 53.9 (17.4) | 46.9 (17.6)
  Week 0: Senescent CD4 Central Memory Cells: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: Senescent CD4 Central Memory Cells | 2.3 (1.9) | 2.2 (1.5) | 2.4 (2.6) | 2.3 (2.7)
  Week 54: Senescent CD4 Central Memory Cells: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: Senescent CD4 Central Memory Cells | 1.9 (1.5) | 2.1 (1.7) | 2.2 (1.9) | 2.4 (2.5)
  Week 80: Senescent CD4 Central Memory Cells: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: Senescent CD4 Central Memory Cells | 2.3 (1.8) | 2.3 (1.6) | 2.1 (1.6) | 2.6 (2.4)
  Week 0: Senescent CD4 Effector Memory Cells: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: Senescent CD4 Effector Memory Cells | 6.9 (5.5) | 6.3 (5.6) | 6.9 (5.4) | 6.7 (6.5)
  Week 54: Senescent CD4 Effector Memory Cells: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: Senescent CD4 Effector Memory Cells | 5.9 (5.8) | 6.7 (6.0) | 6.6 (4.9) | 7.5 (9.0)
  Week 80: Senescent CD4 Effector Memory Cells: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: Senescent CD4 Effector Memory Cells | 6.9 (5.9) | 7.0 (5.2) | 6.4 (4.7) | 7.6 (7.4)
  Week 0: Senescent CD8 Central Memory Cells: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: Senescent CD8 Central Memory Cells | 12.1 (10.1) | 11.5 (9.1) | 12.9 (9.7) | 12.4 (12.7)
  Week 54: Senescent CD8 Central Memory Cells: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: Senescent CD8 Central Memory Cells | 11.7 (9.5) | 10.4 (9.2) | 12.0 (10.2) | 12.2 (14.5)
  Week 80: Senescent CD8 Central Memory Cells: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: Senescent CD8 Central Memory Cells | 12.7 (9.0) | 12.7 (9.9) | 11.3 (9.8) | 12.2 (11.9)
  Week 0: Senescent CD8 Effector Memory Cells: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: Senescent CD8 Effector Memory Cells | 27.3 (14.8) | 27.2 (15.5) | 27.7 (13.6) | 29.1 (17.4)
  Week 54: Senescent CD8 Effector Memory Cells: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: Senescent CD8 Effector Memory Cells | 25.2 (13.1) | 25.1 (14.3) | 26.1 (12.8) | 25.8 (14.7)
  Week 80: Senescent CD8 Effector Memory Cells: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: Senescent CD8 Effector Memory Cells | 27.5 (14.5) | 28.6 (15.7) | 26.5 (14.1) | 26.6 (15.5)
  Week 0: Senescent Naive CD4 T-Cells: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: Senescent Naive CD4 T-Cells | 2.6 (2.7) | 2.9 (3.3) | 2.6 (2.3) | 2.5 (2.3)
  Week 54: Senescent Naive CD4 T-Cells: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: Senescent Naive CD4 T-Cells | 2.5 (2.5) | 3.0 (3.8) | 2.8 (3.0) | 2.7 (2.4)
  Week 80: Senescent Naive CD4 T-Cells: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: Senescent Naive CD4 T-Cells | 3.1 (3.3) | 3.3 (3.8) | 3.1 (3.7) | 3.9 (5.3)
  Week 0: Senescent Naive CD8 T-Cells: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: Senescent Naive CD8 T-Cells | 3.9 (3.4) | 3.6 (3.5) | 3.5 (3.1) | 4.2 (4.4)
  Week 54: Senescent Naive CD8 T-Cells: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: Senescent Naive CD8 T-Cells | 3.5 (2.9) | 3.8 (4.5) | 3.7 (4.3) | 4.2 (3.6)
  Week 80: Senescent Naive CD8 T-Cells: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: Senescent Naive CD8 T-Cells | 4.4 (4.3) | 4.3 (4.7) | 3.8 (3.6) | 4.5 (4.1)
  Week 0: Senescent Naive TREG: number analyzed (Participants) | 65 | 65 | 60 | 67
  Week 0: Senescent Naive TREG | 6.9 (7.9) | 5.5 (3.7) | 7.1 (8.5) | 7.3 (9.3)
  Week 54: Senescent Naive TREG: number analyzed (Participants) | 59 | 52 | 52 | 52
  Week 54: Senescent Naive TREG | 7.2 (10.9) | 6.8 (7.8) | 5.0 (5.5) | 5.6 (5.2)
  Week 80: Senescent Naive TREG: number analyzed (Participants) | 58 | 46 | 53 | 50
  Week 80: Senescent Naive TREG | 6.3 (5.7) | 7.0 (8.9) | 6.0 (7.2) | 7.4 (8.2)
  Week 0: Senescent TEMRA CD4: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: Senescent TEMRA CD4 | 23.3 (19.8) | 21.7 (18.4) | 21.9 (21.7) | 22.0 (20.1)
  Week 54: Senescent TEMRA CD4: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: Senescent TEMRA CD4 | 20.0 (17.1) | 22.8 (18.3) | 23.1 (22.2) | 23.5 (21.7)
  Week 80: Senescent TEMRA CD4: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: Senescent TEMRA CD4 | 21.0 (19.5) | 24.2 (18.1) | 21.7 (21.5) | 25.4 (21.6)
  Week 0: Senescent TEMRA CD8: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: Senescent TEMRA CD8 | 42.8 (20.2) | 40.3 (21.0) | 37.7 (19.4) | 42.0 (23.0)
  Week 54: Senescent TEMRA CD8: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: Senescent TEMRA CD8 | 39.2 (19.8) | 40.7 (21.3) | 38.3 (18.4) | 40.4 (22.9)
  Week 80: Senescent TEMRA CD8: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: Senescent TEMRA CD8 | 42.7 (21.4) | 44.8 (20.9) | 38.7 (20.4) | 43.5 (23.1)
  Week 0: Senescent TEMRA TREG: number analyzed (Participants) | 65 | 65 | 60 | 67
  Week 0: Senescent TEMRA TREG | 3.6 (19.7) | 1.8 (1.9) | 2.8 (4.6) | 4.0 (8.6)
  Week 54: Senescent TEMRA TREG: number analyzed (Participants) | 59 | 52 | 52 | 52
  Week 54: Senescent TEMRA TREG | 3.9 (9.0) | 4.2 (10.4) | 4.6 (10.5) | 4.6 (9.1)
  Week 80: Senescent TEMRA TREG: number analyzed (Participants) | 58 | 46 | 53 | 50
  Week 80: Senescent TEMRA TREG | 2.6 (4.5) | 4.4 (10.4) | 3.2 (5.7) | 4.4 (9.3)
  Week 0: Senescent TREG CM: number analyzed (Participants) | 65 | 65 | 60 | 67
  Week 0: Senescent TREG CM | 0.1 (0.1) | 0.1 (0.1) | 0.1 (0.2) | 0.2 (0.2)
  Week 54: Senescent TREG CM: number analyzed (Participants) | 59 | 52 | 52 | 52
  Week 54: Senescent TREG CM | 0.1 (0.1) | 0.1 (0.1) | 0.1 (0.2) | 0.2 (0.2)
  Week 80: Senescent TREG CM: number analyzed (Participants) | 58 | 46 | 53 | 50
  Week 80: Senescent TREG CM | 0.2 (0.2) | 0.2 (0.1) | 0.1 (0.2) | 0.3 (0.5)
  Week 0: Senescent TREG EM: number analyzed (Participants) | 65 | 65 | 60 | 67
  Week 0: Senescent TREG EM | 0.4 (0.4) | 0.4 (0.3) | 0.4 (0.5) | 0.4 (0.4)
  Week 54: Senescent TREG EM: number analyzed (Participants) | 59 | 52 | 52 | 52
  Week 54: Senescent TREG EM | 0.4 (0.4) | 0.3 (0.3) | 0.3 (0.3) | 0.5 (0.5)
  Week 80: Senescent TREG EM: number analyzed (Participants) | 58 | 46 | 53 | 50
  Week 80: Senescent TREG EM | 0.5 (0.7) | 0.5 (0.9) | 0.5 (0.7) | 0.5 (0.7)
  Week 0: Total Naive TREG: number analyzed (Participants) | 65 | 65 | 60 | 67
  Week 0: Total Naive TREG | 46.8 (18.1) | 42.4 (14.1) | 50.3 (14.2) | 47.7 (17.6)
  Week 54: Total Naive TREG: number analyzed (Participants) | 59 | 52 | 52 | 52
  Week 54: Total Naive TREG | 43.7 (15.6) | 44.3 (15.8) | 49.4 (15.4) | 45.1 (13.7)
  Week 80: Total Naive TREG: number analyzed (Participants) | 58 | 46 | 53 | 50
  Week 80: Total Naive TREG | 46.8 (15.7) | 44.1 (18.3) | 48.7 (17.0) | 43.4 (15.2)
  Week 0: Total TREG: number analyzed (Participants) | 65 | 65 | 60 | 67
  Week 0: Total TREG | 3.9 (1.9) | 3.8 (1.5) | 4.1 (1.6) | 3.5 (1.3)
  Week 54: Total TREG: number analyzed (Participants) | 59 | 52 | 52 | 52
  Week 54: Total TREG | 3.8 (1.5) | 3.5 (1.5) | 4.0 (1.5) | 3.5 (1.2)
  Week 80: Total TREG: number analyzed (Participants) | 58 | 46 | 53 | 50
  Week 80: Total TREG | 3.7 (1.5) | 3.5 (1.3) | 3.4 (1.2) | 3.4 (1.2)
  Week 0: Total TREG CM: number analyzed (Participants) | 65 | 65 | 60 | 67
  Week 0: Total TREG CM | 14.8 (9.2) | 15.8 (8.1) | 14.4 (7.9) | 14.2 (7.9)
  Week 54: Total TREG CM: number analyzed (Participants) | 59 | 52 | 52 | 52
  Week 54: Total TREG CM | 15.5 (9.0) | 15.6 (9.5) | 13.8 (7.8) | 15.0 (6.7)
  Week 80: Total TREG CM: number analyzed (Participants) | 58 | 46 | 53 | 50
  Week 80: Total TREG CM | 15.3 (8.7) | 15.0 (8.2) | 13.8 (7.4) | 15.9 (8.2)
  Week 0: Total TREG EM: number analyzed (Participants) | 65 | 65 | 60 | 67
  Week 0: Total TREG EM | 30.8 (14.6) | 36.4 (11.2) | 28.8 (12.2) | 30.7 (15.2)
  Week 54: Total TREG EM: number analyzed (Participants) | 59 | 52 | 52 | 52
  Week 54: Total TREG EM | 32.4 (14.6) | 32.6 (12.5) | 28.3 (12.9) | 31.9 (13.6)
  Week 80: Total TREG EM: number analyzed (Participants) | 58 | 46 | 53 | 50
  Week 80: Total TREG EM | 30.7 (13.7) | 33.5 (13.9) | 30.2 (15.0) | 32.9 (13.3)
  Week 0: Total TREG TEMRA: number analyzed (Participants) | 65 | 65 | 60 | 67
  Week 0: Total TREG TEMRA | 7.6 (11.5) | 5.5 (3.5) | 6.7 (5.7) | 7.5 (9.0)
  Week 54: Total TREG TEMRA: number analyzed (Participants) | 59 | 52 | 52 | 52
  Week 54: Total TREG TEMRA | 8.5 (11.4) | 7.7 (10.5) | 8.6 (10.4) | 8.2 (10.3)
  Week 80: Total TREG TEMRA: number analyzed (Participants) | 58 | 46 | 53 | 50
  Week 80: Total TREG TEMRA | 7.3 (8.1) | 7.4 (10.3) | 7.5 (6.8) | 7.8 (9.3)
  Week 0: Total Viable CD4 T-Cells: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: Total Viable CD4 T-Cells | 54.7 (10.7) | 53.2 (8.7) | 54.6 (11.3) | 54.6 (11.5)
  Week 54: Total Viable CD4 T-Cells: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: Total Viable CD4 T-Cells | 54.3 (11.3) | 52.1 (12.2) | 54.6 (12.7) | 52.7 (12.7)
  Week 80: Total Viable CD4 T-Cells: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: Total Viable CD4 T-Cells | 51.9 (13.3) | 50.3 (13.8) | 53.1 (12.6) | 52.2 (13.5)
  Week 0: Total Viable CD8 T-Cells: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: Total Viable CD8 T-Cells | 26.1 (8.1) | 28.2 (8.7) | 25.8 (7.6) | 26.6 (8.3)
  Week 54: Total Viable CD8 T-Cells: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: Total Viable CD8 T-Cells | 25.0 (7.9) | 26.7 (9.4) | 24.6 (7.9) | 24.0 (9.8)
  Week 80: Total Viable CD8 T-Cells: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: Total Viable CD8 T-Cells | 24.2 (8.9) | 25.4 (9.5) | 23.5 (8.9) | 23.9 (9.7)
  Week 0: Total Viable T-Cells: number analyzed (Participants) | 70 | 68 | 63 | 71
  Week 0: Total Viable T-Cells | 55.6 (7.1) | 55.2 (8.1) | 55.3 (8.0) | 55.0 (7.2)
  Week 54: Total Viable T-Cells: number analyzed (Participants) | 61 | 55 | 55 | 55
  Week 54: Total Viable T-Cells | 53.6 (7.0) | 55.9 (6.7) | 57.4 (7.7) | 55.5 (8.7)
  Week 80: Total Viable T-Cells: number analyzed (Participants) | 60 | 48 | 55 | 54
  Week 80: Total Viable T-Cells | 52.7 (8.6) | 55.3 (7.9) | 56.2 (8.0) | 55.8 (7.9)

99. Secondary Outcome: Change in Biomarker: Immune Phenotyping- T Follicular Helper (TfH) Cell Panel
Description: TfH cell panel is evaluated by Immune phenotyping of peripheral blood mononuclear cells (PBMC) at baseline (week 0), week 54 and week 80.
  In below table CTFH refer to Circulating T follicular helper; ICOS refers to inducible T-cell co-stimulator; PD refers to Programmed cell death protein; CCR refers to C-C chemokine receptor; CXCR refers to C-X-C chemokine receptor; CD refer to Cluster of Differentiation; CM refers to central memory; EM refers to effector memory, TIGIT refers to T cell immunoreceptor with Ig and ITIM domains.
Time Frame: Week 0, week 54 and week 80
Population: The FAS included all randomised participants. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of TfH cells (%)
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Percentage of TfH cells (%)
  Week 0: Activated cTfh17 Cells: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: Activated cTfh17 Cells | 0.8 (1.2) | 1.0 (2.2) | 0.8 (1.6) | 0.6 (0.9)
  Week 54: Activated cTfh17 Cells: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: Activated cTfh17 Cells | 0.6 (1.2) | 0.4 (0.8) | 0.7 (1.2) | 0.9 (2.0)
  Week 80: Activated cTfh17 Cells: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: Activated cTfh17 Cells | 0.8 (2.0) | 1.1 (2.9) | 0.6 (0.8) | 0.9 (1.4)
  Week 0: Activated cTfh2 Cells: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: Activated cTfh2 Cells | 0.6 (0.6) | 0.6 (0.6) | 0.6 (0.5) | 0.6 (0.6)
  Week 54: Activated cTfh2 Cells: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: Activated cTfh2 Cells | 0.4 (0.4) | 0.4 (0.4) | 0.7 (1.2) | 0.6 (0.6)
  Week 80: Activated cTfh2 Cells: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: Activated cTfh2 Cells | 0.6 (0.6) | 0.5 (0.3) | 0.5 (0.5) | 0.6 (0.6)
  Week 0:Activated PD1+ICOS+ cTfh1: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0:Activated PD1+ICOS+ cTfh1 | 1.3 (1.7) | 1.9 (7.7) | 1.1 (1.2) | 1.0 (1.1)
  Week 54: Activated PD1+ICOS+ cTfh1: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: Activated PD1+ICOS+ cTfh1 | 0.7 (0.6) | 1.0 (1.2) | 1.2 (2.5) | 1.2 (1.4)
  Week 80: Activated PD1+ICOS+ cTfh1: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: Activated PD1+ICOS+ cTfh1 | 0.7 (0.6) | 0.9 (1.0) | 1.0 (2.1) | 1.1 (2.5)
  Week 0: CCR7+ cTfh1 Cells: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: CCR7+ cTfh1 Cells | 96.9 (2.5) | 97.1 (3.5) | 94.7 (13.4) | 97.2 (2.2)
  Week 54: CCR7+ cTfh1 Cells: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: CCR7+ cTfh1 Cells | 97.1 (2.5) | 95.8 (13.1) | 97.1 (4.2) | 97.3 (2.3)
  Week 80: CCR7+ cTfh1 Cells: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: CCR7+ cTfh1 Cells | 97.0 (3.0) | 96.8 (3.0) | 97.4 (2.1) | 97.0 (2.3)
  Week 0: CCR7+ cTfh17 Cells: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: CCR7+ cTfh17 Cells | 97.4 (11.7) | 97.4 (11.9) | 97.4 (12.5) | 97.3 (11.8)
  Week 54: CCR7+ cTfh17 Cells: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: CCR7+ cTfh17 Cells | 98.1 (2.9) | 93.9 (22.3) | 96.9 (12.9) | 95.3 (18.3)
  Week 80: CCR7+ cTfh17 Cells: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: CCR7+ cTfh17 Cells | 98.7 (1.5) | 97.3 (5.9) | 96.8 (13.4) | 98.7 (1.4)
  Week 0: CCR7+ cTfh2 Cells: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: CCR7+ cTfh2 Cells | 98.1 (1.6) | 98.2 (1.4) | 98.2 (1.5) | 98.3 (1.4)
  Week 54: CCR7+ cTfh2 Cells: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: CCR7+ cTfh2 Cells | 98.1 (1.9) | 98.5 (1.2) | 98.3 (1.1) | 98.1 (1.6)
  Week 80: CCR7+ cTfh2 Cells: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: CCR7+ cTfh2 Cells | 98.3 (1.5) | 98.3 (1.8) | 98.4 (1.1) | 98.3 (1.0)
  Week 0: CXCR4+ cTfh1 Cells: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: CXCR4+ cTfh1 Cells | 59.4 (27.6) | 58.0 (25.9) | 54.9 (27.8) | 55.6 (29.2)
  Week 54: CXCR4+ cTfh1 Cells: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: CXCR4+ cTfh1 Cells | 64.5 (28.7) | 64.5 (28.8) | 64.4 (29.3) | 69.4 (25.0)
  Week 80: CXCR4+ cTfh1 Cells: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: CXCR4+ cTfh1 Cells | 70.8 (24.5) | 66.4 (27.4) | 63.5 (30.3) | 66.8 (25.2)
  Week 0: CXCR4+ cTfh17 Cells: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: CXCR4+ cTfh17 Cells | 50.9 (30.4) | 45.8 (27.8) | 43.7 (29.3) | 45.1 (31.4)
  Week 54: CXCR4+ cTfh17 Cells: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: CXCR4+ cTfh17 Cells | 56.1 (31.1) | 54.0 (29.3) | 53.1 (31.4) | 56.4 (29.6)
  Week 80: CXCR4+ cTfh17 Cells: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: CXCR4+ cTfh17 Cells | 60.0 (27.4) | 57.2 (30.3) | 54.6 (31.4) | 57.6 (28.5)
  Week 0: CXCR4+ Ctfh2 Cells: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: CXCR4+ Ctfh2 Cells | 58.8 (26.8) | 56.3 (25.2) | 54.0 (26.3) | 54.5 (28.8)
  Week 54: CXCR4+ Ctfh2 Cells: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: CXCR4+ Ctfh2 Cells | 63.3 (28.2) | 65.2 (27.3) | 63.7 (28.5) | 67.7 (25.3)
  Week 80: CXCR4+ Ctfh2 Cells: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: CXCR4+ Ctfh2 Cells | 69.3 (23.9) | 65.8 (27.1) | 62.7 (29.5) | 66.7 (24.7)
  Week 0: Circulating TFH-Cells (cTfh): number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: Circulating TFH-Cells (cTfh) | 5.5 (3.7) | 5.4 (3.4) | 6.2 (3.3) | 6.1 (3.7)
  Week 54: Circulating TFH-Cells (cTfh): number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: Circulating TFH-Cells (cTfh) | 5.7 (3.3) | 5.6 (3.9) | 6.2 (4.0) | 6.2 (4.4)
  Week 80: Circulating TFH-Cells (cTfh): number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: Circulating TFH-Cells (cTfh) | 5.8 (3.3) | 5.9 (4.1) | 6.1 (4.2) | 5.8 (3.8)
  Week 0: ICOS+ CD4 CM: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: ICOS+ CD4 CM | 0.5 (0.5) | 0.5 (0.5) | 0.4 (0.3) | 0.5 (0.4)
  Week 54: ICOS+ CD4 CM: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: ICOS+ CD4 CM | 0.3 (0.2) | 0.3 (0.2) | 0.4 (0.2) | 0.4 (0.3)
  Week 80: ICOS+ CD4 CM: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: ICOS+ CD4 CM | 0.3 (0.3) | 0.3 (0.2) | 0.3 (0.2) | 0.3 (0.2)
  Week 0: ICOS+ CD4 EM: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: ICOS+ CD4 EM | 0.2 (0.2) | 0.3 (0.6) | 0.2 (0.2) | 0.2 (0.2)
  Week 54: ICOS+ CD4 EM: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: ICOS+ CD4 EM | 0.2 (0.1) | 0.2 (0.1) | 0.2 (0.1) | 0.2 (0.1)
  Week 80: ICOS+ CD4 EM: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: ICOS+ CD4 EM | 0.2 (0.1) | 0.2 (0.1) | 0.2 (0.5) | 0.2 (0.1)
  Week 0: ICOS+ CD4 TEMRA: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: ICOS+ CD4 TEMRA | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Week 54: ICOS+ CD4 TEMRA: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: ICOS+ CD4 TEMRA | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Week 80: ICOS+ CD4 TEMRA: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: ICOS+ CD4 TEMRA | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.1) | 0.0 (0.0)
  Week 0: ICOS+ NAIVE CD4 T-Cells: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: ICOS+ NAIVE CD4 T-Cells | 0.1 (0.1) | 0.1 (0.1) | 0.1 (0.1) | 0.1 (0.1)
  Week 54: ICOS+ NAIVE CD4 T-Cells: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: ICOS+ NAIVE CD4 T-Cells | 0.0 (0.1) | 0.0 (0.0) | 0.0 (0.1) | 0.1 (0.1)
  Week 80: ICOS+ NAIVE CD4 T-Cells: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: ICOS+ NAIVE CD4 T-Cells | 0.0 (0.1) | 0.0 (0.0) | 0.0 (0.1) | 0.0 (0.0)
  Week 0: ICOS+ NAIVE TREG: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: ICOS+ NAIVE TREG | 2.3 (1.8) | 2.7 (3.4) | 1.9 (2.1) | 2.5 (2.8)
  Week 54: ICOS+ NAIVE TREG: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: ICOS+ NAIVE TREG | 2.1 (2.0) | 2.0 (2.4) | 1.9 (2.5) | 2.4 (2.5)
  Week 80: ICOS+ NAIVE TREG: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: ICOS+ NAIVE TREG | 2.2 (2.2) | 2.1 (2.4) | 1.9 (2.3) | 2.7 (2.7)
  Week 0: ICOS+ TREG CM: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: ICOS+ TREG CM | 10.9 (5.3) | 11.3 (5.8) | 10.4 (5.4) | 11.0 (5.9)
  Week 54: ICOS+ TREG CM: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: ICOS+ TREG CM | 10.0 (5.2) | 9.2 (4.4) | 9.7 (4.7) | 10.6 (5.1)
  Week 80: ICOS+ TREG CM: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: ICOS+ TREG CM | 10.1 (4.9) | 9.0 (4.3) | 8.8 (5.2) | 10.5 (4.4)
  Week 0: ICOS+ TREG EM: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: ICOS+ TREG EM | 12.8 (6.4) | 13.3 (6.8) | 13.0 (6.2) | 12.8 (6.5)
  Week 54: ICOS+ TREG EM: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: ICOS+ TREG EM | 11.9 (5.8) | 11.6 (5.9) | 12.8 (6.1) | 12.7 (5.9)
  Week 80: ICOS+ TREG EM: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: ICOS+ TREG EM | 12.0 (5.5) | 11.3 (5.4) | 10.5 (5.3) | 12.0 (5.8)
  Week 0: ICOS+ TREG TEMRA: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: ICOS+ TREG TEMRA | 10.2 (10.6) | 13.0 (18.4) | 10.5 (11.4) | 9.3 (8.6)
  Week 54: ICOS+ TREG TEMRA: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: ICOS+ TREG TEMRA | 8.8 (10.5) | 9.7 (10.7) | 11.0 (12.6) | 12.8 (15.1)
  Week 80: ICOS+ TREG TEMRA: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: ICOS+ TREG TEMRA | 9.9 (9.8) | 9.6 (10.1) | 8.2 (9.2) | 11.0 (10.5)
  Week 0: PD1+ CD4 Central Memory: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: PD1+ CD4 Central Memory | 6.2 (4.0) | 6.7 (4.9) | 7.2 (5.3) | 6.6 (4.3)
  Week 54: PD1+ CD4 Central Memory: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: PD1+ CD4 Central Memory | 6.4 (4.7) | 6.8 (5.4) | 7.2 (5.4) | 6.7 (3.9)
  Week 80: PD1+ CD4 Central Memory: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: PD1+ CD4 Central Memory | 6.7 (5.5) | 7.5 (5.9) | 6.8 (4.8) | 7.2 (5.3)
  Week 0: PD1+ CD4 Effector Memory: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: PD1+ CD4 Effector Memory | 4.0 (3.2) | 4.2 (2.3) | 4.0 (2.8) | 4.1 (2.6)
  Week 54: PD1+ CD4 Effector Memory: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: PD1+ CD4 Effector Memory | 3.7 (3.0) | 3.9 (2.2) | 3.6 (2.3) | 4.0 (2.5)
  Week 80: PD1+ CD4 Effector Memory: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: PD1+ CD4 Effector Memory | 3.9 (2.7) | 4.3 (2.3) | 3.6 (2.2) | 4.3 (2.4)
  Week 0: PD1+ Naive CD4: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: PD1+ Naive CD4 | 3.8 (6.1) | 3.0 (4.7) | 4.2 (6.8) | 3.2 (4.4)
  Week 54: PD1+ Naive CD4: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: PD1+ Naive CD4 | 4.2 (6.2) | 2.9 (4.0) | 4.4 (6.8) | 3.5 (4.6)
  Week 80: PD1+ Naive CD4: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: PD1+ Naive CD4 | 5.0 (8.4) | 3.3 (4.6) | 4.2 (6.6) | 3.8 (6.2)
  Week 0: PD1+ Naive TREG: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: PD1+ Naive TREG | 8.4 (6.8) | 8.7 (7.5) | 8.4 (7.9) | 8.5 (8.0)
  Week 54: PD1+ Naive TREG: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: PD1+ Naive TREG | 9.8 (7.9) | 9.4 (9.5) | 9.1 (8.5) | 9.4 (8.2)
  Week 80: PD1+ Naive TREG: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: PD1+ Naive TREG | 11.0 (9.8) | 10.1 (9.1) | 9.3 (8.2) | 10.7 (9.2)
  Week 0: PD1+ TEMRA TREG: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: PD1+ TEMRA TREG | 22.5 (19.0) | 23.5 (17.5) | 19.8 (15.0) | 19.5 (13.5)
  Week 54: PD1+ TEMRA TREG: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: PD1+ TEMRA TREG | 20.5 (13.7) | 19.7 (16.2) | 18.6 (14.0) | 21.4 (13.9)
  Week 80: PD1+ TEMRA TREG: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: PD1+ TEMRA TREG | 22.5 (15.0) | 25.7 (19.5) | 22.4 (16.6) | 22.7 (13.0)
  Week 0: PD1+ TREG CM: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: PD1+ TREG CM | 16.8 (10.0) | 17.5 (11.5) | 17.3 (11.0) | 17.2 (10.2)
  Week 54: PD1+ TREG CM: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: PD1+ TREG CM | 16.5 (10.5) | 16.7 (10.9) | 16.8 (11.4) | 18.0 (10.6)
  Week 80: PD1+ TREG CM: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: PD1+ TREG CM | 18.1 (13.0) | 18.7 (11.2) | 16.6 (11.0) | 18.8 (11.6)
  Week 0: PD1+ TREG EM: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: PD1+ TREG EM | 20.1 (9.9) | 21.1 (11.4) | 21.6 (10.9) | 20.9 (10.0)
  Week 54: PD1+ TREG EM: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: PD1+ TREG EM | 19.3 (10.5) | 19.8 (10.3) | 21.1 (11.6) | 21.6 (10.7)
  Week 80: PD1+ TREG EM: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: PD1+ TREG EM | 20.6 (12.2) | 21.1 (10.5) | 19.4 (10.6) | 21.9 (10.0)
  Week 0: PD1+ICOSNeg cTfh1: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: PD1+ICOSNeg cTfh1 | 30.0 (14.8) | 28.8 (15.3) | 32.4 (16.5) | 29.7 (13.2)
  Week 54: PD1+ICOSNeg cTfh1: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: PD1+ICOSNeg cTfh1 | 30.5 (16.2) | 29.1 (13.9) | 34.2 (19.0) | 31.0 (13.5)
  Week 80: PD1+ICOSNeg cTfh1: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: PD1+ICOSNeg cTfh1 | 32.4 (18.1) | 30.7 (16.0) | 31.3 (14.0) | 32.8 (13.6)
  Week 0: PD1+ICOSNeg cTfh17: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: PD1+ICOSNeg cTfh17 | 21.8 (16.3) | 22.5 (16.3) | 23.7 (17.1) | 22.3 (15.7)
  Week 54: PD1+ICOSNeg cTfh17: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: PD1+ICOSNeg cTfh17 | 21.8 (17.4) | 21.1 (16.9) | 26.2 (19.7) | 21.7 (15.5)
  Week 80: PD1+ICOSNeg cTfh17: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: PD1+ICOSNeg cTfh17 | 26.8 (19.2) | 24.7 (16.0) | 23.6 (15.8) | 24.3 (15.5)
  Week 0: PD1+ICOSNeg cTfh2: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: PD1+ICOSNeg cTfh2 | 19.1 (12.0) | 18.4 (12.6) | 20.8 (14.3) | 18.5 (11.2)
  Week 54: PD1+ICOSNeg cTfh2: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: PD1+ICOSNeg cTfh2 | 18.4 (13.3) | 18.1 (13.1) | 20.2 (14.4) | 18.8 (11.7)
  Week 80: PD1+ICOSNeg cTfh2: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: PD1+ICOSNeg cTfh2 | 20.2 (16.6) | 19.6 (13.9) | 18.9 (11.7) | 20.2 (13.2)
  Week 0: PD1- ICOS- cTfh1: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: PD1- ICOS- cTfh1 | 68.4 (15.1) | 69.0 (16.3) | 64.6 (17.9) | 68.9 (13.5)
  Week 54: PD1- ICOS- cTfh1: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: PD1- ICOS- cTfh1 | 68.6 (16.4) | 68.0 (16.5) | 64.1 (19.7) | 67.5 (14.1)
  Week 80: PD1- ICOS- cTfh1: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: PD1- ICOS- cTfh1 | 66.7 (18.2) | 68.1 (16.1) | 67.4 (14.4) | 65.9 (14.0)
  Week 0: PD1- ICOS- cTfh17: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: PD1- ICOS- cTfh17 | 75.6 (18.8) | 74.7 (18.2) | 73.4 (19.3) | 75.3 (18.1)
  Week 54: PD1- ICOS- cTfh17: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: PD1- ICOS- cTfh17 | 77.4 (17.9) | 72.9 (23.7) | 70.9 (21.5) | 73.5 (20.9)
  Week 80: PD1- ICOS- cTfh17: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: PD1- ICOS- cTfh17 | 72.1 (20.1) | 74.0 (16.2) | 73.6 (18.7) | 74.6 (15.8)
  Week 0: PD1- ICOS- cTfh2: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: PD1- ICOS- cTfh2 | 80.1 (12.2) | 80.8 (12.8) | 78.3 (14.2) | 80.7 (11.5)
  Week 54: PD1- ICOS- cTfh2: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: PD1- ICOS- cTfh2 | 81.0 (13.3) | 81.3 (13.3) | 78.8 (14.3) | 80.3 (11.9)
  Week 80: PD1- ICOS- cTfh2: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: PD1- ICOS- cTfh2 | 79.1 (16.9) | 79.8 (13.9) | 80.4 (11.9) | 79.0 (13.4)
  Week 0: Potentially Anergic TEMRA CD4: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: Potentially Anergic TEMRA CD4 | 0.7 (2.5) | 0.2 (0.3) | 0.4 (1.0) | 0.3 (0.7)
  Week 54: Potentially Anergic TEMRA CD4: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: Potentially Anergic TEMRA CD4 | 0.8 (3.0) | 0.2 (0.3) | 0.5 (1.3) | 0.3 (0.5)
  Week 80: Potentially Anergic TEMRA CD4: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: Potentially Anergic TEMRA CD4 | 0.8 (2.9) | 0.2 (0.3) | 0.5 (1.4) | 0.3 (0.7)
  Week 0: Regulatory T-Follicular Subset: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: Regulatory T-Follicular Subset | 0.2 (0.2) | 0.2 (0.2) | 0.2 (0.2) | 0.2 (0.2)
  Week 54: Regulatory T-Follicular Subset: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: Regulatory T-Follicular Subset | 0.2 (0.2) | 0.2 (0.2) | 0.2 (0.2) | 0.3 (0.2)
  Week 80: Regulatory T-Follicular Subset: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: Regulatory T-Follicular Subset | 0.2 (0.2) | 0.2 (0.3) | 0.2 (0.3) | 0.3 (0.3)
  Week 0: TH17-Like Circulating T-Follicular cells: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: TH17-Like Circulating T-Follicular cells | 0.5 (0.5) | 0.4 (0.4) | 0.5 (0.5) | 0.5 (0.5)
  Week 54: TH17-Like Circulating T-Follicular cells: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: TH17-Like Circulating T-Follicular cells | 0.4 (0.4) | 0.4 (0.4) | 0.4 (0.5) | 0.4 (0.4)
  Week 80: TH17-Like Circulating T-Follicular cells: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: TH17-Like Circulating T-Follicular cells | 0.4 (0.5) | 0.4 (0.5) | 0.3 (0.3) | 0.4 (0.5)
  Week 0: TH2-Like Circulating T-Follicular Cells: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: TH2-Like Circulating T-Follicular Cells | 3.6 (2.2) | 3.6 (2.0) | 4.0 (2.0) | 4.1 (2.3)
  Week 54: TH2-Like Circulating T-Follicular Cells: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: TH2-Like Circulating T-Follicular Cells | 3.9 (2.0) | 3.6 (2.2) | 4.0 (2.3) | 3.9 (2.5)
  Week 80: TH2-Like Circulating T-Follicular Cells: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: TH2-Like Circulating T-Follicular Cells | 3.8 (2.0) | 3.7 (2.1) | 3.9 (2.2) | 3.8 (2.1)
  Week 0: TIGIT+ cTfh1: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: TIGIT+ cTfh1 | 53.0 (11.6) | 48.5 (13.9) | 53.4 (12.4) | 51.6 (13.1)
  Week 54: TIGIT+ cTfh1: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: TIGIT+ cTfh1 | 51.1 (13.1) | 47.6 (13.9) | 52.2 (14.1) | 50.2 (14.1)
  Week 80: TIGIT+ cTfh1: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: TIGIT+ cTfh1 | 51.4 (11.1) | 48.1 (14.4) | 49.6 (10.4) | 52.7 (12.2)
  Week 0: TIGIT+ cTfh17: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: TIGIT+ cTfh17 | 40.5 (16.2) | 36.2 (13.1) | 39.3 (14.5) | 38.7 (14.9)
  Week 54: TIGIT+ cTfh17: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: TIGIT+ cTfh17 | 37.0 (13.5) | 31.4 (16.5) | 40.7 (14.7) | 35.8 (15.6)
  Week 80: TIGIT+ cTfh17: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: TIGIT+ cTfh17 | 39.4 (14.5) | 35.9 (13.9) | 35.3 (12.7) | 36.8 (13.8)
  Week 0: TIGIT+ cTfh2: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: TIGIT+ cTfh2 | 44.4 (9.5) | 40.9 (9.8) | 44.8 (7.4) | 43.4 (9.8)
  Week 54: TIGIT+ cTfh2: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: TIGIT+ cTfh2 | 41.1 (11.0) | 37.9 (10.9) | 42.0 (9.6) | 41.0 (11.6)
  Week 80: TIGIT+ cTfh2: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: TIGIT+ cTfh2 | 40.7 (10.4) | 38.4 (9.5) | 40.5 (8.4) | 41.9 (9.9)
  Week 0: TOTAL ICOS+ TREG: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: TOTAL ICOS+ TREG | 8.6 (4.4) | 9.6 (5.5) | 8.0 (3.8) | 8.9 (4.5)
  Week 54: TOTAL ICOS+ TREG: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: TOTAL ICOS+ TREG | 8.3 (4.8) | 7.5 (3.5) | 7.6 (3.8) | 8.6 (3.6)
  Week 80: TOTAL ICOS+ TREG: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: TOTAL ICOS+ TREG | 8.3 (4.4) | 7.4 (3.6) | 6.6 (3.3) | 8.6 (3.6)
  Week 0: Th1-Like Circulating T-Follicular Cells: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: Th1-Like Circulating T-Follicular Cells | 1.3 (1.4) | 1.3 (1.2) | 1.6 (1.2) | 1.5 (1.3)
  Week 54: Th1-Like Circulating T-Follicular Cells: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: Th1-Like Circulating T-Follicular Cells | 1.4 (1.2) | 1.6 (1.7) | 1.8 (1.5) | 1.8 (1.9)
  Week 80: Th1-Like Circulating T-Follicular Cells: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: Th1-Like Circulating T-Follicular Cells | 1.5 (1.4) | 1.8 (1.9) | 1.9 (2.0) | 1.6 (1.5)
  Week 0: Total PD1+ TREG: number analyzed (Participants) | 73 | 71 | 63 | 72
  Week 0: Total PD1+ TREG | 14.5 (7.9) | 15.1 (8.2) | 14.7 (8.9) | 14.4 (7.4)
  Week 54: Total PD1+ TREG: number analyzed (Participants) | 62 | 57 | 59 | 58
  Week 54: Total PD1+ TREG | 14.8 (9.1) | 14.3 (8.5) | 14.5 (9.1) | 15.0 (7.6)
  Week 80: Total PD1+ TREG: number analyzed (Participants) | 59 | 51 | 56 | 55
  Week 80: Total PD1+ TREG | 16.0 (10.6) | 15.9 (8.3) | 14.2 (9.0) | 16.1 (8.9)

100. Secondary Outcome: Change in Biomarker: Immune Phenotyping- Myeloid Cell Panel
Description: Myeloid panel is evaluated by Immune phenotyping of peripheral blood mononuclear cells (PBMC) at baseline (week 0), week 54 and week 80.
  In below table HLA refers to Human Leukocyte Antigen; MDSC refers to myeloid-derived suppressor cell; DC refers to Dendritic cells; MYDC refers to Myeloid Dendritic Cells; IMMYE_MDSC refers to Immature myeloid cells & a subset of myeloid suppressor cells within the CD14-HLA class II- myeloid cell population.
Time Frame: Week 0, week 54 and week 80
Population: The FAS included all randomised participants. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of Myeloid cells (%)
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Percentage of Myeloid cells (%)
  Week 0: CD14+ HLA low Myeloid Cells: number analyzed (Participants) | 70 | 69 | 65 | 71
  Week 0: CD14+ HLA low Myeloid Cells | 1.1 (1.5) | 1.0 (1.3) | 0.9 (1.2) | 1.0 (1.4)
  Week 54: CD14+ HLA low Myeloid Cells: number analyzed (Participants) | 60 | 54 | 54 | 54
  Week 54: CD14+ HLA low Myeloid Cells | 1.1 (2.3) | 0.7 (0.9) | 0.7 (1.1) | 0.6 (1.1)
  Week 80: CD14+ HLA low Myeloid Cells: number analyzed (Participants) | 58 | 45 | 54 | 52
  Week 80: CD14+ HLA low Myeloid Cells | 1.0 (2.2) | 0.6 (0.7) | 0.9 (1.2) | 0.8 (1.1)
  Week 0: CD14+ MDSC: number analyzed (Participants) | 70 | 69 | 65 | 71
  Week 0: CD14+ MDSC | 68.2 (20.8) | 69.1 (22.3) | 73.5 (19.4) | 70.3 (18.6)
  Week 54: CD14+ MDSC: number analyzed (Participants) | 60 | 54 | 54 | 54
  Week 54: CD14+ MDSC | 64.0 (23.4) | 67.0 (23.2) | 69.3 (21.4) | 65.9 (20.2)
  Week 80: CD14+ MDSC: number analyzed (Participants) | 58 | 45 | 54 | 52
  Week 80: CD14+ MDSC | 65.7 (22.3) | 62.7 (20.8) | 64.1 (23.3) | 63.9 (23.2)
  Week 0: CD14-HLA II- Myeloid Cells Total Myeloid: number analyzed (Participants) | 70 | 69 | 65 | 71
  Week 0: CD14-HLA II- Myeloid Cells Total Myeloid | 80.4 (11.0) | 82.2 (10.4) | 80.8 (12.1) | 81.8 (11.0)
  Week 54: CD14-HLA II- Myeloid Cells Total Myeloid: number analyzed (Participants) | 60 | 54 | 54 | 54
  Week 54: CD14-HLA II- Myeloid Cells Total Myeloid | 80.9 (11.7) | 80.0 (12.0) | 80.8 (12.7) | 83.5 (10.5)
  Week 80: CD14-HLA II- Myeloid Cells Total Myeloid: number analyzed (Participants) | 58 | 45 | 54 | 52
  Week 80: CD14-HLA II- Myeloid Cells Total Myeloid | 79.0 (12.9) | 81.0 (10.8) | 80.9 (9.7) | 81.3 (8.4)
  Week 0: CD16+ Dendritic Cells: number analyzed (Participants) | 70 | 69 | 65 | 71
  Week 0: CD16+ Dendritic Cells | 12.5 (8.4) | 11.3 (7.5) | 12.9 (10.6) | 11.5 (7.5)
  Week 54: CD16+ Dendritic Cells: number analyzed (Participants) | 60 | 54 | 54 | 54
  Week 54: CD16+ Dendritic Cells | 10.2 (8.1) | 10.3 (7.5) | 11.2 (9.7) | 12.0 (9.7)
  Week 80: CD16+ Dendritic Cells: number analyzed (Participants) | 58 | 45 | 54 | 52
  Week 80: CD16+ Dendritic Cells | 11.7 (10.6) | 9.4 (6.1) | 9.2 (7.1) | 12.1 (8.0)
  Week 0: IMMYE_MDSC: number analyzed (Participants) | 70 | 69 | 65 | 71
  Week 0: IMMYE_MDSC | 0.3 (0.2) | 0.2 (0.2) | 0.2 (0.2) | 0.2 (0.4)
  Week 54: IMMYE_MDSC: number analyzed (Participants) | 60 | 54 | 54 | 54
  Week 54: IMMYE_MDSC | 0.2 (0.3) | 0.2 (0.3) | 0.2 (0.3) | 0.1 (0.2)
  Week 80: IMMYE_MDSC: number analyzed (Participants) | 58 | 45 | 54 | 52
  Week 80: IMMYE_MDSC | 0.2 (0.3) | 0.1 (0.2) | 0.2 (0.2) | 0.2 (0.2)
  Week 0: Intermediate Monocyte Subset: number analyzed (Participants) | 70 | 69 | 65 | 71
  Week 0: Intermediate Monocyte Subset | 8.6 (8.4) | 9.0 (7.8) | 8.3 (8.8) | 7.7 (7.3)
  Week 54: Intermediate Monocyte Subset: number analyzed (Participants) | 60 | 54 | 54 | 54
  Week 54: Intermediate Monocyte Subset | 6.5 (4.8) | 7.3 (6.7) | 6.3 (7.1) | 5.8 (5.4)
  Week 80: Intermediate Monocyte Subset: number analyzed (Participants) | 58 | 45 | 54 | 52
  Week 80: Intermediate Monocyte Subset | 6.0 (5.1) | 6.6 (6.5) | 5.7 (5.4) | 5.8 (4.5)
  Week 0: Non-Classical Monocytes: number analyzed (Participants) | 70 | 69 | 65 | 71
  Week 0: Non-Classical Monocytes | 1.5 (1.3) | 1.3 (0.8) | 1.2 (0.8) | 1.3 (1.0)
  Week 54: Non-Classical Monocytes: number analyzed (Participants) | 60 | 54 | 54 | 54
  Week 54: Non-Classical Monocytes | 1.2 (1.1) | 1.3 (0.8) | 1.1 (0.8) | 1.2 (0.9)
  Week 80: Non-Classical Monocytes: number analyzed (Participants) | 58 | 45 | 54 | 52
  Week 80: Non-Classical Monocytes | 1.2 (0.7) | 1.2 (0.7) | 1.0 (0.6) | 1.3 (0.9)
  Week 0: Total Classical Monocytes: number analyzed (Participants) | 70 | 69 | 65 | 71
  Week 0: Total Classical Monocytes | 87.2 (9.3) | 86.7 (8.1) | 87.6 (9.1) | 88.0 (8.0)
  Week 54: Total Classical Monocytes: number analyzed (Participants) | 60 | 54 | 54 | 54
  Week 54: Total Classical Monocytes | 87.8 (7.9) | 88.1 (7.6) | 88.0 (8.8) | 89.3 (6.8)
  Week 80: Total Classical Monocytes: number analyzed (Participants) | 58 | 45 | 54 | 52
  Week 80: Total Classical Monocytes | 89.3 (6.0) | 88.5 (7.1) | 88.6 (7.0) | 89.7 (5.4)
  Week 0: Total Monocytes in Myeloid Cells: number analyzed (Participants) | 70 | 69 | 65 | 71
  Week 0: Total Monocytes in Myeloid Cells | 14.2 (8.9) | 12.6 (7.8) | 14.1 (9.5) | 13.4 (8.7)
  Week 54: Total Monocytes in Myeloid Cells: number analyzed (Participants) | 60 | 54 | 54 | 54
  Week 54: Total Monocytes in Myeloid Cells | 13.8 (9.3) | 14.9 (9.8) | 14.3 (10.6) | 12.2 (8.3)
  Week 80: Total Monocytes in Myeloid Cells: number analyzed (Participants) | 58 | 45 | 54 | 52
  Week 80: Total Monocytes in Myeloid Cells | 15.5 (10.3) | 13.8 (9.1) | 13.6 (7.6) | 13.5 (6.3)
  Week 0: Total Myeloid DC: number analyzed (Participants) | 70 | 69 | 65 | 71
  Week 0: Total Myeloid DC | 3.8 (2.1) | 3.6 (2.3) | 3.8 (2.8) | 3.4 (2.0)
  Week 54: Total Myeloid DC: number analyzed (Participants) | 60 | 54 | 54 | 54
  Week 54: Total Myeloid DC | 3.7 (2.3) | 3.9 (2.4) | 3.8 (2.4) | 3.2 (2.1)
  Week 80: Total Myeloid DC: number analyzed (Participants) | 58 | 45 | 54 | 52
  Week 80: Total Myeloid DC | 4.1 (2.3) | 4.1 (2.5) | 4.1 (3.0) | 3.9 (2.1)
  Week 0: Total MYDC: number analyzed (Participants) | 70 | 69 | 65 | 71
  Week 0: Total MYDC | 30.4 (9.1) | 31.4 (10.2) | 32.7 (9.2) | 31.0 (9.6)
  Week 54: Total MYDC: number analyzed (Participants) | 60 | 54 | 54 | 54
  Week 54: Total MYDC | 30.4 (11.3) | 31.3 (8.5) | 31.7 (11.9) | 27.2 (9.2)
  Week 80: Total MYDC: number analyzed (Participants) | 58 | 45 | 54 | 52
  Week 80: Total MYDC | 28.7 (10.7) | 30.5 (7.9) | 31.6 (12.0) | 31.9 (10.2)
  Week 0: Total Percent Of Myeloid Cells: number analyzed (Participants) | 70 | 69 | 65 | 71
  Week 0: Total Percent Of Myeloid Cells | 94.6 (3.8) | 94.7 (5.4) | 94.6 (3.4) | 94.6 (4.1)
  Week 54: Total Percent Of Myeloid Cells: number analyzed (Participants) | 60 | 54 | 54 | 54
  Week 54: Total Percent Of Myeloid Cells | 95.1 (3.6) | 95.9 (4.0) | 95.0 (3.8) | 95.6 (3.7)
  Week 80: Total Percent Of Myeloid Cells: number analyzed (Participants) | 58 | 45 | 54 | 52
  Week 80: Total Percent Of Myeloid Cells | 94.8 (5.4) | 95.6 (4.0) | 94.6 (4.4) | 94.1 (5.1)
  Week 0: Total Plasmacytoid Dendritic Cells (PDC): number analyzed (Participants) | 70 | 69 | 65 | 71
  Week 0: Total Plasmacytoid Dendritic Cells (PDC) | 14.3 (5.4) | 12.5 (6.6) | 12.0 (6.3) | 12.9 (7.5)
  Week 54: Total Plasmacytoid Dendritic Cells (PDC): number analyzed (Participants) | 60 | 54 | 54 | 54
  Week 54: Total Plasmacytoid Dendritic Cells (PDC) | 14.4 (6.7) | 13.5 (5.9) | 12.0 (6.1) | 11.8 (6.5)
  Week 80: Total Plasmacytoid Dendritic Cells (PDC): number analyzed (Participants) | 58 | 45 | 54 | 52
  Week 80: Total Plasmacytoid Dendritic Cells (PDC) | 13.5 (6.6) | 12.8 (6.7) | 11.6 (6.3) | 12.5 (6.7)

101. Secondary Outcome: Autoantibodies Against Glutamic Acid Decarboxylase (GAD)
Description: Participants were analyzed for autoantibodies against Glutamic acid decarboxylase (GAD) and were categorized as negative and positive.
Time Frame: Week 0, week 54 and week 80
Population: The FAS included all randomised participants. Number analyzed = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Participants
  Week 0: Negative | 3 | 1 | 5 | 3
  Week 0: Positive | 74 | 76 | 71 | 74
  Week 54: number analyzed (Participants) | 67 | 65 | 68 | 66
  Week 54: Negative | 5 | 4 | 4 | 3
  Week 54: Positive | 62 | 61 | 64 | 63
  Week 80: number analyzed (Participants) | 65 | 64 | 68 | 62
  Week 80: Negative | 4 | 2 | 5 | 1
  Week 80: Positive | 61 | 62 | 63 | 61

102. Secondary Outcome: Autoantibodies Against Zinc-transporter 8 (ZnT8)
Description: Participants were analyzed for autoantibodies against Zinc-transporter 8 (ZnT8) and were categorized as negative and positive.
Time Frame: Week 0, week 54 and week 80
Population: The FAS included all randomised participants. Number analyzed = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Participants
  Week 0: Negative | 29 | 30 | 30 | 36
  Week 0: Positive | 48 | 47 | 46 | 41
  Week 54: number analyzed (Participants) | 68 | 65 | 68 | 66
  Week 54: Negative | 26 | 28 | 27 | 33
  Week 54: Positive | 42 | 37 | 41 | 33
  Week 80: number analyzed (Participants) | 65 | 64 | 68 | 62
  Week 80: Negative | 23 | 30 | 31 | 33
  Week 80: Positive | 42 | 34 | 37 | 29

103. Secondary Outcome: Autoantibodies Against Islet Antigen-2 (IA2)
Description: Participants were analyzed for autoantibodies against Islet antigen-2 (IA2) and were categorized as negative and positive.
Time Frame: Week 0, week 54 and week 80
Population: The FAS included all randomised participants. Number analyzed = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Participants
  Week 0: Negative | 38 | 37 | 31 | 45
  Week 0: Positive | 39 | 40 | 45 | 32
  Week 54: number analyzed (Participants) | 68 | 65 | 68 | 66
  Week 54: Negative | 35 | 33 | 28 | 38
  Week 54: Positive | 33 | 32 | 40 | 28
  Week 80: number analyzed (Participants) | 65 | 64 | 68 | 62
  Week 80: Negative | 32 | 38 | 29 | 35
  Week 80: Positive | 33 | 26 | 39 | 27

104. Secondary Outcome: Autoantibodies Against Insulin Autoantibodies (IAA)
Description: Participants were analyzed for autoantibodies against Insulin autoantibodies (IAA) and were categorized as negative and positive.
Time Frame: Week 0, week 54 and week 80
Population: The FAS included all randomised participants. Number analyzed = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Participants
  Week 0: number analyzed (Participants) | 77 | 76 | 75 | 76
  Week 0: Negative | 35 | 28 | 26 | 36
  Week 0: Positive | 42 | 48 | 49 | 40
  Week 54: number analyzed (Participants) | 68 | 65 | 68 | 66
  Week 54: Negative | 30 | 28 | 22 | 11
  Week 54: Positive | 38 | 37 | 46 | 55
  Week 80: number analyzed (Participants) | 66 | 64 | 68 | 62
  Week 80: Negative | 18 | 24 | 13 | 15
  Week 80: Positive | 48 | 40 | 55 | 47

105. Secondary Outcome: Change in Biomarker: Total Interleukin-21 (IL-21)
Description: IL-21 is evaluated at baseline (week 0), week 54 and week 80.
Time Frame: Week 0, week 54 and week 80
Population: The FAS included all randomised participants. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: picogram per milliliter
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
picogram per milliliter
  Week 0: number analyzed (Participants) | 73 | 74 | 72 | 72
  Week 0 | 28.8 (10.2) | 31.1 (10.8) | 30.9 (10.7) | 30.2 (10.2)
  Week 54: number analyzed (Participants) | 68 | 65 | 68 | 66
  Week 54 | 3993.5 (2145.4) | 4368.2 (2374.9) | 25.0 (0.0) | 34.1 (68.1)
  Week 80: number analyzed (Participants) | 66 | 64 | 67 | 62
  Week 80 | 540.9 (495.3) | 674.1 (648.1) | 28.0 (8.2) | 30.7 (17.2)

106. Secondary Outcome: Change in Biomarker: Serum Vitamin D (1,25 Dehydroxy-calciferol)
Description: Serum vitamin D is evaluated at baseline (week 0), week 54 and week 80.
Time Frame: Week 0, week 54 and week 80
Population: The FAS included all randomised participants. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: picomole per liter
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
picomole per liter
  Week 0: number analyzed (Participants) | 67 | 72 | 67 | 70
  Week 0 | 123 (30) | 122 (39) | 122 (29) | 120 (33)
  Week 54: number analyzed (Participants) | 67 | 62 | 65 | 64
  Week 54 | 117 (31) | 125 (36) | 113 (30) | 119 (32)
  Week 80: number analyzed (Participants) | 64 | 63 | 66 | 62
  Week 80 | 119 (41) | 124 (49) | 121 (38) | 115 (33)

107. Secondary Outcome: Change in Short Form 36 Health Survey (SF-36)
Description: SF-36v2™ questionnaire measured the HRQoL on 8 domains (Bodily Pain, General Health, Mental Health, Physical Functioning, Role Emotion, Physical Health, Social Functioning and Vitality) on individual scale ranges. The scores 0-100 (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. Change from baseline (week 0) to week 54 and week 80 in SF-36 score is presented.The MCS measure is derived from domain scales of vitality, social functioning, role emotional and mental health. The PCS measure is derived from domain scales of physical functioning, role-physical, bodily pain, and general health. A norm-based score of 50 corresponds to the mean score and 10 corresponds to the standard deviation of the 2009 U.S. general population. A positive change score indicate an improvement since baseline.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: The FAS included all randomised participants. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Score on a scale
  Week 54: Bodily pain: number analyzed (Participants) | 76 | 71 | 73 | 72
  Week 54: Bodily pain | -0.8 (8.5) | -2.2 (7.6) | 0.1 (5.2) | 0.6 (9.1)
  Week 80: Bodily Pain: number analyzed (Participants) | 66 | 64 | 68 | 62
  Week 80: Bodily Pain | 0.8 (7.8) | -1.4 (7.0) | -0.5 (6.4) | 0.8 (10.2)
  Week 54: General Health Perception: number analyzed (Participants) | 76 | 71 | 73 | 72
  Week 54: General Health Perception | -1.1 (7.1) | -0.3 (8.4) | -1.6 (7.3) | -1.0 (7.1)
  Week 80: General Health Perception: number analyzed (Participants) | 66 | 64 | 68 | 62
  Week 80: General Health Perception | -0.9 (7.2) | 0.6 (9.0) | -1.7 (7.9) | -1.8 (8.6)
  Week 54: Mental Component Sum: number analyzed (Participants) | 76 | 71 | 73 | 72
  Week 54: Mental Component Sum | 0.5 (9.4) | 0.6 (9.3) | -2.1 (9.0) | -1.3 (7.6)
  Week 80: Mental Component Sum: number analyzed (Participants) | 66 | 64 | 68 | 62
  Week 80: Mental Component Sum | 1.7 (9.8) | -0.4 (8.9) | -2.4 (9.6) | -0.7 (8.7)
  week 54: Mental Health: number analyzed (Participants) | 76 | 71 | 73 | 72
  week 54: Mental Health | 0.7 (8.4) | 0.6 (7.9) | -1.5 (8.6) | -1.3 (6.9)
  Week 80: Mental Health: number analyzed (Participants) | 66 | 64 | 68 | 62
  Week 80: Mental Health | 1.5 (8.6) | -0.2 (8.0) | -1.5 (9.0) | -0.7 (7.6)
  Week 54: Physical Component Sum: number analyzed (Participants) | 76 | 71 | 73 | 72
  Week 54: Physical Component Sum | -0.4 (4.2) | -0.4 (5.3) | -0.1 (3.8) | 0.3 (5.7)
  Week 80: Physical Component Sum: number analyzed (Participants) | 66 | 64 | 68 | 62
  Week 80: Physical Component Sum | -0.1 (3.9) | 0.5 (5.4) | 0.0 (4.3) | 0.0 (6.9)
  Week 54: Physical Functioning: number analyzed (Participants) | 76 | 71 | 73 | 72
  Week 54: Physical Functioning | 0.6 (2.5) | 0.9 (4.4) | 0.0 (2.6) | 0.3 (5.8)
  Week 80: Physical Functioning: number analyzed (Participants) | 66 | 64 | 68 | 62
  Week 80: Physical Functioning | 0.5 (2.9) | 1.1 (4.6) | -0.1 (2.4) | 0.1 (6.4)
  Week 54:Lim Emotion Prob: number analyzed (Participants) | 76 | 71 | 73 | 72
  Week 54:Lim Emotion Prob | 0.3 (10.7) | 0.5 (8.9) | -1.4 (9.0) | -0.1 (8.5)
  Week 80: Lim Emotion Prob: number analyzed (Participants) | 66 | 64 | 68 | 62
  Week 80: Lim Emotion Prob | 1.2 (10.8) | -0.1 (9.8) | -2.2 (9.4) | 0.0 (8.3)
  Week 54: Lim. Phy Health: number analyzed (Participants) | 76 | 71 | 73 | 72
  Week 54: Lim. Phy Health | 0.3 (5.8) | 0.7 (6.9) | -0.6 (5.7) | -0.2 (6.9)
  Week 80: Lim. Phy Health: number analyzed (Participants) | 66 | 64 | 68 | 62
  Week 80: Lim. Phy Health | 0.8 (6.4) | 0.9 (7.0) | -0.2 (5.2) | 0.0 (7.3)
  Week 54: Social Functioning: number analyzed (Participants) | 76 | 71 | 73 | 72
  Week 54: Social Functioning | 0.8 (10.3) | 0.1 (10.0) | -1.4 (7.4) | 0.0 (8.5)
  Week 80: Social Functioning: number analyzed (Participants) | 66 | 64 | 68 | 62
  Week 80: Social Functioning | 2.3 (9.9) | 1.0 (8.3) | -1.2 (7.3) | -0.4 (8.4)
  Week 54: Vitality: number analyzed (Participants) | 76 | 71 | 73 | 72
  Week 54: Vitality | -0.5 (8.2) | 0.5 (7.9) | -2.2 (5.9) | -2.3 (6.9)
  Week 80: Vitality: number analyzed (Participants) | 66 | 64 | 68 | 62
  Week 80: Vitality | 0.5 (7.9) | -1.4 (6.9) | -2.2 (7.1) | -0.7 (6.9)

108. Secondary Outcome: Change in Experience of Treatment Benefits and Barriers (ETBB)
Description: Treatment Benefits and Barriers (ETBB) questionnaire measured diabetes-specific health beliefs on 2 categories: Total Score for Perceived Barriers and Perceived Benefits. The measurement of perceived benefits of, and barriers to, treatment was achieved by creating a pool 28 statements each with a 7-point scale ranging from strongly agree (6) to strongly disagree (0). ETBB benefits score was calculated using the responses from questions 1, 4, 7, 8, 10, and 12 and ETBB barriers score was calculated using the responses from questions 2, 3, 5, 6, 9, and 11. Both was calculated as the sum of responses divided by number of responses received multiplied by the maximum number of responses. Based on the responses used the maximum responses available was 6. The higher score indicates more perceived benefits or more perceived barrier.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: The FAS included all randomised participants. Number analyzed = participants with available data.
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
score on a scale
  Week 54: Total Score for Perceived Barriers: number analyzed (Participants) | 76 | 71 | 73 | 72
  Week 54: Total Score for Perceived Barriers | -1.2 (8.3) | -1.8 (7.7) | -0.2 (8.2) | -0.3 (6.3)
  Week 80: Total Score for Perceived Barriers: number analyzed (Participants) | 66 | 64 | 68 | 62
  Week 80: Total Score for Perceived Barriers | -2.0 (7.8) | -2.0 (7.5) | -0.1 (6.7) | 0.1 (8.3)
  Week 54: Total Score for Perceived Benefits: number analyzed (Participants) | 76 | 71 | 73 | 72
  Week 54: Total Score for Perceived Benefits | 0.6 (5.6) | 1.1 (4.2) | 0.2 (5.7) | -0.5 (6.3)
  Week 80: Total Score for Perceived Benefits: number analyzed (Participants) | 66 | 64 | 68 | 62
  Week 80: Total Score for Perceived Benefits | 0.1 (5.8) | 1.1 (4.8) | 1.3 (6.2) | -0.4 (5.1)

109. Secondary Outcome: Change in Diabetes Treatment Satisfaction Questionnaire (DTSQ)
Description: Change from baseline (week 0) in DTSQ is evaluated at week 54 and 80. The DTSQs items are scored on a 7-point graded response scale ranging from 6 to 0. Higher score indicates a higher level of glycaemia/treatment satisfaction.
Time Frame: (Week 0, week 54) and (week 0, week 80)
Population: The FAS included all randomised participants. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 77 | 77 | 76 | 77
Score on a scale
  Week 54: Perceived frequency of hyperglycaemia: number analyzed (Participants) | 76 | 71 | 73 | 72
  Week 54: Perceived frequency of hyperglycaemia | 0.6 (1.9) | 0.0 (1.5) | 0.0 (1.9) | 0.5 (1.7)
  Week 80: Perceived frequency of hyperglycaemia: number analyzed (Participants) | 66 | 64 | 68 | 62
  Week 80: Perceived frequency of hyperglycaemia | 0.9 (1.8) | 0.5 (1.8) | 0.6 (2.0) | 0.7 (1.9)
  Week 54: Perceived frequency of hypoglycaemia: number analyzed (Participants) | 76 | 71 | 73 | 72
  Week 54: Perceived frequency of hypoglycaemia | -0.7 (2.1) | -0.6 (1.6) | -0.4 (2.1) | -0.2 (1.5)
  Week 80: Perceived frequency of hypoglycaemia: number analyzed (Participants) | 66 | 64 | 68 | 62
  Week 80: Perceived frequency of hypoglycaemia | -0.9 (1.8) | -0.3 (1.7) | -0.4 (1.8) | -0.1 (1.5)
  Week 54: Treatment satisfaction: number analyzed (Participants) | 76 | 71 | 73 | 72
  Week 54: Treatment satisfaction | 1.5 (4.8) | 0.9 (5.2) | 1.3 (4.8) | 0.2 (5.5)
  Week 80: Treatment satisfaction: number analyzed (Participants) | 66 | 64 | 68 | 62
  Week 80: Treatment satisfaction | 1.3 (6.1) | 1.2 (5.7) | 0.0 (5.1) | 0.2 (6.2)

110. Secondary Outcome: Area Under the Concentration-time Curve (AUC) 0-4h of Mixed Meal Tolerance Test (MMTT) Stimulated C-peptide at Week 80 Relative to Baseline
Description: Area under the concentration-time curve, from 0 to 4 hours (AUC0-4h) of a mixed meal tolerance test (MMTT) stimulated C-peptide at week 80 is presented as ratio to baseline. AUC of C-peptide was measured as Nano moles*hour per liter (nmol*h/L).
Time Frame: 0 - 4 hours post-dose on week 0 and week 80
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AUC
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 63 | 64 | 62 | 58
Ratio of AUC | 0.566 (71.3) | 0.598 (70.2) | 0.373 (115.8) | 0.571 (100.9)

111. Secondary Outcome: AUC0-2h of C-peptide at Week 80 Relative to Baseline
Description: Area under the concentration-time curve, from 0 to 2 hours (AUC0-2h) of a MMTT stimulated C-peptide at week 80 is presented as ratio to baseline. AUC of C-peptide was measured as 'nmol*h/L'.
Time Frame: 0-2 hours post-dose on week 0 and week 80
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AUC
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 63 | 64 | 62 | 58
Ratio of AUC | 0.590 (74.5) | 0.619 (71.2) | 0.370 (111.5) | 0.540 (120.6)

112. Secondary Outcome: Cmax of C-peptide at Week 80 Relative to Baseline
Description: Maximum observed concentration (Cmax) of a MMTT stimulated C-peptide at week 80 is presented as ratio to baseline. Cmax of C-peptide was measured as nanomoles per liter (nmol/L).
Time Frame: 0-4 hours post-dose on week 0 and week 80
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of Cmax
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 63 | 64 | 62 | 58
Ratio of Cmax | 0.580 (74.8) | 0.592 (76.8) | 0.389 (109.0) | 0.568 (97.7)

113. Secondary Outcome: AUC0-4h of Glucose at Week 80 Relative to Baseline
Description: Area under the concentration-time curve, from 0 to 4 hours (AUC0-4h) of a MMTT stimulated glucose at week 80 is presented as ratio to baseline. AUC of glucose was measured as Milli moles*hour per liter (mmol*h/L).
Time Frame: 0 - 4 hours post-dose on week 0 and week 80
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AUC
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 63 | 64 | 63 | 58
Ratio of AUC | 1.129 (33.3) | 1.115 (32.6) | 1.136 (39.0) | 1.221 (26.6)

114. Secondary Outcome: AUC0-2h of Glucose at Week 80 Relative to Baseline
Description: Area under the concentration-time curve, from 0 to 2 hours (AUC0-2h) of a MMTT stimulated glucose at week 80 is presented as ratio to baseline. AUC of glucose was measured as 'mmol*h/L'.
Time Frame: 0-2 hours post-dose on week 0 and week 80
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AUC
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 63 | 64 | 63 | 58
Ratio of AUC | 1.119 (28.6) | 1.086 (28.1) | 1.070 (35.5) | 1.166 (21.7)

115. Secondary Outcome: Cmax of Glucose at Week 80 Relative to Baseline
Description: Maximum observed concentration (Cmax) of a MMTT stimulated glucose at week 80 is presented as ratio to baseline. Cmax of C-peptide was measured as 'mmol/L'.
Time Frame: 0-4 hours post-dose on week 0 and week 80
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of Cmax
Arm/Group | NNC0114-0006 + Liraglutide (Experimental) | NNC0114-0006 (Experimental) | Liraglutide (Experimental) | Placebo (Placebo)
Number analyzed (Participants) | 63 | 64 | 63 | 58
Ratio of Cmax | 1.114 (25.6) | 1.074 (28.7) | 1.104 (31.0) | 1.155 (21.5)

ADVERSE EVENTS:
Time Frame: Weeks 0-80
Description: All reported adverse events are treatment-emergent. Results are based on the safety analysis set (SAS) which included all participants who received at least one dose of randomised treatment.
Groups:
- NNC0114-0006 + Liraglutide: Participants received 12 mg/kg dose of NNC0114-0006 every 6 weeks, intravenously for 54 weeks. Participants took 0.6 mg of liraglutide, once daily, subcutaneously, for first two weeks, 1.2 mg for next 2 weeks and 1.8 mg for rest of the treatment period. Participants received treatment for 54 weeks followed by an off-treatment observation period of 26 weeks. Participants continued their pre-trial insulin treatment throughout the trial.
- NNC0114-0006: Participants received 12 mg/kg dose of NNC0114-0006 every 6 weeks, intravenously for 54 weeks. Participants took liraglutide placebo once daily, subcutaneously, with the volume of placebo equivalent to the volume liraglutide 0.6 mg, 1.2 mg and 1.8 mg. Participants received treatment for 54 weeks followed by an off-treatment observation period of 26 weeks. Participants continued their pre-trial insulin treatment throughout the trial.
- Liraglutide: Participants received NNC0114-0006 placebo (volume equivalent to NNC0114-0006 dose of 12 mg/kg) every 6 weeks, intravenously for 54 weeks. Participants took 0.6 mg of liraglutide, once daily, subcutaneously, for first two weeks, 1.2 mg for next 2 weeks and 1.8 mg for rest of the treatment period. Participants received treatment for 54 weeks followed by an off-treatment observation period of 26 weeks. Participants continued their pre-trial insulin treatment throughout the trial.
- Placebo: Participants received NNC0114-0006 placebo (volume equivalent to NNC0114-0006 dose of 12 mg/kg) every 6 weeks, intravenously for 54 weeks. In addition to that, participants took liraglutide placebo once daily subcutaneously, with the volume of placebo equivalent to the volume liraglutide 0.6 mg, 1.2 mg and 1.8 mg. Participants received treatment for 54 weeks followed by an off-treatment observation period of 26 weeks. Participants continued their pre-trial insulin treatment throughout the trial.
Arm/Group | NNC0114-0006 + Liraglutide | NNC0114-0006 | Liraglutide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/77 | 1/76 | 0/77
Serious Adverse Events (participants affected / at risk) | 7/77 | 5/77 | 9/76 | 11/77
Other Adverse Events (participants affected / at risk) | 57/77 | 55/77 | 62/76 | 54/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NNC0114-0006 + Liraglutide (N=77) | NNC0114-0006 (N=77) | Liraglutide (N=76) | Placebo (N=77)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Genital herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ketosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Peritonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Routine health maintenance (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal muscular atrophy (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Traumatic shock (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NNC0114-0006 + Liraglutide (N=77) | NNC0114-0006 (N=77) | Liraglutide (N=76) | Placebo (N=77)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 4 (5) | 4 (4) | 2 (4)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 0 (0) | 4 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 9 (11) | 0 (0) | 4 (4) | 7 (10)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 7 (8) | 4 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (6) | 5 (6) | 2 (3)
Blood creatine phosphokinase increased (Investigations) | 4 (4) | 2 (2) | 2 (2) | 3 (3)
Blood immunoglobulin E increased (Investigations) | 1 (1) | 3 (3) | 7 (7) | 4 (5)
Contusion (Injury, poisoning and procedural complications) | 4 (5) | 1 (2) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 4 (4) | 5 (7) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 14 (15) | 2 (2) | 11 (13) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 15 (21) | 9 (15) | 13 (22) | 9 (11)
Dyspepsia (Gastrointestinal disorders) | 5 (8) | 3 (6) | 3 (5) | 4 (4)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (6)
Fatigue (General disorders) | 4 (4) | 4 (4) | 6 (6) | 2 (4)
Gastroenteritis (Infections and infestations) | 3 (4) | 6 (7) | 5 (6) | 4 (5)
Headache (Nervous system disorders) | 11 (21) | 10 (12) | 10 (11) | 11 (17)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (15) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 6 (7) | 12 (14) | 2 (3) | 2 (2)
Lipase increased (Investigations) | 5 (6) | 1 (1) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 20 (35) | 27 (63) | 25 (50) | 25 (45)
Nausea (Gastrointestinal disorders) | 19 (33) | 6 (10) | 42 (62) | 9 (13)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 13 (18) | 5 (8) | 9 (11)
Pharyngitis (Infections and infestations) | 3 (3) | 4 (5) | 0 (0) | 3 (4)
Pyrexia (General disorders) | 3 (4) | 7 (9) | 7 (12) | 4 (4)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 0 (0) | 5 (6)
Respiratory tract infection viral (Infections and infestations) | 5 (7) | 1 (1) | 3 (6) | 2 (2)
Rhinitis (Infections and infestations) | 5 (5) | 3 (3) | 3 (5) | 5 (6)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (4) | 4 (6)
Sinusitis (Infections and infestations) | 1 (1) | 2 (5) | 1 (1) | 4 (4)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 8 (13) | 5 (9) | 4 (4) | 7 (9)
Vomiting (Gastrointestinal disorders) | 14 (24) | 0 (0) | 17 (34) | 4 (5)
Weight decreased (Investigations) | 4 (4) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-09-17): https://cdn.clinicaltrials.gov/large-docs/55/NCT02443155/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-17): https://cdn.clinicaltrials.gov/large-docs/55/NCT02443155/SAP_001.pdf